| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan 207040 for an open label, randomised, parallel group clinical study to evaluate the effect of the Connected Inhaler System (CIS) on adherence to Relvar/Breo ELLIPTA therapy, in asthmatic subjects with poor control. |
|---|---|---|
| Compound Number | : | GW685698+GW642444 (GSK2285997) |
| <b>Effective Date</b> | : | 21-FEB-2019 |

## **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report (CSR) for Protocol 207040.
- This RAP is intended to describe the study population, efficacy and safety analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the final Statistical Analysis Complete (SAC) deliverable.

## RAP Author(s):

| Author | Date |
|---|---|
| Lead PPD Principal Statistician (Respiratory, Biostatistics UK) | 14 FEB 2019 |
| Co-Authors PPD Associate Statistician, (Respiratory, Biostatistics India) | 15 FEB 2019 |
| Study Statistician (Respiratory, Biostatistics UK) | 14 FEB 2019 |

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## The GlaxoSmithKline group of companies

## **RAP Team Review Confirmations (Method E-mail):**

| Reviewer | Date |
|---|---|
| PPD | |
| Clinical Investigation Leader (Respiratory, Head Unit | 15 FEB 2019 |
| Physician, Clinical Development) | |
| | 15 FED 2010 |
| Clinical Development Director (Respiratory, Head Unit Physician, Clinical Pharmacology and Discovery Medicine) | 15 FEB 2019 |
| PPD PPD | |
| Project Statistician (Respiratory, Biostatistics UK) | 15 FEB 2019 |
| PPD | 18 FEB 2019 |
| Lead Programmer (Respiratory, Biostatistics UK) | 10 FED 2019 |

## **Clinical Statistics and Clinical Programming Line Approvals**

## (Method: Pharma TMF eSignature):

| Approver | Date |
|---------------------------------------------------------------|-------------|
| Senior Statistics Director (Respiratory, Clinical Statistics) | 21 FEB 2019 |
| Programming Manager (Respiratory, Clinical Programming) | 21 FEB 2019 |

## **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | INTRO | DDUCTION | N | 8 |
| 2. | CLIMA | ANDV OF I | KEY PROTOCOL INFORMATION | 0 |
| ۷. | 2.1. | | | |
| | | | to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | | ojectives and Endpoints | |
| | 2.3. | | esign | |
| | 2.4. | Statistica | ıl Hypothesis | 14 |
| 3. | PLAN | NED ANAI | LYSES | 16 |
| | 3.1. | Interim A | nalyses | 16 |
| | 3.2. | Final Ana | alyses | 16 |
| 4. | ٨٨٨١ | veie dod | ULATIONS | 17 |
| 4. | 4.1. | | Deviations | |
| | 4.1. | Protocor | Deviations | 17 |
| 5. | | | ONS FOR DATA ANALYSES AND DATA HANDLING | |
| | | | ) | |
| | 5.1. | | eatment & Sub-group Display Descriptors | |
| | 5.2. | | Definitions | |
| | 5.3. | | re Studies | |
| | 5.4. | Examina | tion of Covariates, Other Strata and Subgroups | 21 |
| | | 5.4.1. | Covariates and Other Strata | |
| | | 5.4.2. | Examination of Subgroups | 21 |
| | 5.5. | Multiple ( | Comparisons and Multiplicity | |
| | 5.6. | Other Co | nsiderations for Data Analyses and Data Handling | |
| | | Conventi | ons | 22 |
| 6. | STUD | Y POPUL | ATION ANALYSES | 23 |
| | 6.1. | Overview | of Planned Study Population Analyses | 23 |
| | 6.2. | | entary Information for Study Population Displays | |
| | | 6.2.1. | Disease and Baseline Characteristics | 23 |
| | | 6.2.2. | Preferred Time of Dosing | |
| | | 6.2.3. | Study Medication Exposure and Compliance | |
| | | 6.2.4. | HCP dashboard review | |
| _ | | NA (ON / A NI A | LVOFO | 0.5 |
| 7. | | | LYSES | |
| | 7.1. | | Efficacy Analysis | |
| | | 7.1.1. | Endpoint | |
| | | 7.1.2. | Summary Measure | |
| | | 7.1.3. | Population of Interest | |
| | | 7.1.4. | Strategy for Intercurrent (Post-Randomisation) Events 7.1.4.1. Events prior to premature discontinuation of | 26 |
| | | | 7.1.4.1. Events prior to premature discontinuation of the ELLIPTA maintenance sensor | 28 |
| | | | 7.1.4.2. Events following premature discontinuation of | 20 |
| | | | the ELLIPTA maintenance sensor | 28 |
| | | 7.1.5. | Statistical Analyses / Methods | |
| | | | 7.1.5.1. Statistical Methodology Specification | |
| | 72 | Seconda | ry Efficacy Analyses | 31 |


| 00=046 |
|--------|
| 207040 |

| 7.2.1. | ELLIPTA | Adherence N | Measure Endpoints | 31 |
|---|---|---|---|---|
| | 7.2.1.1. | | Measure | |
| | 7.2.1.2. | | of Interest | |
| | 7.2.1.3. | | r Intercurrent (Post-Randomisation) | |
| | | | | 32 |
| | | 7.2.1.3.1. | | |
| | | 7.2.1.0.1. | discontinuation of the ELLIPTA | |
| | | | maintenance sensor | 22 |
| | | 70400 | | 32 |
| | | 7.2.1.3.2. | 0 1 | |
| | | | discontinuation of the ELLIPTA | |
| | | | maintenance sensor | |
| | 7.2.1.4. | | Analyses / Methods | 32 |
| | 7.2.1.5. | Statistical Analyses / Methodology | | |
| | | Specification | on | 33 |
| | | 7.2.1.5.1. | The percentage of ELLIPTA doses | |
| | | | taken (daily adherence) between | |
| | | | the beginning of Month 4 and the | |
| | | | end of Month 6 | 33 |
| | | 7.2.1.5.2. | The percentage of ELLIPTA doses | |
| | | 7.2.1.0.2. | taken (daily adherence) between | |
| | | | the beginning of Month 1 and the | |
| | | | end of Month 6 | 35 |
| | | 7.2.1.5.3. | | |
| | | 1.2.1.3.3. | The percentage of ELLIPTA doses | |
| | | | taken (daily adherence) between | |
| | | | the beginning of Month 1 and the | 0- |
| | | | end of Month 3 | |
| 7.2.2. | | | on Use Endpoints | |
| | 7.2.2.1. | | | |
| | 7.2.2.2. | | of Interest | 39 |
| | 7.2.2.3. | | r Intercurrent (Post-Randomisation) | |
| | | | | 40 |
| | | 7.2.2.3.1. | Events following premature | |
| | | | discontinuation of the MDI sensor | 42 |
| | 7.2.2.4. | Statistical / | Analyses / Methods | 42 |
| | 7.2.2.5. | Statistical Analyses / Methodology | | |
| | | Specification | on | 42 |
| 7.2.3. | Asthma ( | | oints | |
| | 7.2.3.1. | | Measure | |
| | 7.2.3.2. | | of Interest | |
| | 7.2.3.3. | | r Intercurrent (Post-Randomisation) | |
| | 7.2.0.0. | | | 45 |
| | | 7.2.3.3.1. | Change from baseline | |
| | | 1.2.3.3.1. | | |
| | | | (Randomisation) in ACT total | 4.5 |
| | | 70000 | score at Month 6 (Visit 10) | 40 |
| | | 7.2.3.3.2. | Percentage of patients becoming | |
| | | | controlled as defined as an | |
| | | | Asthma Control Test score ≥20 at | |
| | | | Month 6 (Visit 10) | 45 |
| | | 7.2.3.3.3. | Percentage of patients with an | |
| | | | increase from baseline ≥ 3 in ACT | |
| | | | total score at Month 6 (Visit 10) | 46 |
| | | | , | |

| | | | 7.2.3.3.4. | Percentage of patients who have either an ACT total score of ≥ 20 and/or an increase from baseline of ≥ 3 in ACT total score at Month 6 (Visit 10) | 46 |
|---|---|---|---|---|---|
| | | 7.2.3.4. | | Analyses / Methodology | |
| | | | 7.2.3.4.1. | Change from baseline in ACT total | |
| | | | | score at month 6 | 47 |
| | | | 7.2.3.4.2. | | 47 |
| | | | 7.2.3.4.3. | | |
| | | | | ACT total score at month 6 | 48 |
| | | | 7.2.3.4.4. | | |
| | | | | increase from baseline of ≥ 3 in | |
| | | | | ACT total score at Month 6 (Visit | |
| | | | | 10) | 49 |
| 7.3. | | | | S | |
| | 7.3.1. | | | Adherence Measure Analyses | |
| | | 7.3.1.1. | | Magazira | |
| | | 7.3.1.2.<br>7.3.1.3. | | Measure | |
| | | 7.3.1.3.<br>7.3.1.4. | | of Interestr Intercurrent (Post-Randomisation) | 50 |
| | | 7.5.1.4. | | | 50 |
| | | | | Events prior to premature | 50 |
| | | | 7.0.1.4.1. | discontinuation of the ELLIPTA | |
| | | | | maintenance sensor | 51 |
| | | | 7.3.1.4.2. | | |
| | | | | discontinuation of the ELLIPTA | |
| | | | | maintenance sensor | 51 |
| | | 7.3.1.5. | Statistical A | Analyses / Methods | |
| | | 7.3.1.6. | | Analyses / Methodology | |
| | | | | on | 52 |
| | | | 7.3.1.6.1. | The percentage of ELLIPTA doses | |
| | | | | taken (daily adherence) between | |
| | | | | the beginning of Month 4 and the | |
| | | | | end of Month 6 | <mark>52</mark> |
| | 7.3.2. | | | re Utilization Analyses | |
| | | 7.3.2.1. | | | |
| | | 7.3.2.2. | | of Interest | |
| | 7.3.3. | | | eported Outcomes (PROs) Analyses | |
| | | 7.3.3.1. | | | |
| | | 7.3.3.2. | | Measure | |
| | | 7.3.3.3. | Population | of Interest | 56 |
| | | 7.3.3.4. | | r Intercurrent (Post-Randomisation) | |
| | | | | Develope of actions and time | 56 |
| | | | 7.3.3.4.1. | 3 - 3 - 6 - | |
| | | | | responder threshold of ≥ 0.09 | |
| | | | | points improvement from baseline (randomisation) for the ASUI total | |
| | | | | score at Month 6 (Visit 10) | 57 |
| | | | | Source at Mortill of Albit 10) | 57 |

| | | | | 7.3.3.4.2. | Change from baseline | |
|---|---|---|---|---|---|---|
| | | | | | (randomisation) in ASUI total | |
| | | | | | score at month 6 (Visit 10) | 57 |
| | | | | 7.3.3.4.3. | Percentage of patients meeting a | |
| | | | | | responder threshold of ≥ 4 points | |
| | | | | | improvement (decrease) from | |
| | | | | | baseline (randomisation) for the | |
| | | | | | SGRQ total score at month 6 (Visit | |
| | | | | | 10) | 57 |
| | | | | 7.3.3.4.4. | Change from baseline | |
| | | | | 7.0.0.1.1. | (Randomisation) in SGRQ total | |
| | | | | | score at Month 6 (Visit 10) | 58 |
| | | | | 7.3.3.4.5. | Change from baseline (Screening) | |
| | | | | 7.5.5. <del>4</del> .5. | in PAM-13, MARS-A, and BMQ | |
| | | | | | total score at Month 6 (Visit 10) | 59 |
| | | | 7225 | Statistical A | | 50 |
| | | | 7.3.3.5. | | Analyses / Methodology | FO |
| | | | | • | on<br>Increase from Baseline of ≥ 0.09 | 50 |
| | | | | 7.3.3.5.1. | | |
| | | | | | in ASUI total score at Month 6 | |
| | | | | 70050 | (Visit 10) | 58 |
| | | | | 7.3.3.5.2. | 3 | |
| | | | | | (Randomisation) in ASUI total | |
| | | | | | score at Month 6 (Visit 10) | 59 |
| | | | | 7.3.3.5.3. | Increase from Baseline of ≥ 4 in | |
| | | | | | SGRQ total score at Month 6 (Visit | |
| | | | | | 10) | 60 |
| | | | | 7.3.3.5.4. | • | |
| | | | | | (Randomisation) in SGRQ total | |
| | | | | | score at Month 6 (Visit 10) | 60 |
| | | 7.3.4. | | | ed Exhaled Nitric Oxide (FeNO) and | |
| | | | • | | (PEF) Analyses | |
| | | | 7.3.4.1. | | | |
| | | | 7.3.4.2. | | Measures | |
| | | | | | of Interest | 62 |
| | | | 7.3.4.4. | 0, | r Intercurrent (Post-Randomisation) | |
| | | | | | | 62 |
| | | | 7.3.4.5. | | Analyses / Methodology | |
| | | | | | on | |
| | | 7.3.5. | Qualitative | e data from e | exit interviews | 63 |
| ^ | 0.4 = == | T\/ | <b>1050</b> | | | 0.4 |
| 8. | | | | | | |
| | 8.1. | | | | | |
| | 8.2. | | | • | est | |
| | 8.3. | | | | | |
| | 8.4. | Otner Sa | atety Measi | ıres | | 65 |
| 9. | REFE | RENCES | | | | 66 |
| 10 | ۸۵۵۲۰ | NDICEC | | | | 67 |
| ıυ. | | | | | es | |
| | 10.1. | | | | edule of Events | |
| | 10.2. | | | | ws | |
| | 10.2. | Appendi | x Z. ASSESS | sineni vvindo | w5 | 1 |


| 20 | 70 | ۱1 | Λ |
|----|-----|----|---|
| 20 | / U | 14 | U |

| | 10.2.1.<br>10.2.2. | General Definitions of Assessment Windows for Adherence and | 71 |
|---|---|---|---|
| | | Rescue Medication Use Analyses | 71 |
| 10.3. | | x 3: Study Phases and Treatment Emergent Adverse | |
| | Events | | |
| | 10.3.1. | Study Phases | |
| | | 10.3.1.1. Study Phases for Concomitant Medication | 73 |
| | | 10.3.1.2. Study Phases for Asthma Exacerbations | |
| | | 10.3.1.3. Treatment Emergent Flag for Adverse Events | 74 |
| 10.4. | Appendi | x 4: Data Display Standards & Handling Conventions | 75 |
| | 10.4.1. | Reporting Process | 7 <mark>5</mark> |
| | 10.4.2. | Reporting Standards | 7 <mark>5</mark> |
| 10.5. | Appendi | x 5: Derived and Transformed Data | <mark>77</mark> |
| | 10.5.1. | General | <mark>77</mark> |
| | 10.5.2. | Study Population | <mark>77</mark> |
| | 10.5.3. | Efficacy | 79 |
| | | 10.5.3.1. ELLIPTA Device Sensor Assessments | <mark>79</mark> |
| | | 10.5.3.2. MDI Device Sensor Assessments | 88 |
| | | 10.5.3.3. Patient Reported Outcomes | 96 |
| | 10.5.4. | Safety | 100 |
| 10.6. | Appendi | x 6: Reporting Standards for Missing Data | 101 |
| | 10.6.1. | Premature Withdrawals | |
| | 10.6.2. | Handling of Missing Data | 101 |
| | 10.6.3. | Handling of Partial Dates | |
| 10.7. | Appendi | x 7: Abbreviations & Trade Marks | |
| | 10.7.1. | Abbreviations | |
| | 10.7.2. | Trademarks | 104 |
| 10.8. | Appendi | x 8: List of Data Displays | 105 |
| | 10.8.1. | Data Display Numbering | 105 |
| | 10.8.2. | Mock Example Shell Referencing | |
| | 10.8.3. | Deliverables | |
| | 10.8.4. | Study Population Tables | 106 |
| | 10.8.5. | Study Population Figures | 112 |
| | 10.8.6. | Efficacy Tables | 112 |
| | 10.8.7. | Efficacy Figures | |
| | 10.8.8. | Safety Tables | |
| | 10.8.9. | ICH Listings | |
| | 10.8.10. | | |
| 10.9. | Appendi | x 9: Example Mock Shells for Data Displays | |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report (CSR) for Protocol 207040 [GlaxoSmithKline Document Number: 2016N307903 01 (Dated: 10SEP2018)].

| Revision Chronology: | | |
|----------------------|-------------|-------------|
| 2016N307903_00 | | |
| 2016N307903_01 | 10-SEP-2018 | Amendment 1 |

All data displays (Tables, Figures & Listings) will use the term "Subject" which reflects CDISC and GSK Data Display Standards terminology.

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the planned statistical analysis specified in protocol amendment 1 are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Duration of run-in included in analysis models as a continuous covariate, measured in days. | Duration of run-in included in analysis models as a categorical covariate of number of visits. | Participants can complete the run-in period in 1, 2 or 3 visits, use of a categorical covariate is more flexible than the assumption of a linear relationship. |
| Missing data due to a medical device incident will be assumed to be missing at random within the last 3 months treatment period. | Missing data due to a medical device incident will be assumed to be missing at random within each month of the treatment period. | Monthly adherence rates are used within the imputation model to allow for variation in adherence over time. |
| Participants who prematurely discontinue from study will have their post-withdrawal daily adherence data imputed using data from the control arm | Participants who prematurely discontinue from use of the ELLIPTA maintenance sensor will have subsequent adherence data imputed using data from the control arm | The ELLIPTA maintenance sensor may be discontinued without withdrawal from the study |
| Protocol Section 11.3 Populations for Analyses | RAP Section 4 Analysis<br>Populations | The analysis populations have been updated to follow the study populations standard definitions and statistical displays |

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| | Mean change from baseline<br>(Randomisation) in ASUI and<br>SGRQ total score at Month 6<br>included in the RAP as an<br>additional endpoint | To support the exploratory summaries and analyses for ASUI and SGRQ continuous endpoint |
| Composite endpoint - Percentage of patients who have either an ACT total score of ≥ 20 or an increase from baseline of ≥ 3 in ACT total score at Month 6 (Visit 10). | Composite endpoint - Percentage of patients who have either an ACT total score of ≥ 20 and/or an increase from baseline of ≥ 3 in ACT total score at Month 6 (Visit 10). | The condition 'and/or' will be applied to the composite ACT endpoint to replace 'or' to clarify that participants who achieve both an ACT total score of ≥ 20 and an increase from baseline of ≥ 3 in ACT total score at Month 6, in addition to those who only achieve one, will be considered a responder. |
| | Change from baseline (Visit 2, 3 or 4) in FeNO measured at Month 1 (Visit 5) and Month 6 (Visit 10) | To support the exploratory summary of impact of adherence on the biomarker Fractionated Exhaled Nitric Oxide (FeNO) |

## 2.2. Study Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To compare the effect of 6 months use of the CIS on adherence to ELLIPTA maintenance therapy when both the participant and the HCP are supplied with data from the maintenance sensor versus no data supplied to the participant and HCP (Arm 1 vs Arm 5) | Percentage of ELLIPTA doses taken (daily adherence <sup>1.</sup> ) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor |
| Secondary Objectives | Secondary Endpoints |
| To compare the effect of 6 months use of the CIS on adherence to ELLIPTA maintenance therapy for the following aspects of the CIS: • Maintenance data only supplied to participants versus no data supplied to the participant (Arm 2 vs Arm 5) • Rescue and Maintenance data supplied to participant and HCP versus no data supplied to the participant and HCP (Arm 3 vs Arm 5) • Rescue and Maintenance data only supplied to participant versus no data supplied to the participant (Arm 4 vs | Percentage of ELLIPTA doses taken (daily adherence <sup>1.</sup> ) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor |

| Objectives | Endpoints |
|---|---|
| Arm 5) | |
| To compare the effect of the CIS on adherence to ELLIPTA maintenance therapy of the individual CIS treatment arms versus no data supplied to the participant and HCP. | <ul> <li>Percentage of ELLIPTA doses taken (daily adherence<sup>1.</sup>) between the beginning of month 1 and the end of month 3</li> <li>Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 1 and the end of month 6</li> </ul> |
| To evaluate the effect of 6 months use of the CIS on a participant's rescue medicine usage | Percentage of rescue free days measured between the beginning of month 4 and the end of month 6 as determined by the rescue sensor records of date, time, and number of inhaler actuations. |
| | <ul> <li>Total rescue use measured between the beginning of<br/>month 4 and the end of month 6 as determined by the<br/>rescue sensor records of date, time, and number of<br/>inhaler actuations.</li> </ul> |
| To evaluate the effect of 6 months use with the CIS on a participant's asthma control | Change from baseline (Randomisation) in ACT total score<br>at Month 6, measured at baseline (Visit 2, 3 or 4) and<br>Month 6 (Visit 10) |
| | <ul> <li>Percentage of patients becoming controlled as defined as<br/>an Asthma Control Test score ≥20 at Month 6 (Visit 10)</li> </ul> |
| | <ul> <li>Percentage of patients with an increase from baseline ≥ 3<br/>in ACT total score at Month 6 (Visit 10)</li> </ul> |
| | <ul> <li>Composite endpoint - Percentage of patients who have<br/>either an ACT total score of ≥ 20 and/or an increase from<br/>baseline of ≥ 3 in ACT total score at Month 6 (Visit 10).</li> </ul> |
| Exploratory and Other Objectives | Exploratory Endpoints |
| To evaluate the effect of 6 months use of the CIS on adherence to ELLIPTA maintenance therapy on the following aspects of the CIS: HCP having access to sensor data Rescue Medication data being available | Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor |
| To evaluate the effect of 6 months use with CIS on health care utilisation | Health care utilisation endpoints will include the following and will be collected from a participant's medical records. |
| | Number of outpatient visits relating to asthma |
| | Number of primary care visits relating to study HCP dashboard review (for relevant study arms) |
| | Number of and duration of hospitalisations, and ER visits due to asthma |
| | Annualised rate of severe exacerbations |
| | Number of unscheduled visits to primary care related to Asthma |
| To evaluate the effect of 6 months use with CIS on the following patient reported | <ul> <li>Percentage of patients meeting a responder threshold of<br/>≥ 0.09 points improvement from baseline</li> </ul> |

| Objectives | Endpoints |
|---|---|
| outcomes (PROs): | (Randomisation) for the ASUI total score at Month 6 |
| <ul><li>Asthma Symptom Utility Index<br/>(ASUI)</li><li>St Georges Respiratory</li></ul> | <ul> <li>Mean change from baseline (Randomisation) in ASUI total score at Month 6</li> </ul> |
| Questionnaire (SGRQ) • Patient Activation Measure (PAM) • Medication Adherence Report | <ul> <li>Percentage of patients meeting a responder threshold of<br/>≥ 4 points improvement from baseline (Randomisation)<br/>for the SGRQ total score at Month 6</li> </ul> |
| Scale for Asthma (MARS-A) • Beliefs in Medicine Questionnaire (BMQ). | <ul> <li>Mean change from baseline (Randomisation) in SGRQ<br/>total score at Month 6</li> </ul> |
| (DIVIQ). | <ul> <li>Mean change from baseline (Screening) in PAM total<br/>score at Month 6</li> </ul> |
| | <ul> <li>Mean change from baseline (Screening) in MARS-A total<br/>score at Month 6</li> </ul> |
| | <ul> <li>Mean change from baseline (Screening) at Month 6 in<br/>BMQ:</li> </ul> |
| | <ul> <li>General Benefit score</li> </ul> |
| | <ul> <li>General Harm score</li> </ul> |
| | <ul> <li>General Overuse score</li> </ul> |
| | <ul> <li>Specific Necessity score</li> </ul> |
| | <ul> <li>Specific Concern score</li> </ul> |
| To assess the reliability and usability of the CIS | <ul> <li>Incidence of Medical Device Incidents between the<br/>beginning of Month 1 and the end of Month 6.</li> </ul> |
| To explore impact of adherence on<br>the biomarker Fractionated Exhaled<br>Nitric Oxide (FeNO) | <ul> <li>FeNO at Screening (Visit 1), Randomisation (Visit 2,3 or 4), Month 1 (Visit 5) and Month 6 (Visit 10).</li> <li>Change from baseline (Visit 2, 3 or 4) in FeNO measured at Month 1 (Visit 5) and Month 6 (Visit 10)</li> </ul> |
| To explore impact of adherence on<br>the physiological marker Peak | <ul> <li>PEF at Screening (Visit 1), Randomisation (Visit 2,3 or 4),<br/>Month 1 (Visit 5) and Month 6 (Visit 10).</li> </ul> |
| Expiratory Flow (PEF) | <ul> <li>Change from baseline (Visit 2, 3 or 4) in PEF measured<br/>at Month 1 (Visit 5) and Month 6 (Visit 10)</li> </ul> |
| To characterize patient experience of the CIS for participants. | <ul> <li>Exit Questionnaires at Month 6 (Visit 10)</li> </ul> |
| the CIS for participants | <ul> <li>Exit Interviews for a sub set of participants at Month 6<br/>(Visit 10)</li> </ul> |
| Safety Objectives | Safety Endpoints |
| To evaluate the incidence of SAEs, Non-<br>Serious Adverse Events that lead to<br>withdrawal from study and Non-Serious<br>Adverse Drug Reactions in asthmatic | <ul> <li>SAEs, Non-Serious Adverse Events that lead to<br/>withdrawal and Non-Serious Adverse Drug Reactions</li> </ul> |
| participants using the CIS | pant taking one dose of Relyar/Breo FLLIPTA within a 2/Lhour |

 Daily adherence is defined as the participant taking one dose of Relvar/Breo ELLIPTA, within a 24-hour period, starting at 12.00am each day

## 2.3. Study Design



| Overview of Study Do | esign and Key Features |
|---|---|
| | [GlaxoSmithKline Document Number 2016N307903_01]. |
| Time & Events | Refer to Appendix 1: Schedule of Activities |
| Treatment<br>Assignment | All randomised participants will receive Relvar/Breo ELLIPTA, at the dose allocated at the run in. Salbutamol Metered Dose Inhaler (MDI) rescue medication will be prescribed to participants to use as needed throughout the study for relief of asthma symptoms as per usual practice |
| | All participants will have sensors attached to both their Relvar/Breo ELLIPTA and salbutamol MDI. It is the type of data provided by the CIS (either Relvar/Breo ELLIPTA alone or Relvar/Breo ELLIPTA and salbutamol MDI), as well as who sees that data, (participant alone or participant and HCP), that defines the treatment arms. |
| | Participants will be randomized 1:1:1:1 to one of the five treatments arms for the duration of the treatment period: |
| | Arm 1: Data on Maintenance use supplied to Participant (app) and HCP (dashboard) |
| | Arm 2: Data on Maintenance use supplied to Participant (app) |
| | <ul> <li>Arm 3: Data on Maintenance and Rescue use supplied to Participant (app) and HCP (dashboard)</li> </ul> |
| | <ul> <li>Arm 4: Data on Maintenance and Rescue use supplied to Participant (app)</li> </ul> |
| | Arm 5: No data supplied to Participant or HCP |
| | The treatment period for the study is 6 months. However, due to the flexible run in period a participant could be on the study for approximately 7, 8 or 9 months in total. |
| | GSK RandAll NG will be used to generate the randomisation schedule. Centralized randomisation will be used. GSK RAMOS NG will be used for treatment allocation. |

## 2.4. Statistical Hypothesis

The main purpose of the study is to compare the effect of 6 months use with the Connected Inhaler System (CIS) on adherence to Relvar/Breo ELLIPTA maintenance therapy with adherence to Relvar/Breo ELLIPTA maintenance therapy without CIS use (sensor alone), in participants with poorly controlled asthma.

All participants receive Relvar/Breo ELLIPTA, either at the dose they are already prescribed or at the equivalent dose to their current ICS/LABA maintenance therapy if switched onto Relvar/Breo ELLIPTA at enrolment. All participants will have sensors attached to both their Relvar/Breo ELLIPTA and Salbutamol MDI. It is the type of data provided by the CIS (either Relvar/Breo ELLIPTA alone or Relvar/Breo ELLIPTA and salbutamol MDI), as well as who sees that data (participant alone or participant and HCP) that defines the treatment arms.

This study aims to demonstrate the superiority of the CIS on adherence to Relvar/Breo ELLIPTA with an app compared to Relvar/Breo ELLIPTA (with sensor alone).

The primary endpoint is mean percentage of ELLIPTA doses taken (daily adherence) between Months 4 and 6 as determined by the maintenance sensor daily adherence over the last three months of the study period (between months 4 to 6).

The test for the primary treatment comparison will be a test between Arm 1 versus Arm 5. This will be based on a two-sided hypothesis testing approach: the null hypothesis is the difference between Arm 1 and Arm 5 is equal to zero. The alternative hypothesis is that the difference is not equal to zero. The hypotheses associated with the statistical test of the primary endpoint are written below:

H0: 
$$Ti - Tj = 0$$

(where  $i = Arm\ 1$  and  $j = Arm\ 5$ ) The null hypothesis: that the difference in response between Arm 1 and Arm 5 is zero.

Ha: 
$$Ti - Tj \neq 0$$

The alternative hypothesis: that the difference is not zero.

Other comparisons of interest for the primary endpoint are the individual comparisons of Arms 2, 3 and 4 with Arm 5 in order to obtain estimated mean treatment differences, 95% confidence intervals (CIs) and p-values. This will be a descriptive comparison to inform on the relative benefits of the individual aspects of the CIS and no formal inference is planned.

The effect on adherence to maintenance therapy between arms with HCP and no HCP interaction i.e. Arm 1 v Arm 2 and Arm 3 v Arm 4, and arms with rescue medication use feedback versus none i.e. Arm 1 v Arm 3 and Arm 2 v Arm 4, will be also assessed.

The comparisons of interest for the other secondary and safety endpoints are as stated above for the primary endpoint. Arms 1, 2, 3 and 4 will be individually compared to Arm


207040

5, as relevant to the endpoint, to obtain estimated mean treatment differences, 95% confidence intervals and p-values. This will be a descriptive comparison and no formal inference is planned.

## 3. PLANNED ANALYSES

To minimize the risk of breaking the study blind during the pre-programming of analysis datasets and displays for the final analyses, an unblinded team of programmers will scramble the data in a secure area according to a pre-defined blinding strategy, before releasing to Clinical Statistics and Programming (S&P).

## 3.1. Interim Analyses

An interim analysis was originally planned to be conducted when 50% of subjects complete 6 months of study treatment in order to conduct a sample size re-estimation. However the requirement for the interim analysis and sample size-re-estimation was decided no longer necessary and removed from the study protocol.

## 3.2. Final Analyses

The final planned analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study or have been withdrawn as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management (DM).
- 3. System Independent (SI) data to Study Data Tabulation Model (SDTM) data conversion has completed by Conversion Service Provider at Source Data Lock (SDL).
- 4. All criteria for unblinding the randomisation codes have been met.
- 5. Randomisation codes have been distributed according to RandAll NG procedures. Release of randomisation code, unblinding of study treatment and participant level treatment of SDTM data, and related quality control activities have been completed by S&P.
- 6. DBF on SDTM datasets has been declared by DM upon receipt of the final, treatment unblinded SDTM data from S&P.

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All participants | All participants who signed the ICF | Study Population |
| Screened | All participants who were screened for eligibility. | Study Population |
| Enrolled | All participants who passed screening and entered the study. Included are: Run-in Failures; Randomized Participants | Study Population Safety |
| | Note screening failures are excluded from the Enrolled population as they did not enter the study. | |
| Randomized | <ul> <li>All participants who were randomly assigned to a treatment arm in the study.</li> <li>This population will be based on the treatment arm the participant was randomised to.</li> </ul> | Study Population |
| Intent-To-Treat<br>(ITT) | <ul> <li>The ITT population comprises all randomised participants, excluding those who were randomised in error. A participant who is recorded as a screen or runin failure but is randomised, and does not receive a dose of study treatment, is considered to have been randomised in error. Any other participant who received a randomisation number will be considered to have been randomised.</li> <li>This population will be based on the treatment arm the participant was randomised to.</li> </ul> | Study Population Efficacy (ELLIPTA Adherence, Rescue Medications Use, PRO, PEF and FeNO) Safety |

Refer to Section 10.8 Appendix 8: List of Data Displays which will detail the population used for each display.

## 4.1. Protocol Deviations

This dataset will be the basis for the summaries and listings of protocol deviations. A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

## 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| | | | | | | Treatment Group Descriptions | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Sensor I | var/Breo ELLIPTA Salbutamol/Rescue<br>Sensor Data MDI Sensor Data<br>Available to Available to | | nsor Data RandAll NG Randomisation System | | RandAll NG Randomisation System | Data Displays for Reporting | | |
| Arm | Participant | НСР | Participant | НСР | Code | Description | Full Description | Short<br>Description | Order<br>in<br>Table,<br>List,<br>Figure<br>(TLF) |
| 1 | Х | Х | | | 1 | Data on Maintenance use supplied to Participant (app) and HCP (dashboard) | Arm 1: Maintenance use data supplied to<br>Participant and HCP | Arm 1 | 1 |
| 2 | Х | | | | 2 | Data on Maintenance use supplied to Participant (app) | Arm 2: Maintenance use data supplied to<br>Participant | Arm 2 | 2 |
| 3 | Х | Х | Х | Х | 3 | Data on Maintenance and Rescue use supplied to Participant (app) and HCP (dashboard) | Arm 3: Maintenance and Rescue use data supplied to Participant and HCP | Arm 3 | 3 |
| 4 | Х | | Х | | 4 | Data on Maintenance and Rescue use supplied to Participant (app) | Arm 4: Maintenance and Rescue use data supplied to Participant | Arm 4 | 4 |
| 5 | | | | | 5 | No data supplied to Participant or HCP | Arm 5: No data supplied to Participant or HCP | Arm 5 | 5 |

Arm 1: Maintenance use data supplied to Participant and HCP, Arm 2: Maintenance use data supplied to Participant, Arm 3: Maintenance and Rescue use data supplied to Participant and HCP, Arm 4: Maintenance and Rescue use data supplied to Participant, Arm 5: No data supplied to Participant or HCP.

All participants will have sensors attached to both their Relvar/Breo ELLIPTA and Salbutamol (albuterol) MDI. It is the type of data provided by the CIS (either Relvar/Breo ELLIPTA alone or Relvar/Breo ELLIPTA and salbutamol MDI), as well as who sees that data (participant alone or participant and HCP) that defines the treatment arms. See Section 5.1 Study Treatment & Sub-group Display Descriptors for a description of what data is fed back to whom for each treatment arm, and the treatment group descriptors.

Where possible the full description will be used in data displays. If it is necessary to use the short description, for example in figure legends, the footnote shown under the table in Section 5.1 Study Treatment & Sub-group Display Descriptors will be included. Where treatment comparisons are included in a data display and the full treatment descriptions do not also appear within the display, the same footnote will be included.

#### 5.2. Baseline Definitions

Baseline adherence will be the percentage of ELLIPTA doses taken (daily adherence) during the last 28 days of the run-in period prior to randomisation. This will be determined using the randomisation date. A minimum of 14 run-in days prior to randomisation will be required to determine baseline adherence otherwise it will be set to missing. Any missing intermittent daily adherence data will be imputed as non-adherent i.e. the participant will be assumed to have not taken their treatment within the 24-hour time period/window, where there is no evidence of a medical device incident having occurred. Missing data due to a medical device incident such as,

- device failure
- technical failure of the ELLIPTA maintenance sensor
- data transmission failure,

will be assumed to be missing at random (MAR). For each participant the baseline percentage adherence measure will be calculated as the number of days a participant is adherent divided by the number of days without medical device incident within the baseline assessment period \* 100. See Section 10.2.2 Definitions of Assessment Windows for Adherence and Rescue Medication Use Analyses, for the definition of the baseline assessment period.

Baseline rescue free days will be the percentage rescue free days (RFDs) during the last 28 days of the run-in period prior to randomisation. This baseline will be determined in the same manner as the adherence baseline.

Where baseline assessments are determined from the randomisation visit, no unscheduled assessments will be considered as the baseline value.

Where baseline assessments are determined from the screening visit, Visit 1 will be used and no unscheduled screening visits will be considered as the baseline value.

If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

| Parameter | Study Asses | sments Consid | | |
|---|---|---|---|---|
| Visit 1 Study Days<br>Screening -28 to -1 | | Randomisation<br>Visit, Study Day<br>1 (Pre-Dose) | Baseline Used in Data<br>Display | |
| Efficacy | | | | |
| ELLIPTA Adherence<br>Endpoints (%) | | Х | | % adherence from Day -28<br>to Day -1 |
| Rescue Free Days (RFDs) (%) | | Х | | % RFDs from Day -28 to<br>Day -1 |
| Total Rescue Use (TRU) (puffs) | | Х | | Total use from Day -28 to<br>Day -1 |
| ACT Total score | | | Х | Randomisation |
| SGRQ Total score | | | Х | Randomisation |
| ASUI Total score | | | Х | Randomisation |
| PAM-13 Total score | Х | | | Screening |
| BMQ Total score | Х | | | Screening |
| MARS-A Total score | Х | | | Screening |
| PEF (litres/minute) | | | Х | Randomisation - use maximum value at visit |
| FeNO (parts per billion) | | | Х | Randomisation - use maximum value at visit |

#### Notes:

- Day 1 is referenced as Day 0 (Randomisation visit at either Visit 2 or 3 or 4) in Section 2.3 and Section 10.1
   Appendix 1: Schedule of Activities but will be reported as Day 1 per Clinical Data Interchange Standards Consortium (CDISC) reporting guidelines.
- Unless otherwise stated, if the baseline for an endpoint is missing it will not be imputed using a different timepoint
  or derivation but will remain missing.

## 5.3. Multicentre Studies

It is likely that many centres will enrol very small number of participants. Consequently, all centres within the same country will be pooled. In addition, if there are any countries enrolling very small numbers in total (<12 in the Intent to Treat population), these countries will be pooled with another country within a similar geographical region. All amalgamations will be finalised and documented prior to unblinding the treatment arm codes. These amalgamations will be used wherever region is incorporated into an analysis or summary.

In this multicentre global study, enrolment will be presented by centre, country and region (if required).

## 5.4. Examination of Covariates, Other Strata and Subgroups

#### 5.4.1. Covariates and Other Strata

Unless otherwise stated, all models used for adherence and rescue free days will allow for fixed effects due to randomised treatment arm, baseline (of the analysis variable), duration of run-in (visits), country, gender, and age (years - determined from screening date). Randomised treatment arm, duration of run-in, country, and gender will be included as categorical covariates; baseline and age will be included as continuous covariates.

The covariates to be considered in the patient reported outcomes (PRO) analyses include randomised treatment arm, age (years - determined from screening date), gender, country and baseline (of the analysis variable), if relevant.

The covariate region will replace country should amalgamation of countries, as described in Section 5.3 Multicentre Studies, be required.

The list of covariates and other strata may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses.

## 5.4.2. Examination of Subgroups

The following outcomes will be summarized by randomised treatment arm within subgroups defined by country.

- Enrollment
- Demographic characteristics
- Ellipta adherence

For these summaries, subgroups will be defined as in Table 2.

Table 2

| Category | Subgroups |
|---|---|
| Country | US, Canada, Germany, Italy, Netherlands, Spain, UK |
| Baseline ACT total score | • <=15, 16 - 19 |
| Age (years – as determine from screening date) | • 18-35, 36-48, 49-58, >58 years |

Notes: Details of the planned summaries are presented in Section 10.8 Appendix 8: List of Data Displays

## 5.5. Multiple Comparisons and Multiplicity

No adjustments for multiplicity will be applied.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 10.1 | Appendix 1: Schedule of Activities |
| 10.2 | Appendix 2: Assessment Windows |
| 10.3 | Appendix 3: Study Phases and Treatment Emergent Adverse Events |
| 10.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 10.5 | Appendix 5: Derived and Transformed Data |
| 10.6 | Appendix 6: Reporting Standards for Missing Data |
| 10.7 | Appendix 7: Abbreviations & Trade Marks |
| 10.8 | Appendix 8: List of Data Displays |

#### 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Study Population Analyses

Study population summaries will be based on the ITT population, unless otherwise specified.

Study population displays including summaries and lists of study populations, screening and run-in status, participant study and study drug disposition, participant enrolment, inclusion and exclusion and important protocol deviations, demographic, age, race and baseline characteristics (including height, weight and BMI), medical conditions, family and smoking history and prior and concomitant medications will be based on GSK Core Data Standards. Details of the planned displays are presented in Section 10.8 Appendix 8: List of Data Displays.

Concomitant medications will be coded using the GSK Drug coding dictionary. Summaries of the number and percentage of participants taking concomitant medications will be displayed by ingredient without regard to Anatomical Therapeutical Chemical (ATC) classifications. These summaries will include single-ingredient medications and will present multi-ingredient medications according to the combination of the component ingredients. Summaries will be split into asthma and non-asthma concomitant medications, as well as into those taken pre-screening, during run-in, whilst on-treatment and post-treatment (as described in Section 10.3.1 Study Phases).

Asthma maintenance concomitant medications taken by participants in the 12 months prior to screening (pre-screening) will also be summarised as well as those used to treat severe exacerbations experienced whilst on study.

## 6.2. Supplementary Information for Study Population Displays

#### 6.2.1. Disease and Baseline Characteristics

Summary of attendance at each scheduled clinic visit will be presented.

Summaries and lists of the Relvar/Breo ELLIPTA and Salbutamol MDI sensor statuses as well as the App status during the study will be presented.

Asthma exacerbation history (12-month history) at screening will be summarised with frequency distributions of the number of exacerbations treated with oral/systemic corticosteroids not involving hospitalization; the number of exacerbations treated without oral/systemic corticosteroids not involving hospitalization; the number of exacerbations requiring hospitalization; and the total number of exacerbations (i.e., those not involving hospitalization and those involving hospitalization).

Asthma duration will also be summarised.

The screening and baseline lung function test and exhaled nitric oxide summaries will include screening (Visit 1) pre-bronchodilator and pre-ICS/LABA, PEF (in litres per minute (L/min)) and FeNO (millilitres per second (mL/sec)). Baseline PEF (L/min) and

FeNO (mL/sec) measured at Randomisation (Visit 2/3/4) will also be summarised. Additionally, screening and baseline PEF will be summarised by country.

Prescription details (12-month history) at screening will be summarised with frequency distributions of the number of asthma maintenance therapy prescriptions requested or prescribed; the number of asthma maintenance therapy requested or prescribed that would need to be 100% compliant. Compliance in the previous 12 months will be calculated as 100 \* (Actual number of prescriptions) / (Number of prescriptions needed to be 100% compliant) and summarised. These data will also be listed.

## 6.2.2. Preferred Time of Dosing

Summary statistics to summarise percentage of total ELLIPTA doses taken at preferred time of dosing for each participant will be presented. A participant is considered as having taken their dose at their preferred time if the actual time of the ELLIPTA dose is recorded  $\pm 1$  hour of their preferred time as captured on the eCRF at screening. A histogram of individual dose deviations (in minutes) from preferred time will also be presented per treatment group. These data will also be listed.

## 6.2.3. Study Medication Exposure and Compliance

Duration (days) of exposure to study medication will be calculated based on randomisation date and latest (stop) of all dates recorded for the participant. Duration will be summarised categorically and with descriptive statistics. Total years exposed to Relvar/Breo after randomisation will also be presented. Further details are presented in Section 10.5 Appendix 5: Derived and Transformed Data

Calculation of Relvar/Breo study medication compliance after randomisation, will be based on the ELLIPTA device dose counter (which displays the number of doses remaining) as described in Section 10.5 Appendix 5: Derived and Transformed Data. Treatment compliance (calculated as a percentage) will be summarised categorically and with descriptive statistics.

All exposure and compliance data will be listed.

A summary of the number of puffs per day as recorded by the ELLIPTA Relvar/Breo and MDI sensors will be summarised and graphically presented.

#### 6.2.4. HCP dashboard review

The actions taken by the HCP post the dashboard data review will be summarized and listed by visit for Arms 1 and 3.

## 7. EFFICACY ANALYSES

## 7.1. Primary Efficacy Analysis

The primary analysis will estimate the treatment arm effect of 6 months use of the Relvar/Breo ELLIPTA maintenance therapy with CIS when both the participant and the HCP are supplied with data from the ELLITPA sensor versus no data supplied to the participant and HCP (Arm 1 vs Arm 5).

#### 7.1.1. Endpoint

The primary endpoint is the percentage of ELLIPTA doses taken (daily adherence) between the beginning of Month 4 and the end of Month 6 as determined by the maintenance sensor. Daily adherence is defined as the participant taking one dose of Relvar/Breo ELLIPTA, within a 24-hour period, starting at 12.00am each day of the runin and treatment period.

## 7.1.2. Summary Measure

The mean difference in daily adherence between Arm 1 and Arm 5 will be estimated from an Analysis of Covariance (ANCOVA) model allowing for effects due to randomised treatment arm, baseline adherence, duration of run-in (visits), country, gender, and age (years).

## 7.1.3. Population of Interest

The primary efficacy analysis will be based on the Intent-To-Treat population.

## 7.1.4. Strategy for Intercurrent (Post-Randomisation) Events

The following steps in Table 3 will be applied sequentially when deriving the primary endpoint. See Section 10.5.3.1 ELLIPTA Device Sensor Assessments for full details of the missing data imputations process.

Table 3

| Intercurrent Event Estimation Rules (to be applied sequentially) | Intercurrent Event (IE) | Strategy with Rationale | Estimation Method following IE |
|---|---|---|---|
| 1 | None (completed as randomised) | Treatment policy: | Data are available; no imputation required |
| | Without discontinuation of CIS feedback or ELLIPTA maintenance sensor • Premature discontinuation from rescue/salbutamol MDI sensor • Change of dose of ELLIPTA Discontinuation of CIS feedback, but not ELLIPTA maintenance sensor • Premature discontinuation from | Directly assessed using observed adherence data while ELLIPTA maintenance sensor is in use, regardless of whether the CIS feedback is discontinued. | |
| | App and/or HCP interaction | | |
| 2 | Discontinuation of ELLIPTA maintenance sensor only | Treatment policy: Without the ELLIPTA maintenance sensor, no | Jump to Reference (J2R) Imputation |
| | | CIS feedback is possible, assume • participants continue to take ELLIPTA as | |

| Intercurrent Event Estimation Rules (to be applied sequentially) | Intercurrent Event (IE) | Strategy with Rationale | Estimation Method following IE |
|---|---|---|---|
| | | <ul> <li>they would have without the CIS intervention</li> <li>adherence will be like that in the control (no CIS feedback) group</li> </ul> | |
| 3 | Discontinuation of ELLIPTA | Whilst on treatment: ELLIPTA adherence is only a relevant measure while ELLIPTA treatment is appropriate. It is assumed that ELLIPTA treatment is no longer appropriate if the participant discontinues ELLIPTA but remains in the study or withdraws for a reason related to ELLIPTA. | Follow-up after ELLIPTA discontinuation is excluded, i.e. no data; adherence is weighted by proportion of months 4 to 6 for which data is included* |
| 4 | Premature withdrawal from the study, not related to ELLIPTA discontinuation or CIS, and concurrent with discontinuation of the ELLIPTA maintenance sensor | Hypothetical: When study withdrawal is unrelated to ELLIPTA or the CIS then reasonable to assume that participant would have continued with ELLIPTA and their CIS intervention, had the unrelated event not occurred | Missing at Random (MAR) Imputation |

<sup>\*</sup> Discontinuation of ELLIPTA prior to the start of month 4 will lead to a participant being excluded from the primary analysis

## 7.1.4.1. Events prior to premature discontinuation of the ELLIPTA maintenance sensor

The treatment policy estimand is directly assessed using the observed adherence data while the ELLIPTA maintenance sensor is in use, regardless of whether the CIS feedback is discontinued.

Any missing intermittent adherence data will be imputed as non-adherent i.e. the participant will be assumed to have not taken their treatment within the 24-hour time period/window, where there is no evidence of device or technical/transmission failure.

Missing intermittent adherence data due to a medical device incident such as device failure, technical failure of the sensor, or data transmission failure will be assumed to be missing at random (MAR). For each participant, the percentage adherence measure will be calculated from the proportion of the number of days a participant is adherent divided by the number of days data provided in that month.

## 7.1.4.2. Events following premature discontinuation of the ELLIPTA maintenance sensor

It is assumed that participants would continue to take ELLIPTA as they would have without the CIS intervention (J2R imputation) following discontinuation of the ELLIPTA maintenance sensor.

It is assumed that ELLIPTA treatment is no longer appropriate if the participant discontinues ELLIPTA but remains in the study or withdraws for a reason related to ELLIPTA. The ELLIPTA adherence endpoint is no longer considered relevant and subsequent follow-up is excluded from the analysis, with participants weighted in the analysis by the proportion of months 4 to 6 for which data is included.

It is assumed that participants would continue to take ELLIPTA as they would have with their allocated CIS intervention (MAR imputation) following concurrent discontinuation of the ELLIPTA maintenance sensor and withdrawal unrelated to ELLIPTA or CIS.

See Section 10.5.3.1 ELLIPTA Device Sensor Assessments for further derivation details.

#### 7.1.5. Statistical Analyses / Methods

Details of the planned displays will be provided in Section 10.8, Appendix 8: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints /variables defined in Section 7.1.1, Endpoint will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 7.1.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

The primary endpoint is the percentage of ELLIPTA doses taken (daily adherence) between the beginning of Month 4 and the end of Month 6 as determined by the maintenance sensor. Daily adherence is defined as the participant taking one dose of Relvar/Breo ELLIPTA within a 24 hour period, starting at 12.00am each day of treatment period.

#### **Multiple Imputation Specification**

Imputation will be carried out using monthly adherence rates for months 1 to 6. 1000 draws will be used. For each draw, four intermediate imputation datasets will be created to allow for the handling of fully unobserved months (using set A imputations) and partially unobserved months (using set B imputations).

- Set A where the partially observed month is directly estimated under the MAR assumption as the
  proportion of the number of days a participant is adherent divided by the number of days data
  provided in that month.
  - J2R imputations
  - MAR imputations
- Set B where the partially observed month is set to missing.
  - J2R imputations
  - MAR imputations

The timing of the intercurrent events of discontinuation of the ELLIPTA maintenance sensor, discontinuation of ELLIPTA and withdrawal from study will be used to identify the proportion of each month to be assigned as observed data, J2R imputed data, MAR imputed data, or no data. The strategy for handling intercurrent events is described in Section 7.1.4 Strategy for Intercurrent (Post-Randomisation) Events.

Within each imputation draw, for each month, the observed and any imputed data will be combined to provide a percentage adherence value. The values for months 4 to 6 will be combined to create the value for the primary analysis and the weight to be assigned to each participant.

Multiple imputation using Rubin's rules will be used to estimate the treatment effect and associated standard error, by performing the ANCOVA analysis described below on the primary endpoint within each dataset.

The multiple imputation will be implemented using the methods described in Carpenter, 2013, using the macros available from https://missingdata.lshtm.ac.uk/2017/04/06/gsk-five-macros/..

#### **Model Specification**

The analysis will be performed on the percentage adherence between Months 4 and 6 using an Analysis of Covariance (ANCOVA) model allowing for effects due to randomised treatment arm, baseline adherence, duration of run-in (visits), country, gender, and age (years).

Baseline adherence will be the percentage ELLIPTA doses taken (daily adherence) during the last 28 days of the run-in period prior to randomisation. Randomised treatment arm, duration of run-in (visits), country, and gender will be included as categorical covariates; baseline adherence and age (years) will be included as continuous covariates.

Each participant will be weighted by the proportion of months 4 to 6 for which data is included in the percentage adherence endpoint (both observed and imputed data are accounted for in the weighting).

Data from all 5 treatment arms will be included in the model and used to estimate the difference between Arm 1 and Arm 5 for the primary objective.

#### **Model Checking & Diagnostics**

Normality assumptions underlying the ANCOVA model used for analysis will be examined in a limited number of imputed datasets by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.

If there are any departures from the distributional assumptions, alternative models may be explored using appropriately transformed data.

Interactions with treatment will be explored for other model covariates and tests for interactions will be at the 2-sided 10% significance level. Any significant interactions that are found will be thoroughly investigated and where necessary, extra outputs will be produced.

#### Model Results Presentation

Summary statistics (n, mean, standard deviation, median, minimum, maximum) of the primary endpoint will be provided, based on the observed percentages.

The adjusted means for each treatment and the estimated treatment difference for the primary treatment comparison of Arm 1 versus Arm 5 will be presented together with a 95% confidence interval for the difference and corresponding Wald test statistic and p-value from the multiple imputation procedure.

#### Subgroup Analyses

For the analysis by baseline total ACT score (<=15, 16-19), the model will additionally include the baseline ACT total score category and randomised treatment arm-by-baseline ACT total score category interaction as covariates.

For the analysis by age group (18-35, 36-48, 49-58, >58 years), the model will additionally include age group and randomised treatment arm-by-age group interaction as covariates.

The adjusted means for each treatment and the estimated treatment difference for the treatment comparisons of Arm 2 versus Arm 5, Arm 3 versus Arm 5 and Arm 4 versus Arm 5 will be presented together with the 95% confidence interval for the differences and corresponding p-values from the multiple imputation procedure.

#### **Sensitivity Analysis**

 A sensitivity analysis will be performed estimating the treatment effect by utilizing a generalized linear model (GLM) and not running the multiple imputation process. The model will follow a binomial distribution with the logit link function. The covariates included in the GLM will be the same as those included in the primary analysis. Model assumptions will be checked using standardised residual plots, and model results presentation will be the same as described for the primary analysis. Missing data will be assumed to be MAR.

## 7.2. Secondary Efficacy Analyses

The secondary analysis of daily adherence during month 4 to 6 will estimate the treatment effect of 6 months use of the ELLIPTA maintenance therapy with CIS for the following aspects of the CIS:

- Maintenance data only supplied to participants versus no data supplied to the participant (Arm 2 vs Arm 5)
- Rescue and Maintenance data supplied to participant and HCP versus no data supplied to the participant and HCP (Arm 3 vs Arm 5)
- Rescue and Maintenance data only supplied to participant versus no data supplied to the participant (Arm 4 vs Arm 5)

In addition, secondary analyses of daily adherence during month 1 to 6 and month 1 to 3 will estimate the treatment effect of 6 months use of the ELLIPTA maintenance therapy with CIS when the participant and the HCP are supplied with data from maintenance and rescue sensors versus no data supplied to participant and HCP (Arm 1, 2, 3, 4 vs Arm 5).

Secondary analysis to evaluate the effect of 6 months use of the CIS on a participant's rescue medication usage will be conducted, as well as an evaluation of the effect of 6 months use with the CIS on participant's asthma control.

## 7.2.1. ELLIPTA Adherence Measure Endpoints

The adherence secondary endpoints are:

- The percentage of ELLIPTA doses taken (daily adherence) between the beginning of Month 4 and the end of Month 6 as determined by the maintenance sensor. Daily adherence is defined as the participant taking one dose of Relvar/Breo ELLIPTA, within a 24-hour period, starting at 12.00am each day of the run-in and treatment period.
- The percentage of ELLIPTA doses taken (daily adherence) between the beginning of Month 1 and the end of Month 6 as determined by the maintenance sensor. Daily adherence is defined as the participant taking one dose of Relvar/Breo ELLIPTA, within a 24-hour period, starting at 12.00am each day of the run-in and treatment period.
- The percentage of ELLIPTA doses taken (daily adherence) between the beginning of Month 1 and the end of Month 3 as determined by the maintenance sensor. Daily adherence is defined as the participant taking one dose of Relvar/Breo ELLIPTA, within a 24-hour period, starting at 12.00am each day of the run-in and treatment period.

#### 7.2.1.1. Summary Measure

The mean difference in daily adherence between the comparisons of interest will be estimated from an Analysis of Covariance (ANCOVA) model allowing for effects due to randomised treatment, baseline adherence, duration of run-in (visits), country, gender, and age (years).

#### 7.2.1.2. Population of Interest

The secondary efficacy analyses will be based on the Intent-To-Treat population.

## 7.2.1.3. Strategy for Intercurrent (Post-Randomisation) Events

The steps detailed in Section 7.1.4 Strategy for Intercurrent (Post-Randomisation) Events will be applied sequentially when deriving the secondary adherence endpoints.

## 7.2.1.3.1. Events prior to premature discontinuation of the ELLIPTA maintenance sensor

The treatment policy estimand is directly assessed using the observed adherence data while the ELLIPTA maintenance sensor is in use, regardless of whether the CIS feedback is discontinued.

Any missing intermittent adherence data will be imputed as non-adherent i.e. the participant will be assumed to have not taken their treatment within the 24-hour time period/window, where there is no evidence of device or technical/transmission failure.

Missing intermittent adherence data due to a medical device incident such as device failure, technical failure of the sensor, or data transmission failure will be assumed to be missing at random (MAR). For each participant, the percentage adherence measure will be calculated from the proportion of the number of days a participant is adherent divided by the number of days data provided in that month.

## 7.2.1.3.2. Events following premature discontinuation of the ELLIPTA maintenance sensor

It is assumed that participants would continue to take ELLIPTA as they would have without the CIS intervention (J2R imputation) following discontinuation of the ELLIPTA maintenance sensor.

It is assumed that ELLIPTA treatment is no longer appropriate if the participant discontinues ELLIPTA but remains in the study or withdraws for a reason related to ELLIPTA. The ELLIPTA adherence endpoint is no longer considered relevant and subsequent follow-up is excluded from the analysis, with participants weighted in the analysis by the proportion of months 4 to 6 for which data is included.

It is assumed that participants would continue to take ELLIPTA as they would have with their allocated CIS intervention (MAR imputation) following concurrent discontinuation of the ELLIPTA maintenance sensor and withdrawal unrelated to ELLIPTA or CIS.

See Section 10.5.3.1 ELLIPTA Device Sensor Assessments further derivation details.

#### 7.2.1.4. Statistical Analyses / Methods

Details of the planned displays will be provided in Section 10.8, Appendix 8: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints /variables defined in Section 7.1.1, Endpoint will be summarised using descriptive statistics, graphically presented (where appropriate) and listed

## 7.2.1.5. Statistical Analyses / Methodology Specification

## 7.2.1.5.1. The percentage of ELLIPTA doses taken (daily adherence) between the beginning of Month 4 and the end of Month 6

#### **Endpoint / Variables**

Percentage of ELLIPTA doses taken (daily adherence) between the beginning of Month 4 and the end of Month 6 as determined by the maintenance sensor for the following treatment arm comparisons:

- Arm 2 vs Arm 5
- Arm 3 vs Arm 5
- Arm 4 vs Arm 5

Daily adherence is defined as the participant taking one dose of Relvar/Breo ELLIPTA within a 24-hour period, starting at 12.00am each day of treatment period.

#### **Multiple Imputation Specification**

Imputation will be carried out using monthly adherence rates for months 1 to 6. 1000 draws will be used. For each draw, four intermediate imputation datasets will be created to allow for the handling of fully unobserved months (using set A imputations) and partially unobserved months (using set B imputations).

- Set A where the partially observed month is directly estimated under the MAR assumption as the proportion of the number of days a participant is adherent divided by the number of days data provided in that month.
  - J2R imputations
  - MAR imputations
- Set B where the partially observed month is set to missing.
  - J2R imputations
  - MAR imputations

The timing of the intercurrent events of discontinuation of the ELLIPTA maintenance sensor, discontinuation of ELLIPTA and withdrawal from study will be used to identify the proportion of each month to be assigned as observed data, J2R imputed data, MAR imputed data, or no data. The strategy for handling intercurrent events is described in Section 7.1.4 Strategy for Intercurrent (Post-Randomisation) Events.

Within each imputation draw, for each month, the observed and any imputed data will be combined to provide a percentage adherence value. The values for months 4 to 6 will be combined to create the value for the secondary analysis and the weight to be assigned to each participant.

Multiple imputation using Rubin's rules will be used to estimate the treatment effect and associated standard error, by performing the ANCOVA analysis described below on the secondary endpoint within each dataset.

The multiple imputation will be implemented using the methods described in Carpenter, 2013, using the macros available from <a href="https://missingdata.lshtm.ac.uk/2017/04/06/gsk-five-macros/">https://missingdata.lshtm.ac.uk/2017/04/06/gsk-five-macros/</a>.

#### **Model Specification**

The analysis will be performed on the percentage adherence between Months 4 and 6 using an Analysis of Covariance (ANCOVA) model allowing for effects due to randomised treatment arm, baseline adherence, duration of run-in (visits), country, gender, and age (years).

Baseline adherence will be the percentage ELLIPTA doses taken (daily adherence) during the last 28 days of the run-in period prior to randomisation. Randomised treatment, duration of run-in (visits), country, and gender will be included as categorical covariates; baseline adherence and age (years) will be included as continuous covariates.

Each participant will be weighted by the proportion of months 4 to 6 for which data is included in the percentage adherence endpoint (both observed and imputed data are accounted for in the weighting).

Data from all 5 treatment arms will be included in the model, and used to estimate the difference between:

- Arm 2 and Arm 5
- Arm 3 and Arm 5
- Arm 4 and Arm 5

#### **Model Checking & Diagnostics**

Normality assumptions underlying the ANCOVA model used for analysis will be examined in a limited number of imputed datasets by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.

If there are any departures from the distributional assumptions, alternative models may be explored using appropriately transformed data.

Interactions with treatment will be explored for other model covariates and tests for interactions will be at the 2-sided 10% significance level. Any significant interactions that are found will be thoroughly investigated and where necessary, extra outputs will be produced.

#### **Model Results Presentation**

Summary statistics (mean, standard deviation, median, minimum, maximum) of the primary endpoint will be provided, based on the observed percentages.

The adjusted means for each treatment and the estimated treatment difference for the treatment comparisons of Arm 2 versus Arm 5, Arm 3 versus Arm 5 and Arm 4 versus Arm 5 will be presented together with the 95% confidence interval for the differences and corresponding p-values from the multiple imputation procedure.

#### Subgroup Analyses

For the analysis by baseline total ACT score (<=15, 16-19), the model will additionally include the baseline ACT total score category and randomised treatment arm-by-baseline ACT total score category interaction as covariates.

For the analysis by age group (18-35, 36-48, 49-58, >58 years), the model will additionally include age group and randomised treatment arm-by-age group interaction as covariates.

The adjusted means for each treatment and the estimated treatment difference for the treatment comparisons of Arm 2 versus Arm 5, Arm 3 versus Arm 5 and Arm 4 versus Arm 5 will be presented together with the 95% confidence interval for the differences and corresponding p-values from the multiple imputation procedure.

#### Sensitivity Analysis

 A sensitivity analysis will be performed estimating the treatment effect by utilizing a generalized linear model (GLM) and not running the multiple imputation process. The model will follow a binomial distribution with the logit link function. The covariates included in the GLM will be the same as those included in the primary analysis. Model assumptions will be checked using standardised residual plots, and model results presentation will be the same as described for the primary analysis. Missing data will be assumed to be MAR.

## 7.2.1.5.2. The percentage of ELLIPTA doses taken (daily adherence) between the beginning of Month 1 and the end of Month 6

#### **Endpoint / Variables**

Percentage of ELLIPTA doses taken (daily adherence) between the beginning of Month 1 and the end of Month 6 as determined by the maintenance sensor for the following treatment arm comparisons:

- Arm 1 vs Arm 5
- Arm 2 vs Arm 5
- Arm 3 vs Arm 5
- Arm 4 vs Arm 5

Daily adherence is defined as the participant taking one dose of Relvar/Breo ELLIPTA within a 24-hour period, starting at 12.00am each day of treatment period.

#### **Multiple Imputation Specification**

Imputation will be carried out using monthly adherence rates for months 1 to 6. 1000 draws will be used. For each draw, four intermediate imputation datasets will be created to allow for the handling of fully unobserved months (using set A imputations) and partially unobserved months (using set B imputations).

- Set A where the partially observed month is directly estimated under the MAR assumption as the
  proportion of the number of days a participant is adherent divided by the number of days data
  provided in that month.
  - J2R imputations
  - MAR imputations
- Set B where the partially observed month is set to missing.
  - J2R imputations
  - MAR imputations

The timing of the intercurrent events of discontinuation of the ELLIPTA maintenance sensor, discontinuation of ELLIPTA and withdrawal from study will be used to identify the proportion of each month to be assigned as observed data, J2R imputed data, MAR imputed data, or no data. The strategy for handling intercurrent

events is described in Section 7.1.4 Strategy for Intercurrent (Post-Randomisation) Events.

Within each imputation draw, for each month, the observed and any imputed data will be combined to provide a percentage adherence value. The values for months 4 to 6 will be combined to create the value for the primary analysis and the weight to be assigned to each participant.

Multiple imputation using Rubin's rules will be used to estimate the treatment effect and associated standard error, by performing the ANCOVA analysis described below on the primary endpoint within each dataset.

The multiple imputation will be implemented using the methods described in Carpenter, 2013, using the macros available from <a href="https://missingdata.lshtm.ac.uk/2017/04/06/gsk-five-macros/">https://missingdata.lshtm.ac.uk/2017/04/06/gsk-five-macros/</a>.

### **Model Specification**

The analysis will be performed on the percentage adherence between Months 1 and 6 using an Analysis of Covariance (ANCOVA) model allowing for effects due to randomised treatment arm, baseline adherence, duration of run-in (visits), country, gender, and age (years).

Baseline adherence will be the percentage ELLIPTA doses taken (daily adherence) during the last 28 days of the run-in period prior to randomisation. Randomised treatment, duration of run-in (visits), country, and gender will be included as categorical covariates; baseline adherence and age (years) will be included as continuous covariates.

Each participant will be weighted by the proportion of months 1 to 6 for which data is included in the percentage adherence endpoint (both observed and imputed data are accounted for in the weighting).

Data from all 5 treatment arms will be included in the model, and used to estimate the difference between:

- Arm 1 and Arm 5
- Arm 2 and Arm 5
- Arm 3 and Arm 5
- Arm 4 and Arm 5

#### **Model Checking & Diagnostics**

Normality assumptions underlying the ANCOVA model used for analysis will be examined in a limited number of imputed datasets by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.

If there are any departures from the distributional assumptions, alternative models may be explored using appropriately transformed data.

Interactions with treatment will be explored for other model covariates and tests for interactions will be at the 2-sided 10% significance level. Any significant interactions that are found will be thoroughly investigated and where necessary, extra outputs will be produced.

#### **Model Results Presentation**

Summary statistics (n, mean, standard deviation, median, minimum, maximum) of the primary endpoint will be provided, based on the observed percentages.
The adjusted means for each treatment arm and the estimated treatment arm difference for the treatment comparisons of Arm 1 versus Arm 5, Arm 2 versus Arm 5, Arm 3 versus Arm 5 and Arm 4 versus Arm 5 will be presented together with the 95% confidence interval for the differences and corresponding p-values from the multiple imputation procedure.

### **Sensitivity Analysis**

A sensitivity analysis will be performed estimating the treatment effect by utilizing a generalized linear
model (GLM) and not running the multiple imputation process. The model will follow a binomial
distribution with the logit link function. The covariates included in the GLM will be the same as those
included in the primary analysis. Model assumptions will be checked by using standardised residual
plots, and the model results presentation will be the same as described for the primary analysis.
Missing data will be assumed to be MAR.

# 7.2.1.5.3. The percentage of ELLIPTA doses taken (daily adherence) between the beginning of Month 1 and the end of Month 3

#### **Endpoint / Variables**

Percentage of ELLIPTA doses taken (daily adherence) between the beginning of Month 1 and the end of Month 3 as determined by the maintenance sensor for the following treatment arm comparisons:

- Arm 1 vs Arm 5
- Arm 2 vs Arm 5
- Arm 3 vs Arm 5
- Arm 4 vs Arm 5

Daily adherence is defined as the participant taking one dose of Relvar/Breo ELLIPTA within a 24-hour period, starting at 12.00am each day of treatment period.

#### Multiple Imputation Specification

Imputation will be carried out using monthly adherence rates for months 1 to 6. 1000 draws will be used. For each draw, four intermediate imputation datasets will be created to allow for the handling of fully unobserved months (using set A imputations) and partially unobserved months (using set B imputations).

- Set A where the partially observed month is directly estimated under the MAR assumption as the
  proportion of the number of days a participant is adherent divided by the number of days data
  provided in that month.
  - J2R imputations
  - MAR imputations
- Set B where the partially observed month is set to missing.
  - J2R imputations
  - MAR imputations

The timing of the intercurrent events of discontinuation of the ELLIPTA maintenance sensor, discontinuation of ELLIPTA and withdrawal from study will be used to identify the proportion of each month to be assigned as observed data, J2R imputed data, MAR imputed data, or no data. The strategy for handling intercurrent

events is described in Section 7.1.4 Strategy for Intercurrent (Post-Randomisation) Events.

Within each imputation draw, for each month, the observed and any imputed data will be combined to provide a percentage adherence value. The values for months 4 to 6 will be combined to create the value for the primary analysis and the weight to be assigned to each participant.

Multiple imputation using Rubin's rules will be used to estimate the treatment effect and associated standard error, by performing the ANCOVA analysis described below on the primary endpoint within each dataset.

The multiple imputation will be implemented using the methods described in Carpenter, 2013, using the macros available from <a href="https://missingdata.lshtm.ac.uk/2017/04/06/gsk-five-macros/">https://missingdata.lshtm.ac.uk/2017/04/06/gsk-five-macros/</a>.

# **Model Specification**

The analysis will be performed on the percentage adherence between Months 1 and 3 using an Analysis of Covariance (ANCOVA) model allowing for effects due to randomised treatment arm, baseline adherence, duration of run-in (visits), country, gender, and age (years).

Baseline adherence will be the percentage ELLIPTA doses taken (daily adherence) during the last 28 days of the run-in period prior to randomisation. Randomised treatment arm, duration of run-in (visits), country, and gender will be included as categorical covariates; baseline adherence and age (years) will be included as continuous covariates.

Each participant will be weighted by the proportion of months 1 to 3 for which data is included in the percentage adherence endpoint (both observed and imputed data are accounted for in the weighting).

Data from all 5 treatment arms will be included in the model, and used to estimate the difference between:

- Arm 1 and Arm 5
- Arm 2 and Arm 5
- Arm 3 and Arm 5
- Arm 4 and Arm 5

#### **Model Checking & Diagnostics**

Normality assumptions underlying the ANCOVA model used for analysis will be examined in a limited number of imputed datasets by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.

If there are any departures from the distributional assumptions, alternative models may be explored using appropriately transformed data.

Interactions with treatment will be explored for other model covariates and tests for interactions will be at the 2-sided 10% significance level. Any significant interactions that are found will be thoroughly investigated and where necessary, extra outputs will be produced.

#### Model Results Presentation

Summary statistics (n, mean, standard deviation, median, minimum, maximum) of the primary endpoint will be provided, based on the observed percentages.

The adjusted means for each treatment and the estimated treatment difference for the treatment comparisons of Arm 1 versus Arm 5, Arm 2 versus Arm 5, Arm 3 versus Arm 5 and Arm 4 versus Arm 5 will be presented together with the 95% confidence interval for the differences and corresponding p-values from the multiple imputation procedure.

#### Sensitivity Analysis

A sensitivity analysis will be performed estimating the treatment effect by utilizing a generalized linear
model (GLM) and not running the multiple imputation process. The model will follow a binomial
distribution with the logit link function. The covariates included in the GLM will be the same as those
included in the primary analysis. Model assumptions will be checked by using standardised residual
plots, and the model results presentation will be the same as described for the primary analysis.
Missing data will be assumed to be MAR.

# 7.2.2. MDI Rescue Medication Use Endpoints

- Percentage of rescue free days measured between the beginning of month 4 and the end of month 6 as determined by the MDI rescue sensor records of date, time, and number of inhaler actuations.
- Total rescue use measured between the beginning of month 4 and the end of month 6 as determined by the MDI rescue sensor records of date, time, and number of inhaler actuations.

# 7.2.2.1. Summary Measure

The rescue medicine summary measures are:

- The mean difference in percentage of rescue free days between the treatment arms will be estimated from an Analysis of Covariance (ANCOVA) model allowing for effects due to randomised treatment, baseline rescue-free, duration of run-in (visits), country, gender, and age (years).
- The mean total rescue use for the treatment arms will be summarised using summary statistics (n, mean, SD, median, min, max) for each treatment arm for each Month separately, and totalled Month 4-6.

#### 7.2.2.2. Population of Interest

These secondary efficacy analyses will be based on the Intent-To-Treat population.

# 7.2.2.3. Strategy for Intercurrent (Post-Randomisation) Events

It is assumed that salbutamol MDI rescue medication use does not permanently discontinue for asthmatic participants, regardless of whether they are used in addition to maintenance therapy or not.

The following steps in Table 4 will be applied sequentially when deriving the rescue free days endpoint. See Section 10.5.3.2 MDI Device Sensor Assessments for full details of the missing data imputations process.

Table 4

| Intercurrent Event Estimation Rules (to be applied sequentially) | Intercurrent Event (IE) | Strategy with Rationale | Estimation Method following IE |
|---|---|---|---|
| 1 | None (completed as randomised) | Treatment policy: | Data are available; no imputation required |
| | <ul> <li>Without discontinuation of CIS feedback or MDI eSensor</li> <li>Premature discontinuation from ELLIPTA eSensor</li> <li>Premature discontinuation from ELLIPTA</li> <li>Change of dose of ELLIPTA</li> </ul> | Directly assessed using observed rescue data while MDI sensor is in use, regardless of whether the CIS feedback is discontinued. | |
| | Discontinuation of CIS feedback, but not MDI eSensor • Premature discontinuation from App and/or HCP interaction | | |

| Intercurrent Event Estimation Rules (to be applied sequentially) | Intercurrent Event (IE) | Strategy with Rationale | Estimation Method following IE |
|---|---|---|---|
| 2 | Discontinuation from MDI eSensor but not the study | Hypothetical: Without the sensor, no CIS feedback is possible and so it is assumed that rescue use will be like that in the control group for those randomised to Arm 3 and 4. Since Arms 1 and 2 never have CIS feedback, without the sensor it is assumed that rescue use will continue as before. | MAR imputation (Arms 1&2)<br>J2R imputation (Arms 3&4) |
| 3 | Premature withdrawal from the study | Hypothetical: Without the sensor, no CIS feedback is possible and so it is assumed that rescue use will be like that in the control group for those randomised to Arm 3 and 4. Since Arms 1 and 2 never have CIS feedback, without the sensor it is assumed that rescue use will continue as before. | MAR imputation (Arms 1&2)<br>J2R imputation (Arms 3&4) |
| 4 | Premature withdrawal from the study<br>not related to CIS, and concurrent with<br>discontinuation of the MDI sensor | Hypothetical: When study withdrawal is unrelated to the CIS then it is reasonable to assume that the participant would have continued with MDI and the Sensor, had the unrelated event not occurred. | Missing at Random (MAR) Imputation |

# 7.2.2.3.1. Events following premature discontinuation of the MDI sensor

It is assumed that participants would continue to take MDI as they would have without the CIS intervention (jump to reference imputation) following discontinuation of the MDI sensor if receiving treatment Arms 3 and 4, otherwise continue to take MDI as they would have with their allocated CIS interventions (MAR).

It is assumed that participants would continue to take MDI as they would have with their allocated CIS interventions (MAR) following concurrent discontinuation of MDI sensor and withdrawal from study if unrelated to CIS.

# 7.2.2.4. Statistical Analyses / Methods

Details of the planned displays will be provided in Section 10.8, Appendix 8: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints /variables defined in Section 7.2.2 MDI Rescue Medication Use Endpoints, Section 7.1.1 Endpoint will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

### 7.2.2.5. Statistical Analyses / Methodology Specification

#### **Endpoint / Variables**

The percentage of rescue free days measured between the beginning of month 4 and the end of month 6 as determined by the MDI rescue sensor for the following treatment arm comparisons

#### **Multiple Imputation Specification**

Imputation will be carried out using monthly rescue free rates for months 1 to 6. 1000 draws will be used. For each draw, four intermediate imputation datasets will be created to allow for the handling of fully unobserved months (using set A imputations) and partially unobserved months (using set B imputations).

- Set A where the partially observed month is directly estimated under the MAR assumption as the
  proportion of the number of days a participant is adherent divided by the number of days data
  provided in that month.
  - J2R imputations
  - MAR imputations
- Set B where the partially observed month is set to missing.
  - J2R imputations
  - MAR imputations

The timing of the intercurrent events of discontinuation of the MDI sensor and withdrawal from study will be used to identify the proportion of each month to be assigned as observed data, J2R imputed data or MAR imputed data. The strategy for handling intercurrent events is described in Section 7.2.2.3 Strategy for Intercurrent (Post-Randomisation) Events.

Within each imputation draw, for each month, the observed and any imputed data will be combined to provide a percentage rescue free day value. The values for months 4 to 6 will be combined to create the value for the secondary analysis and the weight to be assigned to each participant.

Multiple imputation using Rubin's rules will be used to estimate the treatment effect and associated standard error, by performing the ANCOVA analysis described below on the secondary endpoint within each dataset.

The multiple imputation will be implemented using the methods described in Carpenter, 2013, using the macros available from <a href="https://missingdata.lshtm.ac.uk/2017/04/06/gsk-five-macros/">https://missingdata.lshtm.ac.uk/2017/04/06/gsk-five-macros/</a>.

#### **Model Specification**

The analysis will be performed on the percentage of rescue free days between Months 4 and 6 using an Analysis of Covariance (ANCOVA) model allowing for effects due to randomised treatment arm, baseline rescue free days percentage, duration of run-in (visits), country, gender, and age (years).

Baseline rescue free days will be the percentage rescue free days during the last 28 days of the run-in period prior to randomisation. Randomised treatment, duration of run-in (visits), country, and gender will be included as categorical covariates; baseline rescue free days percentage and age (years) will be included as continuous covariates.

Each participant will be weighted by the proportion of months 4 to 6 for which data is included in the percentage rescue free days endpoint (both observed and imputed data are accounted for in the weighting).

Data from all 5 treatment arms will be included in the model, and used to estimate the difference between:

- Arm 1 and Arm 5
- Arm 2 and Arm 5
- Arm 3 and Arm 5
- Arm 4 and Arm 5

#### **Model Checking & Diagnostics**

Normality assumptions underlying the ANCOVA model used for analysis will be examined in a limited number of imputed datasets by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.

If there are any departures from the distributional assumptions, alternative models may be explored using appropriately transformed data.

Interactions with treatment will be explored for other model covariates and tests for interactions will be at the 2-sided 10% significance level. Any significant interactions that are found will be thoroughly investigated and where necessary, extra outputs will be produced.

#### **Model Results Presentation**

Summary statistics (mean, standard deviation, median, minimum, maximum) of the primary endpoint will be provided, based on the observed percentages.

The adjusted means for each treatment and the estimated treatment difference for the treatment comparisons of Arm 1 versus Arm 5, Arm 2 versus Arm 5, Arm 3 versus Arm 5 and Arm 4 versus Arm 5 will be presented together with the 95% confidence interval for the differences and corresponding p-values from

the multiple imputation procedure.

#### **Endpoint / Variables**

Total rescue use measured between the beginning of month 4 and the end of month 6 as determined by the MDI rescue sensor

#### **Summary**

The endpoint will be summarised using descriptive statistics (n, mean, SD, median, min, max) for each treatment arm.

To explore the effect of 6 months use of the CIS on a participant's rescue medicine usage, the following displays will be presented,

- Summary statistics (n, mean, SD, median, min, max) of Total rescue use measured between the beginning of month 4 and the end of month 6 as determined by the MDI rescue sensor
- Total rescue use will be summarized by each individual month (Month 1 Month 6) and then displayed as a total between month 4 – 6.

# 7.2.3. Asthma Control Endpoints

The asthma control secondary endpoints are:

- Change from baseline (Randomisation) in ACT total score at Month 6 (Visit 10), measured at baseline (Visit 2, 3 or 4) and Month 6 (Visit 10)
- Percentage of patients becoming controlled as defined as an Asthma Control Test score ≥20 at Month 6 (Visit 10)
- Percentage of patients with an increase from baseline ≥ 3 in ACT total score at Month 6 (Visit 10)
- Percentage of patients who have either an ACT total score of  $\geq 20$  and/or an increase from baseline of  $\geq 3$  in ACT total score at Month 6 (Visit 10)

# 7.2.3.1. Summary Measure

The asthma control summary measures are:

- The difference in LS means of the change from baseline in ACT total score at month 6, along with a 95% confidence interval and p-value for the difference, analysed using an MMRM model.
- An adjusted odds ratio on percentage of patients becoming controlled as defined as an ACT total score ≥ 20 at Month 6, along with a 95% confidence interval and p-value for the percentage, analysed using a logistic regression model.
- An adjusted odds ratio on percentage of patients with an increase from baseline ≥ 3 in ACT total score at Month 6, along with a 95% confidence interval and p-value for the percentage, analysed using a logistic regression model.
- An adjusted odds ratio on percentage of patients who have either an ACT total score of ≥ 20 and/or an increase from baseline of ≥ 3 in ACT total score at Month 6, along with a 95% confidence interval and p-value for the percentage, analysed using a logistic regression model.

# 7.2.3.2. Population of Interest

The asthma control analyses will be based on the Intent-to-Treat population.

# 7.2.3.3. Strategy for Intercurrent (Post-Randomisation) Events

Intercurrent events for the asthma control outcomes were identified as:

- Early discontinuation of ELLIPTA
- Early discontinuation of the APP
- Early discontinuation of ELLIPTA sensor
- Early discontinuation of MDI sensor
- Early withdrawal from study
- Use of MDI rescue medication
- Use of prohibited medications
- Change of dose of ELLIPTA

The "Treatment policy" strategy will be applied to handle the "Early discontinuation of ELLIPTA sensor", "Early discontinuation of the APP", "Early discontinuation of MDI sensor", "Use of MDI rescue medication", "Use of prohibited medications" and "change of dose of ELLIPTA" for all asthma control exploratory endpoints. The strategy implies direct use of ACT data irrespective of the occurrence of these intercurrent events.

# 7.2.3.3.1. Change from baseline (Randomisation) in ACT total score at Month 6 (Visit 10)

The "treatment policy" strategy will be applied to all handle all the intercurrent events listed in Section 7.2.3.3 Strategy for Intercurrent (Post-Randomisation) Events. In other words, all observed data before early discontinuation of the study respective of treatment arm status (on-treatment) or CIS discontinuation status will be included in the analysis. No missing data will be imputed, missing data will be considered MAR. Therefore, the primary treatment arm effect to be estimated will be the mean change from baseline in ACT total score at month 6 and remaining on study.

# 7.2.3.3.2. Percentage of patients becoming controlled as defined as an Asthma Control Test score ≥20 at Month 6 (Visit 10)

The "Composite" strategy will be used for the "Early discontinuation of ELLIPTA" and 'Early discontinuation of study" intercurrent events. In the occurrence of these intercurrent events, the effect to be estimated will be the effect on the outcome of achieving an ACT total score of  $\geq 20$  at month 6 and remaining on ELLIPTA (off-ELLIPTA treatment data is not collected). Participants who do not meet the improvement threshold, have missing values for their ACT total score at month 6, or prematurely discontinue using ELLIPTA or the study will be classified as non-responders in all planned analyses for this endpoint.

The "Treatment policy" strategy will be used to handle discontinuation of the APP/sensor. This means direct assessment of ACT total score at month 6 against the responder criteria, irrespective of CIS discontinuation status.

# 7.2.3.3.3. Percentage of patients with an increase from baseline ≥ 3 in ACT total score at Month 6 (Visit 10)

The "Composite" strategy will be used for the "Early discontinuation of ELLIPTA" and 'Early discontinuation of study" intercurrent events. In the occurrence of these intercurrent events, the effect to be estimated will be the effect on the outcome of achieving an increase from baseline of  $\geq 3$  in ACT total score at month 6 and remaining on ELLIPTA (off-ELLIPTA treatment data is not collected). Participants who do not meet the improvement threshold, have missing values for their ACT total score at month 6, or discontinue using ELLIPTA or the study will be classified as non-responders in all planned analyses for this endpoint.

The "Treatment policy" strategy will be used to handle discontinuation of the APP/sensor. This means direct assessment of ACT total score at month 6 against the responder criteria, irrespective of CIS discontinuation status.

# 7.2.3.3.4. Percentage of patients who have either an ACT total score of ≥ 20 and/or an increase from baseline of ≥ 3 in ACT total score at Month 6 (Visit 10)

The "Composite" strategy will be used for the "Early discontinuation of ELLIPTA" and 'Early discontinuation of study" intercurrent events. In the occurrence of these intercurrent events, the effect to be estimated will be the effect on the composite outcome of achieving an ACT total score of  $\geq 20$  and/or an increase from baseline of  $\geq 3$  in ACT total score at month 6 and remaining on ELLIPTA (off-ELLIPTA treatment data is not collected). Participants who do not meet the improvement threshold, have missing values for their ACT total score at month 6, or discontinue using ELLIPTA during or the study will be classified as non-responders in all planned analyses for this endpoint.

The "Treatment policy" strategy will be used to handle discontinuation of the APP/sensor. This means direct assessment of ACT total score at month 6 against the responder criteria, irrespective of CIS discontinuation status.

# 7.2.3.4. Statistical Analyses / Methodology Specification

Details of the planned displays will be provided in 10.8 Appendix 8: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints/variables defined in Section 7.2.3.1 Summary Measure will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

### 7.2.3.4.1. Change from baseline in ACT total score at month 6

#### **Endpoint / Variables**

Change from baseline in ACT total score Month 6 (visit 10)

#### **Model Specification**

This endpoint will be analysed using a mixed model repeated measures (MMRM) model utilising the REML estimation approach and the default unstructured covariance matrix structure. Whilst missing data are not implicitly imputed in this analysis, there is an underlying assumption that the data are MAR. All non-missing data for a participant will be used within the analysis and, via modelling of the within-participant correlation structure, the derived treatment differences will be adjusted to take into account missing data.

Terms fitted in the model will include:

- Dependent Variable: change from baseline in ACT total score
- Covariates:
  - Fixed categorical: randomised treatment arm, visit (month 1 and 6), gender and country.
  - Fixed continuous: baseline ACT total score and age
  - Interaction terms: randomised treatment arm-by-visit, baseline ACT total score-by-visit
  - Random effect: participant

#### **Model Checking & Diagnostics**

- If this model fails to converge, alternative correlation structures may be considered
- Appropriate graphs will be reviewed as part of the model checking process to ensure that distributional
  assumptions hold. These will include a normal probability plot of the residuals and a plot of the
  residuals versus the fitted values (checking the normality assumption and constant variance
  assumption of the model, respectively).
- Interactions with treatment will be explored for other model covariates and tests for interactions will be at the 2-sided 10% significance level. Any significant interactions that are found will be thoroughly investigated and where necessary, extra outputs will be produced.

#### **Model Results Presentation**

Adjusted mean change from baseline values for each treatment arm will be presented with their associated standard errors. The estimated treatment difference along with corresponding standard error, 95% confidence interval (CI) and p-value will be presented for the treatment comparisons at month 6 (Visit 10).

#### 7.2.3.4.2. ACT total score ≥20 at month 6

#### **Endpoint / Variables**

Percentage of patients becoming controlled as defined as an Asthma Control Test score ≥20 at Month 6 (Visit 10)

#### **Model Specification**

This endpoint will be analysed using a logistic regression model. Only the month 6 (visit 10) data will be included in the model. Month 1 (visit 5) data will not be implemented since by this timepoint participants may not have reverted to steady medicating behaviour.

Will not be included since participants may not have reverted to normally medicating practise within one month's use of the CIS/

#### Terms in the model:

Dependent variable: ACT total score ≥20 responder/non-responder at month 6 (binary score)

- Covariates:
  - Categorical: randomised treatment arm, gender and country
  - Continuous: baseline ACT total score and age.

Patients who have a missing ACT total score at month 6 (visit 10) (i.e. no ACT data on-treatment) will be classified as non-responders at that visit.

Computation of confidence intervals for the odds ratios is based in the individual Wald tests.

#### **Model Checking & Diagnostics**

If the likelihood maximisation algorithm fails to converge due to complete or quasi-complete separation of the data then Firth's penalized likelihood (Firth, 1993) will be implemented by use of the FIRTH option on the MODEL statement in PROC LOGISTIC.

The fit of the logistic regression model will be assessed by examining the ROC curve and other diagnostic plots

#### **Model Results Presentation**

The number and percentage of participants with a response within each randomised treatment arm will be presented by visit, together with the adjusted odds ratio comparing CIS Arms 1, 2, 3, 4 with Arm 5, associated 95% CIs and p-values.

#### 7.2.3.4.3. Increase from Baseline of ≥ 3 in ACT total score at month 6

### **Endpoint**

Percentage of patients with an increase from baseline ≥ 3 in ACT total score at Month 6 (Visit 10)

#### **Model Specification**

This endpoint will be analysed using a logistic regression model. Only the month 6 (visit 10) data will be included in the model. Month 1 (visit 5) data will not be implemented since by this timepoint participants may not have reverted to steady medicating behaviour.

Terms in the model:

- Dependent variable: Increase from baseline of ≥ 3 in ACT total score at month 6 responder/nonresponder (binary score)
- Covariates:
  - Categorical: randomised treatment arm, gender and country
  - Continuous: baseline ACT total score and age.

Patients who have a missing ACT total score at month 6 (visit 10) (i.e. no ACT data on-treatment) will be classified as non-responders at that visit.

Computation of confidence intervals for the odds rations is based in the individual Wald tests.

#### **Model Checking & Diagnostics**

If the likelihood maximisation algorithm fails to converge due to complete or quasi-complete separation of the data then Firth's penalized likelihood (Firth, 1993) will be implemented by use of the FIRTH option on the MODEL statement in PROC LOGISTIC.

The fit of the logistic regression model will be assessed by examining the ROC curve and other diagnostic plots

#### **Model Results Presentation**

The number and percentage of participants with a response within each randomised treatment arm will be presented by visit, together with the adjusted odds ratio comparing CIS Arms 1, 2, 3, 4 with Arm 5, associated 95% CIs and p-values.

# 7.2.3.4.4. ACT total score of $\geq$ 20 and/or an increase from baseline of $\geq$ 3 in ACT total score at Month 6 (Visit 10).

#### **Endpoint**

Percentage of patients who have either an ACT total score of  $\geq$  20 and/or an increase from baseline of  $\geq$  3 in ACT total score at Month 6 (Visit 10).

# **Model Specification**

This endpoint will be analysed using a logistic regression model. Only the month 6 (visit 10) data will be included in the model. Month 1 (visit 5) data will not be implemented since by this timepoint participants may not have reverted to steady medicating behaviour.

Terms in the model:

- Dependent variable: Composite ACT total score ≥ 20 and/or increase from baseline of ≥ 3 in ACT total score at month 6 responder/non-responder (binary score)
- Covariates:
  - Categorical: randomised treatment arm, gender and country
  - Continuous: baseline ACT total score and age.

Patients who have a missing ACT total score at month 6 (visit 10) (i.e. no ACT data on-treatment) will be classified as non-responders at that visit.

Computation of confidence intervals for the odds rations is based in the individual Wald tests.

#### **Model Checking & Diagnostics**

If the likelihood maximisation algorithm fails to converge due to complete or quasi-complete separation of the data then Firth's penalized likelihood (Firth, 1993) will be implemented by use of the FIRTH option on the MODEL statement in PROC LOGISTIC.

The fit of the logistic regression model will be assessed by examining the ROC curve and other diagnostic plots.

#### **Model Results Presentation**

The number and percentage of participants with a response within each randomised treatment arm will be presented by visit, together with the adjusted odds ratio comparing CIS Arms 1, 2, 3, 4 with Arm 5, associated 95% CIs and p-values.

# 7.3. Exploratory and Other Analyses

The impact of the HCP having access to sensor data on percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor will be assessed by the following comparisons:

• Arm 1 vs Arm 2

• Arm 3 vs Arm 4

The impact of having Rescue Medication data being available on the percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor will be assessed by the following comparisons:

- Arm 1 vs Arm 3
- Arm 2 vs Arm 4

These estimates will be generated from the multiple imputation analysis used to assess the primary endpoint.

The effect of 6 months use with CIS on health care utilisation will be explored as well as its effect on the following patient reported outcomes (PROs); asthma system utility index (ASUI). St. Georges Respiratory Questionnaire (SGRQ), Patient Activation Measure (PAM), Medication Adherence Report Scale for Asthma (MARS-A), Beliefs in Medicine Questionnaire (BMQ).

The reliability and usability of the CIS, as well as the impact of the adherence on Fractional exhaled nitric oxide (FeNO) and Peak Expiratory Flow (PEF) will be assessed.

### 7.3.1. Exploratory ELLIPTA Adherence Measure Analyses

### **7.3.1.1.** Endpoint

The percentage of ELLIPTA doses taken (daily adherence) between the beginning of Month 4 and the end of Month 6 as determined by the maintenance sensor. Daily adherence is defined as the participant taking one dose of Relvar/Breo ELLIPTA, within a 24-hour period, starting at 12.00am each day of the run-in and treatment period

# 7.3.1.2. Summary Measure

The mean difference in daily adherence between the comparisons of interest will be estimated from an Analysis of Covariance (ANCOVA) model allowing for effects due to randomised treatment, baseline adherence, duration of run-in (visits), country, gender, and age (years).

# 7.3.1.3. Population of Interest

The exploratory adherence analyses will be based on the Intent-To-Treat population.

# 7.3.1.4. Strategy for Intercurrent (Post-Randomisation) Events

The steps detailed in Section 7.1.4 Strategy for Intercurrent (Post-Randomisation) Events will be applied sequentially when deriving the secondary adherence endpoints. See Section 10.5.3.1 ELLIPTA Device Sensor Assessments for further derivation details.

# 7.3.1.4.1. Events prior to premature discontinuation of the ELLIPTA maintenance sensor

The treatment policy estimand is directly assessed using the observed adherence data while the ELLIPTA maintenance sensor is in use, regardless of whether the CIS feedback is discontinued.

Any missing intermittent adherence data will be imputed as non-adherent i.e. the participant will be assumed to have not taken their treatment within the 24-hour time period/window, where there is no evidence of device or technical/transmission failure.

Missing intermittent adherence data due to a medical device incident such as device failure, technical failure of the sensor, or data transmission failure will be assumed to be missing at random (MAR). For each participant, the percentage adherence measure will be calculated from the proportion of the number of days a participant is adherent divided by the number of days data provided in that month.

# 7.3.1.4.2. Events following premature discontinuation of the ELLIPTA maintenance sensor

It is assumed that participants would continue to take ELLIPTA as they would have without the CIS intervention (J2R imputation) following discontinuation of the ELLIPTA maintenance sensor.

It is assumed that ELLIPTA treatment is no longer appropriate if the participant discontinues ELLIPTA but remains in the study or withdraws for a reason related to ELLIPTA. The ELLIPTA adherence endpoint is no longer considered relevant and subsequent follow-up is excluded from the analysis, with participants weighted in the analysis by the proportion of months 4 to 6 for which data is included.

It is assumed that participants would continue to take ELLIPTA as they would have with their allocated CIS intervention (MAR imputation) following concurrent discontinuation of the ELLIPTA maintenance sensor and withdrawal unrelated to ELLIPTA or CIS.

# 7.3.1.5. Statistical Analyses / Methods

Details of the planned displays will be provided in Section 10.8, Appendix 8: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints /variables defined in Section 7.3.1.1 Endpoint will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

### 7.3.1.6. Statistical Analyses / Methodology Specification

# 7.3.1.6.1. The percentage of ELLIPTA doses taken (daily adherence) between the beginning of Month 4 and the end of Month 6

#### **Endpoint / Variables**

The percentage of ELLIPTA doses taken (daily adherence) between the beginning of Month 4 and the end of Month 6 as determined by the maintenance sensor for the following treatment arm comparisons:

- HCP having access to sensor data
  - Arm 1 vs Arm 2
  - Arm 3 vs Arm 4
- Rescue medication data being available
  - Arm 1 vs Arm 3
  - Arm 2 vs Arm 4

Daily adherence is defined as the participant taking one dose of Relvar/Breo ELLIPTA within a 24-hour period, starting at 12.00am each day of treatment period.

#### **Multiple Imputation Specification**

Imputation will be carried out using monthly adherence rates for months 1 to 6. 1000 draws will be used. For each draw, four intermediate imputation datasets will be created to allow for the handling of fully unobserved months (using set A imputations) and partially unobserved months (using set B imputations).

- Set A where the partially observed month is directly estimated under the MAR assumption as the
  proportion of the number of days a participant is adherent divided by the number of days data
  provided in that month.
  - J2R imputations
  - MAR imputations
- Set B where the partially observed month is set to missing.
  - J2R imputations
  - MAR imputations

The timing of the intercurrent events of discontinuation of the ELLIPTA maintenance sensor, discontinuation of ELLIPTA and withdrawal from study will be used to identify the proportion of each month to be assigned as observed data, J2R imputed data, MAR imputed data, or no data. The strategy for handling intercurrent events is described in Section 7.1.4 Strategy for Intercurrent (Post-Randomisation) Events.

Within each imputation draw, for each month, the observed and any imputed data will be combined to provide a percentage adherence value. The values for months 1 to 6 will be combined to create the value

for the secondary analysis and the weight to be assigned to each participant.

Multiple imputation using Rubin's rules will be used to estimate the treatment effect and associated standard error, by performing the ANCOVA analysis described below on the secondary endpoint within each dataset.

The multiple imputation will be implemented using the methods described in Carpenter, 2013, using the macros available from <a href="https://missingdata.lshtm.ac.uk/2017/04/06/gsk-five-macros/">https://missingdata.lshtm.ac.uk/2017/04/06/gsk-five-macros/</a>.

#### **Model Specification**

The analysis will be performed on the percentage adherence between Months 4 and 6 using an Analysis of Covariance (ANCOVA) model allowing for effects due to randomised treatment arm, baseline adherence, duration of run-in (visits), country, gender, and age (years).

Baseline adherence will be the percentage ELLIPTA doses taken (daily adherence) during the last 28 days of the run-in period prior to randomisation. Randomised treatment, duration of run-in (visits), country, and gender will be included as categorical covariates; baseline adherence and age (years) will be included as continuous covariates.

Each participant will be weighted by the proportion of months 4 to 6 for which data is included in the percentage adherence endpoint (both observed and imputed data are accounted for in the weighting).

Data from five individual CIS treatment arms will be included in the model, and used to estimate the difference between:

- Arm 1 and Arm 2
- Arm 3 and Arm 4
- Arm 1 and Arm 3
- Arm 2 and Arm 4

#### **Model Checking & Diagnostics**

Normality assumptions underlying the ANCOVA model used for analysis will be examined in a limited number of imputed datasets by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.

If there are any departures from the distributional assumptions, alternative models may be explored using appropriately transformed data.

Interactions with treatment will be explored for other model covariates and tests for interactions will be at the 2-sided 10% significance level. Any significant interactions that are found will be thoroughly investigated and where necessary, extra outputs will be produced.

#### **Model Results Presentation**

Summary statistics (mean, standard deviation, median, minimum, maximum) of the primary endpoint will be provided, based on the observed percentages.

The adjusted means for each treatment arm and the estimated treatment arm difference for the treatment arm comparisons of interest will be presented together with the 95% confidence interval for the differences

and corresponding p-values from the multiple imputation procedure.

# 7.3.2. Exploratory Health Care Utilization Analyses

### **7.3.2.1.** Endpoints

- Number of outpatient visits relating to asthma
- Number of primary care visits relating to study HCP dashboard review (for relevant study arms)
- Number of and duration of hospitalisations, and ER visits due to asthma
- Annualised rate of severe exacerbations
- Number of unscheduled visits to primary care related to Asthma

# 7.3.2.2. Population of Interest

The exploratory analyses will be based on the Intent-To-Treat population.

#### **Endpoint**

Healthcare Utilisation -

- Number of outpatient visits relating to asthma
- Number of and duration of hospitalisations, and ER visits due to asthma
- Number of unscheduled visits to primary care related to Asthma

### Summary

- The number and percentage of participants by frequency of unscheduled healthcare resource contacts (0, 1, 2, 3, 4, >4) will be summarized by contact type and treatment arm to characterize the level of healthcare associated with an asthma exacerbation. The frequency counts for each participant will be the total sum of contacts (or days in hospital) by type.
- The following types of healthcare contact for an exacerbation are recorded in the eCRF:
  - Number of telephone calls
  - Number of home/day visits
  - Number of home/night visits
  - Number of physician office/practice visits
  - Number of urgent care/outpatient visits
  - Number of emergency room visits
  - Number of inpatient hospitalisation days
  - Number of contacts due to an exacerbation

#### **Endpoint**

Healthcare Utilisation -

• Number of primary care visits relating to study HCP dashboard review (for relevant study arms)

#### **Summary**

• The number and percentage of participants by frequency of unscheduled healthcare resource contacts (0, 1, 2, 3, 4, >4) will be summarized by contact type and treatment arm to characterize the level of healthcare associated with an asthma exacerbation. The frequency counts for each participant will be the total sum of contacts (or days in hospital) by type.

#### **Endpoint**

Healthcare Utilisation -

Annual rate of severe asthma exacerbations

#### Summary

- The number and percentage of participants reporting an asthma exacerbation (on-treatment and post-treatment) will be summarised by treatment arm.
- The number and percentage of participants with each number of exacerbations (0, 1, 2, 3, 4, >4) and the total number of exacerbations per treatment arm will also be summarised.
- For the purposes of summarizing these data, the annualized rate of severe asthma exacerbations for the ITT population will be calculated for each participant as
  - o the number of exacerbations / time on Relvar/Breo (in years) from randomisation.
- The summaries will include on-treatment exacerbations, from randomisation date to min(stop date of exposure + 1 day, date of study discontinuation).
- The number and percentage of participants with an exacerbation that led to withdrawal of study, hospitalization, systemic/oral corticosteroids/antibiotics/medication being taken, or emergency room visit will be summarised by treatment arm.
- A listing of severe exacerbations will be provided.

# 7.3.3. Exploratory Patient Reported Outcomes (PROs) Analyses

#### **7.3.3.1.** Endpoints

- Percentage of patients meeting a responder threshold of  $\geq 0.09$  points improvement from baseline (randomisation) for the ASUI total score at month 6
- Change from baseline (randomisation) in ASUI total score at month 6
- Percentage of patients meeting a responder threshold of  $\geq 4$  points improvement (decrease) from baseline (randomisation) for the SGRQ total score at month 6
- Change from baseline (randomisation) in SRGO total score at month 6
- Change from baseline (screening) in PAM total score at month 6
- Change from baseline (screening) in MARS-A total score at month 6
- Change from baseline (screening) in BMQ General Benefit score at month 6
- Change from baseline (screening) in BMQ General Harm score at month 6
- Change from baseline (screening) in BMQ General Overuse score at month 6
- Change from baseline (screening) in BMQ Specific Necessity score at month 6
- Change from baseline (screening) in BMQ Specific Concern score at month 6

### 7.3.3.2. Summary Measure

The PRO summary measures to determine treatment arm effect are:

- An adjusted odds ratio on percentage of patients meeting a responder threshold of
   ≥ 0.09 points improvement from baseline for the ASUI total score at Month 6,
   along with a 95% confidence interval and p-value for the percentage, analysed
   using a logistic regression model.
- The difference in LS means of the change from baseline in ASUI total score at month 6, along with a 95% confidence interval and p-value for the difference, analysed using an MMRM model.
- An adjusted odds ratio on percentage of patients meeting a responder threshold of  $\geq 4$  points improvement (decrease) from baseline for the SGRQ total score at Month 6, along with a 95% confidence interval and p-value for the percentage, analysed using a logistic regression model.
- The difference in LS means of the change from baseline in SGRQ total score at month 6, along with a 95% confidence interval and p-value for the difference, analysed using an MMRM model.
- Mean change from baseline (screening) in PAM-13 total score at month 6.
- Mean change from baseline (screening) in MARS-A total score at month 6
- Mean change from baseline (screening) in BMQ General Benefit score at month
- Mean change from baseline (screening) in BMQ General Harm score at month 6
- Mean change from baseline (screening) in BMQ General Overuse score at month 6
- Mean change from baseline (screening) in BMQ Specific Necessity score at month 6
- Mean change from baseline (screening) in BMQ Specific Concern score at month 6

#### 7.3.3.3. Population of Interest

The PRO exploratory summaries and analysis will be based on the "Intent-to-Treat" population.

### 7.3.3.4. Strategy for Intercurrent (Post-Randomisation) Events

Intercurrent events for the ASUI and SGRQ outcomes were identified as:

- Early discontinuation of ELLIPTA
- Early discontinuation of the APP
- Early discontinuation of ELLIPTA sensor
- Early discontinuation of MDI sensor
- Early withdrawal from study
- Use of MDI rescue medication
- Use of prohibited medications
- Change of dose of ELLIPTA

The "Treatment policy" strategy will be applied to handle the "Early discontinuation of ELLIPTA sensor", "Early discontinuation of the APP", "Early discontinuation of MDI sensor", "Use of MDI rescue medication", "Use of prohibited medications" and "change of dose of ELLIPTA" for all PRO exploratory endpoints. The strategy implies direct use of PRO data irrespective of the occurrence of these intercurrent events.

# 7.3.3.4.1. Percentage of patients meeting a responder threshold of ≥ 0.09 points improvement from baseline (randomisation) for the ASUI total score at Month 6 (Visit 10)

The "Composite" strategy will be used for the "Early discontinuation of ELLIPTA" and 'Early discontinuation of study" intercurrent events. In the occurrence of these intercurrent events, the effect to be estimated will be the effect on the outcome of achieving an improvement from baseline of  $\geq 0.09$  in ASUI total score at month 6 and remaining on ELLIPTA (off-ELLIPTA treatment data is not collected). Participants who do not meet the improvement threshold, have missing values for their ASUI total score at month 6, or discontinue using ELLIPTA or the study will be classified as non-responders in all planned analyses for this endpoint.

The "Treatment policy" strategy will be used to handle discontinuation of the APP/sensor. This means direct assessment of ASUI total score at month 6 against the responder criteria, irrespective of CIS discontinuation status.

# 7.3.3.4.2. Change from baseline (randomisation) in ASUI total score at month 6 (Visit 10)

The "treatment policy" strategy will be applied to all handle all the intercurrent events listed in 7.4.3.4. In other words, all observed data before early discontinuation of the study respective of treatment status (on-treatment) or CIS discontinuation status will be included in the analysis. No missing data will be imputed, missing data will be considered MAR. Therefore, the primary treatment effect to be estimated will be the mean change from baseline in ASUI total score at month 6 and remaining on the study.

# 7.3.3.4.3. Percentage of patients meeting a responder threshold of ≥ 4 points improvement (decrease) from baseline (randomisation) for the SGRQ total score at month 6 (Visit 10)

The "Composite" strategy will be used for the "Early discontinuation of ELLIPTA" and 'Early discontinuation of study" intercurrent events. In the occurrence of these intercurrent events, the effect to be estimated will be the effect on the outcome of achieving an improvement from baseline of  $\geq 4$  in SGRQ total score at month 6 and remaining on ELLIPTA (off-ELLIPTA treatment data is not collected). Participants who do not meet the improvement threshold, have missing values for their SGRQ total score at month 6, or discontinue using ELLIPTA or the study will be classified as non-responders in all planned analyses for this endpoint.

The "Treatment policy" strategy will be used to handle discontinuation of the APP/sensor. This means direct assessment of SGRQ total score at month 6 against the responder criteria, irrespective of CIS discontinuation status.

# 7.3.3.4.4. Change from baseline (Randomisation) in SGRQ total score at Month 6 (Visit 10)

The "treatment policy" strategy will be applied to all handle all the intercurrent events listed in 7.4.3.4. In other words, all observed data before early discontinuation of the study respective of treatment status (on-treatment) or CIS discontinuation status will be included in the analysis. No missing data will be imputed, missing data will be considered MAR. Therefore, the primary treatment effect to be estimated will be the mean change from baseline in SGRQ total score at month 6 and remaining on the study.

# 7.3.3.4.5. Change from baseline (Screening) in PAM-13, MARS-A, and BMQ total score at Month 6 (Visit 10)

The mean change from baseline in PAM-13, MARS-A and all scales for the BMQ questionnaires at month 6 will be summarised using descriptive statistics (n, mean, SD, median, min, max) for each treatment arm. The "treatment policy" strategy will be applied to all handle all the intercurrent events listed in 7.4.3.4. In other words, all observed data before early discontinuation of the study respective of treatment status (ontreatment) or CIS discontinuation status will be included in the analysis. No missing data will be imputed, missing data will be considered MAR. Therefore, the primary treatment arm effect to be estimated will be the mean change from baseline in total score at month 6 and remaining on the study.

No formal statistical analyses will be performed for these endpoints.

# 7.3.3.5. Statistical Analyses / Methodology Specification

Details of the planned displays will be provided in Section 10.8, Appendix 8: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.3.3.1, Endpoints, will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

# 7.3.3.5.1. Increase from Baseline of ≥ 0.09 in ASUI total score at Month 6 (Visit 10)

#### **Endpoint / Variables**

Percentage of patients meeting a responder threshold of  $\geq$  0.09 points improvement from baseline for the ASUI total score at Month 6 (Visit 10)

#### **Model Specification**

This endpoint will be analysed using a logistic regression model. Only the month 6 (visit 10) data will be included in the model. Month 1 (visit 5) data will not be implemented since by this timepoint participants may not have reverted to steady medicating behaviour

Terms in the model:

- Dependent variable: ASUI responder/non-responder score (binary score)
- Covariates:
  - Categorical: randomised treatment arm, gender and country
  - Continuous: baseline ASUI total score and age.

Patients who have a missing ASUI total score at month 6 (visit 10) (i.e. no ASUI data on-treatment) will be classified as non-responders at that visit. This rule will apply to all above analyses.

Computation of confidence intervals for the odds ratios is based in the individual Wald tests.

#### **Model Checking & Diagnostics**

If the likelihood maximisation algorithm fails to converge due to complete or quasi-complete separation of the data then Firth's penalized likelihood (Firth, 1993) will be implemented by use of the FIRTH option on the MODEL statement in PROC LOGISTIC.

The fit off the logistic regression model will be assessed by examining the ROC curve and other diagnostic plots.

#### **Model Results Presentation**

The number and percentage of participants with a response within each randomised treatment arm will be presented by visit, together with the adjusted odds ratio comparing CIS Arms 1, 2, 3, 4 with Arm 5, associated 95% CIs and p-values.

# 7.3.3.5.2. Change from baseline (Randomisation) in ASUI total score at Month 6 (Visit 10)

#### **Endpoint / Variables**

Mean change from baseline in ASUI total score at Month 6 (Visit 10)

#### **Model Specification**

This endpoint will be analysed using a mixed model repeated measures (MMRM) model utilising the REML estimation approach and the default unstructured covariance matrix structure. Whilst missing data are not implicitly imputed in this analysis, there is an underlying assumption that the data are MAR. All non-missing data for a participant will be used within the analysis and, via modelling of the within-participant correlation structure, the derived treatment differences will be adjusted to take into account missing data.

Terms fitted in the model will include:

- Dependent Variable: change from baseline in ASUI total score at month 6
- Covariates:
  - Fixed categorical: randomised treatment arm, visit (month 1 and 6), gender and country.
  - Fixed continuous: baseline ASUI total score and age
  - o Interaction terms: randomised treatment arm-by-visit, baseline ASUI total score-by-visit
  - Random effect: participant

#### **Model Checking & Diagnostics**

- If this model fails to converge, alternative correlation structures may be considered
- Appropriate graphs will be reviewed as part of the model checking process to ensure that distributional
  assumptions hold. These will include a normal probability plot of the residuals and a plot of the residuals
  versus the fitted values (checking the normality assumption and constant variance assumption of the
  model, respectively).
- Interactions with treatment will be explored for other model covariates and tests for interactions will be at the 2-sided 10% significance level. Any significant interactions that are found will be thoroughly investigated and where necessary, extra outputs will be produced.

#### **Model Results Presentation**

Adjusted mean change from baseline values for each treatment arm will be presented with their associated standard errors. The estimated treatment difference along with corresponding standard error, 95% confidence interval (CI) and p-value will be presented for the treatment comparisons at month 6 (Visit 10).

#### 7.3.3.5.3. Increase from Baseline of $\geq 4$ in SGRQ total score at Month 6 (Visit 10)

#### **Endpoint / Variables**

Percentage of patients meeting a responder threshold of  $\geq 4$  points improvement from baseline for the SGRQ total score at month 6

#### **Model Specification**

This endpoint will be analysed using a logistic regression model. Only the month 6 (visit 10) data will be included in the model. Month 1 (visit 5) data will not be implemented since by this timepoint participants may not have reverted to steady medicating behaviour

Terms in the model:

- Dependent variable: SGRQ responder/non-responder score (binary score)
- Covariates:
  - Categorical: randomised treatment arm, gender and country
  - Continuous: baseline SGRQ total score and age.

Patients who have a missing SGRQ total score at month 6 (visit 10) (i.e. no SGRQ data on-treatment) will be classified as non-responders at that visit. This rule will apply to all above analyses.

Computation of confidence intervals for the odds ratios is based in the individual Wald tests.

#### **Model Checking & Diagnostics**

If the likelihood maximisation algorithm fails to converge due to complete or quasi-complete separation of the data then Firth's penalized likelihood (Firth, 1993) will be implemented by use of the FIRTH option on the MODEL statement in PROC LOGISTIC.

The fit of the logistic regression model will be assessed by examining the ROC curve and other diagnostic plots.

#### **Model Results Presentation**

The number and percentage of participants with a response within each randomised treatment arm will be presented by visit, together with the adjusted odds ratio comparing CIS Arms 1, 2, 3, 4 with Arm 5, associated 95% CIs and p-values.

# 7.3.3.5.4. Change from baseline (Randomisation) in SGRQ total score at Month 6 (Visit 10)

#### **Endpoint / Variables**

Mean change from baseline in SGRQ total score at Month 6 (Visit 10)

### **Model Specification**

This endpoint will be analysed using a mixed model repeated measures (MMRM) model utilising the REML estimation approach and the default unstructured covariance matrix structure. Whilst missing data are not implicitly imputed in this analysis, there is an underlying assumption that the data are MAR. All non-missing data for a participant will be used within the analysis and, via modelling of the within-participant correlation

structure, the derived treatment differences will be adjusted to take into account missing data.

Terms fitted in the model will include:

- Dependent Variable: change from baseline in SGRQ total score at month 6
- Covariates:
  - Fixed categorical: randomised treatment arm, visit (month 1 and 6), gender and country.
  - Fixed continuous: baseline SGRQ total score and age
  - o Interaction terms: randomised treatment arm-by-visit, baseline SGRQ total score-by-visit
  - Random effect: participant

#### **Model Checking & Diagnostics**

- If this model fails to converge, alternative correlation structures may be considered
- Appropriate graphs will be reviewed as part of the model checking process to ensure that
  distributional assumptions hold. These will include a normal probability plot of the residuals and a
  plot of the residuals versus the fitted values (checking the normality assumption and constant
  variance assumption of the model, respectively).
- Interactions with treatment will be explored for other model covariates and tests for interactions will be at the 2-sided 10% significance level. Any significant interactions that are found will be thoroughly investigated and where necessary, extra outputs will be produced.

#### **Model Results Presentation**

Adjusted mean change from baseline values for each treatment arm will be presented with their associated standard errors. The estimated treatment difference along with corresponding standard error, 95% confidence interval (CI) and p-value will be presented for the treatment comparisons at month 6 (Visit 10).

# 7.3.4. Exploratory Fractionated Exhaled Nitric Oxide (FeNO) and Peak Expiratory Flow (PEF) Analyses

#### **7.3.4.1.** Endpoints

- FeNO at Screening (Visit 1), Randomisation (Visit 2,3 or 4), Month 1 (Visit 5) and Month 6 (Visit 10).
- Change from baseline (randomisation) in FeNO measured at Month 1 (Visit 5) and Month 6 (Visit 10)
- PEF at Screening (Visit 1), Randomisation (Visit 2,3 or 4), Month 1 (Visit 5) and Month 6 (Visit 10).
- Change from baseline (randomisation) in PEF measured at Month 1 (Visit 5) and Month 6 (Visit 10)

### 7.3.4.2. Summary Measures

The FeNO and PEF summary measures are:

• Summary statistics (n, mean, SD, median, min, max) for each treatment arm of screening (Visit 1), Randomisation (Visit 2,3 or 4), Month 1 (Visit 5) and Month 6 (Visit 10) and changes from baseline (screening) at month 1 (visit 5) and month 6 (visit 10)

# 7.3.4.3. Population of Interest

The FeNO and PEF exploratory summaries will be based on the Intent-to-Treat population.

# 7.3.4.4. Strategy for Intercurrent (Post-Randomisation) Events

Intercurrent events for the FeNO and PEF outcomes were identified as:

- Early discontinuation of ELLIPTA
- Early discontinuation of the APP
- Early discontinuation of ELLIPTA sensor
- Early discontinuation of MDI sensor
- Early withdrawal from study
- Use of MDI rescue medication
- Use of prohibited medications
- Change of dose of ELLIPTA

The "Treatment policy" strategy will be applied to handle all intercurrent event for the FeNO and PEF exploratory endpoints. The strategy implies direct use of FeNO and PEF data irrespective of the occurrence of these intercurrent events.

# 7.3.4.5. Statistical Analyses / Methodology Specification

Details of the planned displays will be provided in Section 10.8, Appendix 8: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.3.4.1 Endpoints will be summarised using descriptive statistics, graphically presented (where appropriate) and listed. No formal statistical analyses will be performed for these endpoints.

#### **Endpoint**

- FeNO at Screening (Visit 1), Randomisation (Visit 2,3 or 4), Month 1 (Visit 5) and Month 6 (Visit 10)
- Change from baseline (randomisation) in FeNO measured at Month 1 (Visit 5) and Month 6 (Visit 10)
- PEF at Screening (Visit 1), Randomisation (Visit 2,3 or 4), Month 1 (Visit 5) and Month 6 (Visit 10)
- Change from baseline (randomisation) in PEF measured at Month 1 (Visit 5) and Month 6 (Visit 10)

#### Summary

All endpoints to be summarised using descriptive statistics (n, mean, SD, median, min, max) for each randomised treatment arm.

To explore the impact of maintenance adherence levels on FeNO and PEF, the following displays will be presented,

 Summary statistics (n, mean, SD, median, min, max) of change from baseline at Month 6 (Visit 10) in FeNO per quartile of the observed primary endpoint measure, percentage of ELLIPTA doses taken (daily adherence) between the beginning of Month 4 and the end of Month 6 as determined by the

#### maintenance sensor

- Summary statistics (n, mean, SD, median, min, max) of change from baseline at Month 6 (Visit 10) in PEF per quartile of the observed primary endpoint measure, percentage of ELLIPTA doses taken (daily adherence) between the beginning of Month 4 and the end of Month 6 as determined by the maintenance sensor
- Note: the quartiles of a ranked adherence data values are four subsets whose boundaries are the three quartile points (25th, 50th and 75th percentiles)
- A scatter plot of the change from baseline at Month 6 (Visit 10) in FeNO by observed primary endpoint measure will be presented. This will be repeated for change from baseline at Month 6 (Visit 10) in PEF.

#### 7.3.5. Qualitative data from exit interviews

Analysis of the qualitative data from exit interviews will be analyzed following a separate qualitative analysis plan and presented in a separate Clinical Study Report (CSR).

# 8. SAFETY ANALYSES

Safety analyses will be based on the ITT Population and will include all study data (runin, on and post-treatment), unless otherwise specified.

Safety endpoints will include:

- Incidence and type of serious adverse events
- Incidence and type of adverse drug reactions (ADR)
- Incidence and type of non-serious adverse events leading to study withdrawal

# 8.1. Adverse Events Analyses

SAEs, AEs leading to withdrawal and non-serious ADRs will be collected.

The incidence of any given adverse event (SAE, ADR or non-serious AEs leading to withdrawal) for each treatment group is defined as the proportion of participants in that group who have experienced at least one such adverse event during the study period.

Adverse event (SAE or ADR) summaries including the summary of adverse drug reactions (ADRs), Serious (SAEs) and non-serious adverse events leading to withdrawal of study will be based on GSK Core Data Standards. The details of the planned displays are provided in Section 10.8 Appendix 8: List of Data Displays.

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) coding dictionary. The version of MedDRA used in reporting will be noted in a footnote of the AE overview table.

For the standard on-treatment and post-treatment AE tables, the number and percentage of participants with all AEs (regardless of causality) will be summarized for each treatment group by system organ class (SOC) and preferred term (PT). The ordering of the SOCs and the PTs within the SOCs will both be in descending order of total incidence. A SOC will not be presented when the overall incidence for any AE within the particular system is zero. If the total incidence for any two or more AEs is equal, the events will be presented in alphabetical order.

# 8.2. Adverse Events of Special Interest

A comprehensive list of MedDRA terms based on clinical and safety review will be used to identify AEs of special interest to FF and Relvar/Breo. Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting and/or emerging data from on-going studies may highlight additional AEs of special interest; therefore, the list of terms to be used for each event of interest and the specific events of interest will be based on the clinical and safety review agreements documented and in place at time of reporting and prior to unblinding the study. The details of the planned displays are provided in Section 10.8 Appendix 8: List of Data Displays.

The number and percentage of participants with on-treatment AEs of special interest will be summarized for each treatment group by special interest term, subgroup and PT. The ordering of the special interest terms, the subgroups and the PTs within them will all be in descending order of total incidence. If the total incidence for any two or more AEs is equal, the events will be presented in alphabetical order. This summary will be produced for non-serious ADRs, and repeated for serious ADRs, all ADRs and SAEs. The list of MedDRA terms used to identify AEs of special interest will be displayed.

# 8.3. Pregnancy

Any pregnancies reported during the study will be summarized in CSR case narratives. Any pregnancy complication or elective termination of a pregnancy for medical reasons will be recorded as an AE or SAE and included in summaries and listings of AEs/SAEs.

# 8.4. Other Safety Measures

All Relvar/Breo ELLIPTA inhaler device malfunction data for participants reporting at least one inhaler malfunction will be listed.

# 9. REFERENCES

Bime, C., Wei, C., Holbrook, J., Sockrider, M., Revicki, D. and Wise, R. Asthma Symptom Utility Index: Reliability, validity, responsiveness, and the minimal important difference in adult asthmatic patients. *Journal of Allergy and Clinical Immunology*. 2012; 130(5):1078-1084.

Carpenter, JR, Roger, J, and Kenward, MG. Analysis of longitudinal trials with missing data: A framework for relevant, accessible assumptions, and inference via multiple imputation. *Journal of Biopharmaceutical Statistics* 2013;23:1352–71.

Cohen J, Mann D, Wisnivesky J. Assessing the validity of self-reported medication adherence among inner-city asthmatic adults: The Medication Adherence Report Scale for Asthma. *Annals of Allergy Asthma Immunology*. 2009 Oct;103(4):325-31.

Firth D. Bias Reduction of Maximum Likelihood Estimates. Biometrika. 1993;80:27–38.

GlaxoSmithKline Document Number 2016N307903\_01: Study 207040; An open label, randomised, parallel group clinical study to evaluate the effect of the Connected Inhaler System (CIS) on adherence to Relvar/Breo ELLIPTA therapy, in asthmatic participants with poor control.

Hibbard J, Stockard J, Mahoney R, and Tusler M. Development of the Patient Activation Measure (PAM): Conceptualizing and Measuring Activation in Patients and Consumers. *HSR: Health Services Research* 2004; 39:4, Part I

Jones P, Francis H, Quirk H et al. A Self-Complete Measure of Health Status for Chronic Airflow Limitation; The St. George's Respiratory Questionnaire. *American Review of Respiratory Disease* 1992; 145:1321-1327

Nathan R, Sorkness C, Kosinski M et al. Development of the asthma control test: A survey for assessing asthma control. Journal of Allergy and Clinical Immunology. Volume 113, Issue 1, January 2004, Pages 59–65

Revicki D A, Leidy N K, Et al. Integrating patient preferences into health outcomes assessment: The multivariable Asthma Symptoim Utility Index. Chest. 1998;114:998-1007.

Schatz M, Kosinski M, Yarlas AS, Hanlon J, Watson ME, Jhingran P. The minimally important difference of the Asthma Control Test, The Journal of allergy and clinical immunology (2009)

# 10. APPENDICES

# 10.1. Appendix 1: Schedule of Activities

# 10.1.1. Protocol Defined Schedule of Events

| Procedures | Screen | Run-In | 1 | | | 1 | reatme | nt Perio | d | | EW | Follow<br>-up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit/Contact | V1 | V2 | V3 | V4 | V5 | V6 | <b>V</b> 7 | V8 | V9 | V10 | | V11 | Conditional Visits: V3 & V4 are only required if a |
| Month of Study | -1 | 0 | 0 | 0 | 1 | 2 | 3 | 4 | 5 | 6 | | | participant is not included at prior run in visit. |
| Day of Study | -28 | 0 | 0 | 0 | 28 | 56 | 84 | 112 | 140 | 168 | | 175 | V6, V7, V8 & V9 are only required for Treatment |
| Visit Window (days) | | ±2 | ±2 | ±2 | ±2 | ±7 | ±7 | ±7 | ±7 | ±7 | | ±2 | arms 1 & 3. Randomisation to treatment arms will |
| Conditional Visits | | | Х | Х | | Х | Х | Х | Х | | | | occur at Visit 2,3 or 4 when randomisation criteria have been met |
| SCREENING ASSESSMENT | TS | • | - | • | - | • | • | • | • | * | - | - | |
| Written Informed Consent | Х | | | | | | | | | | | | Signed by the participant and HCP/ designee prior to any other study assessments. May be completed at a separate visit to screening if required. |
| Participant Demography | Х | | | | | | | | | | | | |
| Medical History | Х | | | | | | | | | | | | |
| Asthma History | Х | | | | | | | | | | | | Including exacerbation history for previous 12 months and those involving hospitalisation |
| Therapy History | Х | | | | | | | | | | | | Maintenance therapy over previous 12 months, including number of prescriptions requested or provided |
| Physical Exam | Х | | | | | | | | | | | | Full physical including height, weight and vital signs |
| Inclusion/Exclusion<br>Criteria | Х | Х | Х | Х | | | | | | | | | ACT assessment for inclusion required at run-in visits |
| Randomisation | | Х | Х | Х | | | | | | | | | Participant randomised to treatment at only one of V2, V3 or V4 once ACT criteria is met |

| Procedures | Screen | Run-In | 1 | | | Ţ | reatme | nt Perio | d | | EW | Follow<br>-up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit/Contact | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | V10 | | V11 | Conditional Visits: V3 & V4 are only required if a |
| Month of Study | -1 | 0 | 0 | 0 | 1 | 2 | 3 | 4 | 5 | 6 | | | participant is not included at prior run in visit. |
| Day of Study | -28 | 0 | 0 | 0 | 28 | 56 | 84 | 112 | 140 | 168 | | 175 | V6, V7, V8 & V9 are only required for Treatment |
| Visit Window (days) | | ±2 | ±2 | ±2 | ±2 | ±7 | ±7 | ±7 | ±7 | ±7 | | ±2 | arms 1 & 3. Randomisation to treatment arms will |
| Conditional Visits | | | Х | Х | | Х | Х | Х | Х | | | | occur at Visit 2,3 or 4 when randomisation criteria have been met |
| SAFETY ASSESSMENTS | | | | | | | | | | | | | |
| Concomitant Medication | | | | | | Х | | | | | | | |
| Urine Pregnancy Test | Χ | Х | Х | Х | Х | | | | | Х | Х | | |
| SAEs | Х | | • | • | • | • | Х | • | | | • | | |
| Non-Serious Adverse<br>Events that leads to<br>withdrawal | Х | | | | | | | | | Non-serious adverse events that leads to dose modification, drug discontinuation, or withdrawal from the trial. Collected from start of run in | | | |
| Non-serious Adverse<br>Drug Reactions | Х | | | | | | Х | | | | | | Collected from start of run in |
| Exacerbations | Х | | | | | | Χ | | | | | | Severe Exacerbation are to be reviewed and recorded. Collected from start of run in |
| Unscheduled HCP visits | | | | | | | Х | | | | | | All secondary care contacts and all primary care contacts related to Asthma |
| QUESTIONNAIRES & Patie | nt Reporte | d Outcor | nes (PR | Os) (Pei | formed | in the o | order gi | ven her | e) | | | | |
| ACT | Х | Х | Х | Х | Х | | | | | Х | Х | | ACT performed at V2, V3 or V4 to confirm inclusion for randomisation |
| ASUI | <b>X</b> 1 | <b>X</b> <sup>2</sup> | <b>X</b> <sup>2</sup> | <b>X</b> <sup>2</sup> | Х | | | | | Χ | Х | | PRO's only performed at screening once a |
| SGRQ | | <b>X</b> 2 | <b>X</b> 2 | <b>X</b> 2 | Х | | | | | Χ | Х | | participant is included. 2. The PRO's are only performed at the run-in visit (V2, V3 or V4) if a participant is randomised to treatment |
| PAM | <b>X</b> 1 | <b>X</b> <sup>2</sup> | <b>X</b> <sup>2</sup> | <b>X</b> <sup>2</sup> | Χ | | | | | Χ | Χ | | |
| MARS-A | <b>X</b> 1 | <b>X</b> <sup>2</sup> | <b>X</b> <sup>2</sup> | <b>X</b> <sup>2</sup> | Х | | | | | Χ | Χ | | |
| BMQ | <b>X</b> 1 | <b>X</b> <sup>2</sup> | <b>X</b> 2 | <b>X</b> 2 | Х | | | | | Χ | Х | | |
| EXIT Questionnaire | | | | | | | | | | Χ | Х | | |

| Procedures | Screen | Run-In | 1 | | | T | reatme | nt Perio | d | | EW | Follow<br>-up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit/Contact | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | V10 | | V11 | Conditional Visits: V3 & V4 are only required if a |
| Month of Study | -1 | 0 | 0 | 0 | 1 | 2 | 3 | 4 | 5 | 6 | | | participant is not included at prior run in visit. |
| Day of Study | -28 | 0 | 0 | 0 | 28 | 56 | 84 | 112 | 140 | 168 | | 175 | V6, V7, V8 & V9 are only required for Treatment |
| Visit Window (days) | | ±2 | ±2 | ±2 | ±2 | ±7 | ±7 | ±7 | ±7 | ±7 | | ±2 | arms 1 & 3. Randomisation to treatment arms will |
| Conditional Visits | | | Х | Х | | Х | Х | Х | Х | | | | occur at Visit 2,3 or 4 when randomisation criteria have been met |
| Exit Interview | | | | | | | | | | Х | Х | Х | Interview is for sub-set of participants who agree to take part and can be performed at V10 or V11 for logistical reason. There is a 14 day window for vendor to schedule and conduct exit interviews. |
| ASSESSMENTS | _ | - | - | | - | | - | - | | | _ | - | |
| Fractional exhaled Nitric Oxide (FeNO) | <b>X</b> <sup>1</sup> | <b>X</b> <sup>2</sup> | <b>X</b> <sup>2</sup> | X <sup>2</sup> | Х | | | | | Х | Х | | 1.PEF & FeNO only performed once a participant is included. |
| Peak Expiratory Flow<br>(PEF) | <b>X</b> 1 | <b>X</b> <sup>2</sup> | <b>X</b> <sup>2</sup> | <b>X</b> <sup>2</sup> | Х | | | | | Х | Х | | 2.PEF and FeNO is only performed at the Run-in visit if a participant is randomised FeNO performed prior to PEF |
| HCP dashboard review | | | | | Х | Х | Х | Х | Х | Х | | | Participants in treatment arms 1 and 3 only. HCP will record action and outcome of review. |
| INVESTIGATIONAL PRODU | JCT | | | | | | | | | | | | |
| Dispense Sensors | Х | | | | | | | | | | | | Sensors must be attached and switched on in clinic. |
| Dispense Relvar/Breo<br>ELLIPTA | Х | | • | | Х | | • | • | • | | | | All participants will attend independent dispensing visits to collect their next Relvar/Breo ELLIPTA |
| Dispense Salbutamol MDI | Х | require visits. | | | | | | and/or salbutamol MDI as required. Patients are required to bring the sensor to the dispensing visits. The sensor will be attached to the new device and switched on at the dispensing visit. | | | | | |
| Training in CIS | Х | Х | X | X | X | | | | | | | | Participants are trained in fitting the sensors at screening. Following randomisation, participants will be trained in CIS as relevant for their treatment arm. Retraining can be provided at V5. |

| Procedures | Screen | Run-In | ١ | | | ī | reatme | nt Perio | d | | EW | Follow<br>-up | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit/Contact | V1 | V2 | V3 | V4 | V5 | V6 | <b>V</b> 7 | V8 | V9 | V10 | | V11 | Conditional Visits: V3 & V4 are only required if a |
| Month of Study | -1 | 0 | 0 | 0 | 1 | 2 | 3 | 4 | 5 | 6 | | | participant is not included at prior run in visit. |
| Day of Study | -28 | 0 | 0 | 0 | 28 | 56 | 84 | 112 | 140 | 168 | | 175 | V6, V7, V8 & V9 are only required for Treatment |
| Visit Window (days) | | ±2 | ±2 | ±2 | ±2 | ±7 | ±7 | ±7 | ±7 | ±7 | | ±2 | arms 1 & 3. Randomisation to treatment arms will |
| Conditional Visits | | | Х | X | | X | X | Х | X | | | | occur at Visit 2,3 or 4 when randomisation criteria have been met |
| Training in ELLIPTA & MDI correct use | Х | | | | Х | | | | | | | | Once included a participant should be trained in correct use of ELLIPTA and MDI devices |
| Correct Use Assessment for ELLIPTA and MDI | Х | | | | Х | | | | | | | | Inhaler use technique will be assessed for correct use. This need only be recorded in source. |
| Return Sensors | | | | | | | | | | Х | Х | | · |
| Return Relvar/Breo<br>ELLIPTA | | | | | | X | | | | | Х | | Patients are required to return their devices at the independent dispensing visits. Doses remaining on each returned ELLIPTA inhaler will be recorded. |
| Return Salbutamol MDI | | | | | | Χ | | | | | Χ | | Patients to return used MDI at dispensing visits. |

# 10.2. Appendix 2: Assessment Windows

#### 10.2.1. General

Clinic visits are scheduled to take place as specified in Appendix 1: Schedule of Activities. Individual measurements will be reported based on the visits they are assigned to in the study database without adjustment. Measurements outside visit windows will not be excluded from analyses.

If a circumstance should arise where multiple measurements have been collected and recorded against the same timepoint, then the first valid value will be used for that timepoint.

The maximum value obtained from the multiple PEF and FeNO assessments at a visit will be used in summaries and analyses. Participants who withhold a daily dose of maintenance therapy and rescue medication for 6 hours prior to the assessment will have value included in the summaries.

# 10.2.2. Definitions of Assessment Windows for Adherence and Rescue Medication Use Analyses

All participants have a sensor on their maintenance and rescue medication to consistently measure their adherence to maintenance and level of rescue medication use in the study. The sensors are attached to participants ELLIPTA Relvar/Breo maintenance treatment and MDI rescue medication from start of Visit 1 until Visit 10. The sensors record the time and date when the Relvar/Breo ELLIPTA cover is opened and closed and the salbutamol MDI rescue medication is actuated.

Study day 1 is defined as the day of randomisation. This could be the day of Visit 2, 3 or 4, dependent on the length of the run-in period. Study day for all other visits, assessments and events are calculated relative to this.

The following information in Table 5 displays which sensor records are summarised for each analysis time period (Analysis Month). Any sensor data recorded post the Month 6 (day 168) time period will not be included in the analysis of ELLIPTA adherence or salbutamol MDI rescue medication use of sensor data.

 Table 5
 Sensor Data Assessment Windows

| Sensor Data Assessment Windows | | |
|---|---|---|
| Analysis | Analysis Po | eriod |
| Month | Beginning Timepoint | Ending Timepoint |
| Baseline | Latest of either Day -28 or day after Visit 1 (minimum of 14 days must be present to create a baseline) | Day -1<br>(Day prior to randomisation) |
| 1 | Day 1<br>(Day of randomisation) | Day 28 or discontinuation from adherence/rescue assessment if within month 1 |
| 2 | Day 29 | Day 56 or discontinuation from adherence/rescue assessment if within month 2 |
| 3 | Day 57 | Day 84 or discontinuation from adherence/rescue assessment if within month 3 |
| 4 | Day 85 | Day 112 or discontinuation from adherence/rescue assessment if within month 4 |
| 5 | Day 113 | Day 140 or discontinuation from adherence/rescue assessment if within month 5 |
| 6 | Day 141 | Earliest of either day of visit 10, Day 168 or discontinuation from adherence/rescue assessment if within month 6 if participant is a completer OTHERWISE Day 168 or discontinuation from adherence/rescue assessment if within month 6 |

Note: 'Discontinuation from adherence/rescue assessment' occurs at the earliest of premature discontinuation from use of the ELLIPTA /MDI sensor, premature discontinuation of ELLIPTA (for adherence measures), or premature withdrawal from the study.
# 10.3. Appendix 3: Study Phases and Treatment Emergent Adverse Events

## 10.3.1. Study Phases

Since participants are on Relvar/Breo study treatment from the time they enter run-in, assessments and events will be classified according to time of occurrence relative to the randomisation date and last stop date of Relvar/Breo treatment. The randomisation and latest exposure treatment stop dates will be used to determine whether an assessment or event was during pre-screening treatment, run-in treatment, on-treatment or post-treatment. If it is not possible to tell whether an assessment or event was on-treatment or not, it will be considered as on-treatment.

### 10.3.1.1. Study Phases for Concomitant Medication

A medication will be summarised in every study phase (pre-screening, run-in, on- or post-treatment) in which it was taken, so a medication that was started during the run-in period and stopped during the post-randomisation treatment period will appear in both the run-in-treatment and the on-treatment summaries.

On-treatment will be considered to be from the day of randomisation to treatment arm until the last (Relvar/Breo) treatment stop date. Post-treatment will be considered to be from the day after the last treatment stop date and onward. Run-in-treatment will be considered from the screening visit until prior to randomisation to treatment arm date. If a participant's last treatment stop date is missing, this will be assumed to the date of the last recorded on-treatment visit up to Visit 10 (not including the Follow-up visit) or the return of the last Relvar/Breo container, whichever is later.

| Study Phase | Definition |
|---|---|
| Pre-Screening<br>Treatment | Date of Medication < Screening Visit Date |
| Run-in Treatment | (Date of Medication ≥ Screening Visit date) and (Date of Medication < Randomisation Date) |
| On-Treatment | (Date of Medication ≥ Randomisation Date) and (Date of Medication ≤ Last Treatment Stop Date) |
| Post-Treatment | Date of Medication > Last Treatment Stop Date |

# 10.3.1.2. Study Phases for Asthma Exacerbations

| Study Phase | Definition |
|---|---|
| Run-in-Treatment | (Exacerbation Onset Date ≥ Screening Visit date) and (Exacerbation Onset Date < |
| | Randomisation Date) |
| On-Treatment | (Exacerbation Onset Date ≥ Randomisation Date) and (Exacerbation Onset Date ≤ |
| | Last Treatment Stop Date)+1 |
| Post-Treatment | Exacerbation Onset Date > Last Treatment Stop Date+1 |

# 10.3.1.3. Treatment Emergent Flag for Adverse Events

| Study Phase | Definition |
|---|---|
| Run-in-<br>Treatment* | (AE Start Date ≥ Screening Visit date) and (AE Start Date < Randomisation Date) |
| On-Treatment | (AE Start Date ≥ Randomisation Date) and (AE Start Date ≤ Last Treatment Stop Date)+1 |
| Post-Treatment | AE Start Date > Treatment Stop Date + 1 |
| Onset Time Since<br>First Dose (days)* | <ul> <li>Time Since First Dose will be derived as followed:</li> <li>If Randomisation Date or AE Onset Date are missing =&gt; missing</li> <li>If Randomisation Date &gt; AE Onset Date then =&gt; AE Onset Date – Randomisation Date</li> <li>If Randomisation Date ≤ AE Onset Date then =&gt; AE Onset Date – Randomisation Date + 1</li> </ul> |

<sup>\*</sup>For participants who enter the run-in treatment phase but do not get randomised, use the last run-in date instead of randomisation date for the "Run-in-Treatment" phase and "Onset Time Since First Dose (days)" as the participants would not have a randomisation date.

# 10.4. Appendix 4: Data Display Standards & Handling Conventions

# 10.4.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | uksal1x00175 |
| HARP Compound | arenv/arprod/gw685698_gw642444/mid207040/final_01 |
| Analysis Datasets | |
| <ul> <li>Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 &amp; ADaM IG<br/>Version 1.0). If the Study Data Standardization Plan (SDSP) exists for a study, ensure the CDISC<br/>versions are consistent.</li> </ul> | |
| Generation of RTF Files | |
| Rich Text Format | Rich Text Format (RTF) files will be generated for final reporting effort. |

#### 10.4.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

All data displays (Tables, Figures & Listings) will use the term "Subject" which reflects CDISC and GSK Data Display Standards terminology

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.
- All data will be reported according to the treatment the participant was randomised to unless otherwise stated.
- Numeric data will be reported (in listings) at the precision collected in the eCRF or recorded in the raw dataset if from non-eCRF sources.

| Specification of Number of Decimal Places for Descriptive Statistics | | |
|---|---|---|
| Label | Description | Number of decimal places (dp) more than raw data |
| N | Number of participants in the treatment group | Always present to 0 dp |
| n | Number of participants with non-<br>missing values | Always present to 0 dp |
| Mean | Arithmetic Mean | 1 dp |

| | I a | Ι |
|---|---|---|
| SD | Standard Deviation | 2 dp |
| Median | Median | 1 dp |
| Min. | Minimum | 0 dp |
| Max. | Maximum | 0 dp |
| Specification of Number of Decin | nal Places for Statistical Analysis | |
| Label | Description | Number of decimal places (dp) more than raw data |
| LS Mean | Adjusted mean for the treatment group | 1 dp |
| LS Mean Change | Adjusted mean change from baseline for the treatment group | 1 dp |
| Std Err | Standard error | 2 dp |
| Difference | Treatment difference | 1 dp |
| Odds Ratio | Treatment odds ratio | Always present to 2 dp |
| Relative Risk | Treatment relative risk | Always present to 2 dp |
| 95% CI | 95% Confidence interval around difference/ratio/relative risk | Same number of dp as the difference/ratio/relative risk |
| p-value | p-value | Always present to 3 dp<br>(or <0.001 or >0.999) |

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to treatment dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the participant's listings.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables and/or figures.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Craphical Diaplaya | |

#### **Graphical Displays**

- Refer to IDSL Statistical Principals 7.01 to 7.13.
- The programs for statistical analysis tables will create SAS datasets with the unrounded numbers from
  the statistical models to be used in any graphs. This will include all LS means, standard errors,
  treatment differences or ratios and confidence intervals. This will be done for all analysis tables
  regardless of whether or not a figure is planned as part of statistical analysis complete (SAC).
- The programs for all graphical displays will additionally create a CSV file with the final data that is used in the graph in order to allow the graph to be redrawn for any potential future publication requirement

### 10.5. Appendix 5: Derived and Transformed Data

#### 10.5.1. General

#### Study Day

- Calculated as the number of days from first randomisation:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Randomisation Date → Study Day = Ref Date Randomisation Date
  - Ref Date ≥ Randomisation Date → Study Day = Ref Date (Randomisation Date) + 1

#### **Change from Baseline**

 Calculated as the difference between the value of the endpoint at the timepoint of interest and the baseline value as defined in Section 5.2 Baseline Definitions

#### **Time Since First Dose**

- Calculated as the number of days from first dose date of post randomisation treatment:
  - Ref Date = Missing → Time Since First Dose = Missing
  - Ref Date < Randomisation Date → Time Since First Dose = Ref Date Randomisation Date</li>
  - Ref Date ≥ Randomisation Date → Time Since First Dose = Ref Date (Randomisation Date) +1

#### **Study Treatment Start and Stop Dates**

- In this study, participants who permanently discontinue Relvar/Breo study treatment, any sensors or the App may continue in the study attending the remaining visits and completing the scheduled assessments.
- Data displays will state if pre-screening, run-in treatment, on-treatment, post-treatment, or both ontreatment and post-treatment data are included in the summary or analysis, when applicable. Ontreatment is defined as Relvar/Breo study treatment from the date of randomisation to treatment arm.
- Relvar/Breo on-treatment start date will be defined as the randomisation date and Relvar/Breo
  Treatment Stop Date will be defined as the latest treatment stop date (from the study treatment
  compliance eCRF log and treatment discontinuation eCRF page). These dates will be used to
  determine whether a measurement is run-in, on or post-treatment. (See Section 10.3.1 Study Phases).

#### Multiple Measurements at One Analysis Time Point

 PEF and FeNO assessments are performed multiple times per visit. The maximum value obtained at the visit will be included in summaries of these data.

### 10.5.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any participant with a missing day will have this imputed as day '15'.
  - Any participant with a missing date and month will have this imputed as PPD

#### **Demographics**

- Birth date will be presented in listings as 'YYYY'.
- Completely missing dates of birth will remain as missing, with no imputation applied. Consequently, the age of the participant will not be calculated and will remain missing.
- Age, in whole years, will be calculated with respect to the date of screening (Visit 1).

#### **Body Mass Index**

Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

#### Race

- The five high level Food and Drug Administration (FDA) race categories and designated Asian subcategories are:
  - 1. African American/African Heritage
  - 2. American Indian or Alaska Native
  - 3. Asian
    - a. Central/South Asian Heritage
    - b. Japanese/East Asian Heritage/South East Asian Heritage
    - c. Mixed Asian Heritage (only required if data exists)
  - 4. Native Hawaiian or other Pacific Islander
  - 5. White
- These categories and subcategories will be summarized along with all combinations of high level categories which exist in the data. All five of the high level race categories and the two Asian subcategories must appear on the display even if there are no participants in a particular category, but combinations that do not exist in the data do not need to be represented. Combinations will be represented as the concatenation of the high level category terms, e.g., "White & Asian." The designated Asian subcategories will not be summarized as combinations with other categories.
- In addition, the standard race categories collected per IDSL will be summarized along with categories for mixed race. The categories are:
  - 1. African American/African Heritage
  - 2. American Indian or Alaska Native
  - 3. Asian Central/South Asian Heritage
  - 4. Asian East Asian Heritage
  - 5. Asian Japanese Heritage
  - 6. Asian South East Asian Heritage
  - 7. Asian Mixed Race
  - 8. Native Hawaiian or other Pacific Islander
  - 9. White Arabic/North African Heritage
  - 10. White White/Caucasian/European Heritage
  - 11. White Mixed Race
  - 12. Mixed Race
- "Asian Mixed Race" is only used if more than one Asian category is selected, but no non-Asian
  races. Similarly, "White Mixed Race" is only used if both of the White categories are selected, and no
  non-White races. If multiple races of different types are selected, then the overall "Mixed Race"
  category is used.
- A participant will only be represented in a single category. A participant who selects a combination of
  races will be counted as "Asian Mixed Race," "White Mixed Race," or "Mixed Race," but not in
  each of the constituent terms. Therefore, the counts will add up to the total number of participants with
  a response, and the percentages will add to 100%.

#### **Treatment Compliance**

- Relvar/Breo treatment compliance, calculated as a percentage, will be based on the total number of inhalations taken from the study drug inhaler(s) and the expected number of inhalations to be taken.
- The expected number of inhalations will be derived as the expected number of inhalations per day (1 for OD dosing) multiplied by the number of days on study drug based on treatment start date and treatment stop date.
- The total number of inhalations taken will be based on the dose counters of the inhalers, which are resupplied during the study. If there is no dose counter information at all then the compliance will be missing, however, as long as the information from one dose counter is present, treatment compliance will be calculated. If a dose counter start count is missing then it will be assumed to be 30. All inhalers dispensed will be used, provided the dose counter stop counts are non-missing.
- Treatment compliance will be calculated based on the formula:

$$Compliance = \left(\frac{\textit{Total \_Number\_of \_Inhalations \_Taken}}{\textit{Expected \_Inhalations} \times (\textit{Stop \_Date} - \textit{Start \_Date} + 1)}\right) \times 100$$

where *Total\_Number\_of\_Inhalations\_Taken* is the total number of doses taken from all inhalers, *Expected\_Inhalations* is equal to 1 and *Start\_Date* and *Stop\_Date* are the earliest treatment start date on or post randomisation and the latest treatment stop date recorded for all the inhalers used in the calculation.

#### **Extent of Exposure and Study Duration**

- Relvar/Breo on-treatment start date will be defined as the randomisation date and Relvar/Breo Treatment
  Stop Date will be defined as the latest treatment stop date (from the study treatment compliance eCRF
  log and treatment discontinuation eCRF page) for the participant. These dates will be used to determine
  whether a measurement is run-in, on or post-treatment. (See Section 10.3.1 Study Phases). Study
  conclusion is defined as completion or withdrawal, as applicable.
- Duration of exposure to study drug will be calculated as:
  - Duration of Exposure (days) = Treatment Stop Date Randomisation Date + 1
- Duration of post-treatment time spent in the study will be calculated as:
  - Duration of Post-Treatment Study Time (days) = Study Conclusion Date Treatment Stop Date
- Duration of total time spent in the study will be calculated as:
  - Duration of Study Time (days) = Study Conclusion Date Randomisation Date + 1
- Years exposed will be calculated as:
  - Last treatment stop date Randomisation Date +1 / 365.25.
  - o Total Years Exposed will be the sum of the year exposed per treatment arm.

# 10.5.3. Efficacy

#### 10.5.3.1. ELLIPTA Device Sensor Assessments

# Percentage of ELLIPTA doses taken (daily adherence) Endpoint

#### **Overview of Calculation**

- 1. Create a dataset (Observed Data A) to calculate the monthly <u>observed</u> percentage of ELLIPTA adherence values (from month 1 to month 6) accounting for the following,
  - a. number of days adherent to ELLIPTA (as prescribed)
  - b. number of days post ELLLIPTA maintenance sensor permanent discontinuation
  - c. the intermittent missing daily adherence data due to device incident.
  - d. Non-adherent days (i.e. none of the above and those days with more than one dose in 24-hour period).

- 2. Duplicate the observed monthly adherence values dataset (Observed Dataset A). Using the values in the duplicate dataset (Dataset B), impute the month where the sensor was permanently discontinued before the end of that month (and therefore presents a monthly adherence rate based on partly observed sensor data for that month) as missing unless the participant is a study completer.
- 3. Using each of the two observed datasets (Observed Dataset A and Observed Dataset B), create four separate imputed datasets (J2R-Dataset A, J2R-Dataset B, MAR-Dataset A, MAR-Dataset B) that account for the two imputation methods (J2R or MAR) that may be applied to participants' data after discontinuation of the maintenance sensor, ELLIPTA or withdrawal from study. Imputation will be carried out using observed monthly adherence rates for months 1 to 6. 1000 draws will be used. Completely missing intermediate monthly values will be assumed MAR. The multiple imputation will be implemented using the methods described in Carpenter, 2013, using the macros (Part1A, Part1B, Part2A and Part2B) available from <a href="https://missingdata.lshtm.ac.uk/2017/04/06/gsk-five-macros/using-seeds-documented-in-the-RAP">https://missingdata.lshtm.ac.uk/2017/04/06/gsk-five-macros/using-seeds-documented-in-the-RAP for the respective endpoint.</a>
- 4. The Observed Datasets (A and B), imputed datasets (J2R-Dataset A, J2R-Dataset B, MAR-Dataset A, MAR-Dataset B) and the timing of the intercurrent events; permanent discontinuation of the ELLIPTA maintenance sensor; permanent discontinuation of ELLIPTA treatment and withdrawal from study; will be used to create an analysis dataset (Dataset C) that identifies the proportion of each month to be assigned as observed data, J2R imputed data, MAR imputed data, or no data. The strategy for handling intercurrent events is described in Section 7.1.4 Strategy for Intercurrent (Post-Randomisation) Events.

Within each imputation draw, for each missing month, the observed and any imputed data will be combined to provide a percentage adherence value. The values for months 4 to 6, months 1-3 and months 1-6, will be combined to create the value for the respective primary and secondary endpoint analyses and the weight to be assigned to each participant.

- 5. Analyse using Multiple Imputation macro Part3
  - a. Perform ANCOVA on the endpoint for each imputed dataset to obtain treatment effect estimate and standard error
  - b. Combine estimates across imputations using Rubin's rules

The intercurrent events identified as part of the primary endpoint estimand and derivation are detailed in full in Section 7.2.1.3 Strategy for Intercurrent (Post-Randomisation) Events. Below are two schematics of the intercurrent event patterns and their estimation rules.

#### **Intercurrent Event Patterns**



#### Intercurrent Event 'Estimation Rules' 1-4



No data if withdrawal related to ELLIPTA; J2R imputation if withdrawal related to CIS; MAR imputation if withdrawal not related to ELLIPTA or CIS

#### Intercurrent Events related to Relvar/Breo or CIS

In order to implement the intercurrent event strategy detailed in Section 7.1.4 Strategy for Intercurrent (Post-Randomisation) Events, it is necessary to determine if and when the reasons for permanent discontinuations related to CIS or ELLIPTA Relvar/Breo treatment occur.

The date and reason for permanently withdrawing from ELLIPTA treatment will be determined from the study treatment (Relvar/Breo ELLIPTA) discontinuation page of the eCRF.

ELLIPTA discontinuation reasons classified as not related to ELLIPTA are as follows:

- AE not treatment related (determine from the AE that lead to withdrawal to treatment if study treatment related, on the AE eCRF page)
- Protocol deviation not related to study treatment
- Participant reached protocol defined stopping criteria not related to study treatment
- Study closed/terminated
- Lost to follow-up
- Investigator discretion not related to study treatment
- Decision by participant or proxy not related to study treatment

ELLIPTA discontinuation reasons classified as related to ELLIPTA are as follows:

- AE treatment related (determine from the AE that lead to withdrawal to treatment if study treatment related, on the AE eCRF page)
- Lack of efficacy
- Protocol deviation related to study treatment
- Participant reached protocol defined stopping criteria (except pregnancy) related to study treatment
- Investigator discretion related to study treatment
- Decision by participant or proxy related to study treatment

The date and reason for withdrawing from the study will be determined from the study conclusion page of the eCRF.

Study discontinuation reasons classified as related to CIS are as follows:

Withdrew consent – dissatisfaction with the connected inhaler system (CIS)

#### Monthly Percentage of ELLIPTA doses taken (daily adherence) - Calculation

STEP 1: Creating the observed adherence dataset (Observed Dataset A)

To determine the monthly <u>observed</u> percentage of ELLIPTA adherence values (Observed Dataset A) the following should be applied for each month:

For Baseline Analysis Month, for each participant create a count of each of the following types of Days

- D1 = Adherence recorded
- D2 = Device incident
- D3 = Post discontinuation of maintenance Sensor
- D4 = Non-adherent (including those imputed as non-adherent)
  - D5=D1 + D2 + D3 + D4, i.e. The total number of days within the Baseline Analysis Month; the total number of days between Beginning Timepoint and Ending Timepoint as defined in Table 5 in Section 10.2 Appendix 2: Assessment Windows.

For Analysis Month 1, 2, 3, 4 and 5, for each participant create a count of each of the following types of days:

- D1 = Adherence recorded
- D2 = Device incident
- D3 = Post discontinuation of maintenance Sensor
- D4 = Non-adherent (including those imputed as non-adherent)
- D5 = D1 + D2 + D3 + D4, i.e. The total number of days within the Analysis Month; the total number of days between Beginning Timepoint and Ending Timepoint as defined in Table 5 in Section 10.2 Appendix 2: Assessment Windows.

For Analysis Month 6, for each participant create a count of each of the following types of days:

- D1 = Adherence recorded
- D2 = Device incident
- D3 = Post discontinuation of maintenance sensor
- D4 = Non-adherent (including those imputed as non-adherent)
- D5 = D1 + D2 + D3 + D4, i.e. the total number of days within Analysis Month 6; the total number of days between Beginning Timepoint and Ending Timepoint as defined in Table 5 in Section 10.2 Appendix 2: Assessment Windows.

The following observations from the sensor and eCRF will be required to determine the above Days and the differences between missing at random due to device/sensor incident and non-adherent days.

- Device malfunction date
- Sensor malfunction date
- Permanent discontinuation of maintenance sensor
- First and last individual sensor synchronisation dates

The first and last individual sensor synchronisation dates will be provided in the sensor dataset. These dates will be used to assess whether missing observations are due to non-adherent days or data being missing at random due to device/sensor malfunction.

For each Analysis Month, the Observed adherence for that month will be calculated as follows:

Monthly observed maintenance adherence (%) =  $\left(\frac{D1}{D5 - D2 - D3}\right) \times 100$ 

#### STEP 2: Creating the modified observed adherence dataset (Observed Dataset B)

The Observed Dataset A will be duplicated. Using the values in the duplicate dataset (Observed Dataset B) the Analysis Month where the maintenance sensor was permanently discontinued before the end of that month (and therefore presents a monthly adherence rate based on partly observed sensor data for that month) will be imputed as missing; i.e.in Dataset B, if within an Analysis Month (D3>0 and D3<D5) then set monthly value for that Analysis Month to missing. (Note: unless the participant is a completer in which case do not set the value to missing for that Analysis Month)

#### STEP 3: Creating the reference imputed datasets under MAR and J2R method

Using each of the two observed datasets (Observed Dataset A and Observed Dataset B) monthly values, create four separate reference imputed datasets (J2R-Dataset A, J2R-Dataset B, MAR-Dataset A, MAR-Dataset B) that account for the two imputation methods (J2R or MAR). Completely missing intermediate monthly values will be assumed MAR.

The multiple imputation will be implemented using the methods described in Carpenter, 2013 using macros, Part1A, Part1B, Part2A and Part2B (available from

https://missingdata.lshtm.ac.uk/2017/04/06/gsk-five-macros/). The seeds are documented at the end of Section 10.5.3.1. and 1000 draws will be used in the relevant macros parameters.

Due to the range of the monthly adherence percentages being limited between 0 and 100, the multiple imputation process can generate percentages outside the possible range of values (< 0% or > 100%). A cap will be put in place where values imputed < 0 will be set as 0 and values imputed as > 100 set as 100.

#### STEP 4: Creating the Monthly Analysis values dataset

For each month within each participant create a count of each of the following durations based on intercurrent events: Let,

m1 = maintenance sensor still in use

m2 = maintenance sensor discontinued, but ELLIPTA Relvar/Breo not discontinued

m3 = ELLIPTA Relvar/Breo discontinued (includes days post withdrawal from the study). Note, if participant is a completer then for Analysis Month 6, m3=0.

m4 = m1 + m2 + m3

Calculate the proportion of days the sensor was still in use from the total number of days ELLIPTA was in use within a month, m1/(m1+m2)

Calculate the proportion of days the sensor was discontinued from the total number of days ELLIPTA was in use within a month, m2/(m1+m2)

Set participants monthly values to observed, MARA, MARB, J2RA, J2RB imputation, no data each with an m1, m2, m3 and m4 duration.

Examples include to following;

 A participant who prematurely discontinues sensor after 15 days of Analysis Month 5 and concurrently discontinues ELLIPTA maintenance therapy and study withdrawal after 10 days of Analysis Month 6

| Subject<br>Id | Draw | Month | Α | В | J2RA | J2RB | MARA | MARB | m1 | m2 | m3 | m4 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| X | 1 | 1 | 77 | 77 | 77 | 77 | 77 | 77 | 28 | 0 | 0 | 28 |
| Х | 1 | 2 | 82 | 82 | 82 | 82 | 82 | 82 | 28 | 0 | 0 | 28 |
| Х | 1 | 3 | 87 | 87 | 87 | 87 | 87 | 87 | 28 | 0 | 0 | 28 |
| Х | 1 | 4 | 77 | 77 | 77 | 77 | 77 | 77 | 28 | 0 | 0 | 28 |
| Х | 1 | 5 | 71 | | 71 | 77 | 71 | 78 | 15 | 13 | 0 | 28 |
| Χ | 1 | 6 | | | 80 | 79 | 77 | 76 | 0 | 10 | 18 | 28 |

 A participant who concurrently prematurely discontinues sensor, ELLIPTA maintenance therapy and study withdrawal after 15 days of Analysis Month 5

| Subject<br>Id | Draw | Month | Α | В | J2RA | J2RB | MARA | MARB | m1 | m2 | m3 | m4 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Χ | 1 | 1 | 77 | 77 | 77 | 77 | 77 | 77 | 28 | 0 | 0 | 28 |
| Х | 1 | 2 | 80 | 80 | 80 | 80 | 80 | 80 | 28 | 0 | 0 | 28 |
| Х | 1 | 3 | 79 | 79 | 79 | 79 | 79 | 79 | 28 | 0 | 0 | 28 |
| Х | 1 | 4 | 75 | 75 | 75 | 75 | 75 | 75 | 28 | 0 | 0 | 28 |
| Χ | 1 | 5 | 83 | | 83 | 77 | 83 | 79 | 15 | 0 | 13 | 28 |
| Χ | 1 | 6 | | | 77 | 77 | 75 | 80 | 0 | 0 | 28 | 28 |

• A participant who completes the study after 26 days in Analysis Month 6

| Subject<br>Id | Draw | Month | Α | В | J2RA | J2RB | MARA | MARB | m1 | m2 | m3 | m4 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Χ | 1 | 1 | 77 | 77 | 77 | 77 | 77 | 77 | 28 | 0 | 0 | 28 |
| Х | 1 | 2 | 82 | 82 | 82 | 82 | 82 | 82 | 28 | 0 | 0 | 28 |
| Х | 1 | 3 | 87 | 87 | 87 | 87 | 87 | 87 | 28 | 0 | 0 | 28 |
| Х | 1 | 4 | 77 | 77 | 77 | 77 | 77 | 77 | 28 | 0 | 0 | 28 |
| Χ | 1 | 5 | 80 | 80 | 80 | 80 | 80 | 80 | 28 | 0 | 0 | 28 |
| X | 1 | 6 | 82 | 82 | 82 | 82 | 82 | 82 | 15 | 11 | 0 | 26 |

If the sensor is in use for at least a day within a month, m1>0 then let the analysis value be a
combined value (weighted average) of the J2RA observed and J2RB imputed values, by taking a
proportion of each value based on the proportion of days sensor was still in use and discontinued
whilst on ELLIPTA respectively;

Analysis value = m1/m1+m2 x (value from J2RA) + m2/m1+m2 x (value from J2RB) Note the weight is, m1 + m2

Else if the sensor was not used in the month, m1=0 then let the analysis value be the imputed value, Analysis value = value from J2RA dataset (which is the imputed value)

Implement special cases of J2R post-discontinuation of ELLIPTA by identifying participants where ELLIPTA is prematurely discontinued and the participant concurrently withdraws from the study, and ELLIPTA discontinuation reason is not related to ELLIPTA:

• If the sensor is in use for at least a day within a month, m1>0 then let the analysis value be a combined value (weighted average) of the J2RA observed and J2RB imputed values, by taking a proportion of each value based on the proportion of days the sensor is in use and not in use in that month

Analysis value =  $m1/m4 \times (value from J2RA) + (m2+m3)/m4 \times (value from J2RB)$ Note the weight is, m4

• Else if the sensor was not used in the month, m1=0 then let the analysis value be the imputed value, Analysis value = value from J2RA dataset (which is the imputed value)

Implement special case of MAR post-discontinuation of ELLIPTA by identify participants where ELLIPTA is prematurely discontinued and the participant concurrently discontinues the maintenance eSensor and concurrently withdraws from the study, and ELLIPTA discontinuation reason is not related to ELLIPTA and study withdrawal is not related to CIS.

Where ELLIPTA has not been discontinued after the sensor but on the same day, m2=0.

• If the sensor is in use for at least a day within a month, m1>0 then let the analysis value be a combined value (weighted average) of the J2RA observed and MARB imputed values, by taking a proportion of each value based on the proportion of days the ELLIPTA was in use and not in use in that month

Analysis Value = m1/m4 x (value from J2RA) + m3/m4 x (value from MARB)

Else

Analysis Value =  $m1/m4 \times (value from J2RA) + m3/m4 \times (value from MARA)$ 

Note the weights are m4

STEP 5: Primary and Secondary Percentage of ELLIPTA doses taken Endpoints calculation

The calculations presented in the previous steps support the final derivation of the following primary and secondary endpoints, the percentage of ELLIPTA doses taken between

- the beginning of Month 4 and the end of Month 6
- the beginning of Month 1 and the end of Month 6
- the beginning of Month 1 and the end of Month 3

For participants who complete the study treatment (i.e. no premature discontinuation of ELLIPTA Relvar/Breo) during the endpoint period of interest:

Analysis Endpoint is the average of monthly Analysis Values over the number of months in the endpoint period of interest, i.e.

- Month 4 to Month 6
- Month 1 to Month 6
- Month 1 to Month 3

For participants who prematurely discontinue ELLIPTA during the endpoint period of interest for reasons related to ELLIPTA, then the weight is the total duration on ELLIPTA within the endpoint period of interest and applied to each analysis month based on the duration within that month. This weight should be applied to each monthly Analysis value within the period of interest and results summed together to produce the final endpoint/response variable for modelling within macro Part 3.

Note the weight is, total duration of ELLIPTA use within the period of interest . The proportion of weight to apply per monthly Analysis value is m1+m2/total duration of ELLIPTA use within the period of interest

For participants who prematurely discontinue ELLIPTA during the endpoint period of interest for reasons not related to ELLIPTA or CIS, or just related to CIS, the MAR or J2R imputation assumes participants would have continued taking ELLIPTA until the end of the period of interest. The weight is the total duration within the endpoint period of interest. This weight will be applied to each monthly Analysis value within the period of interest and results summed together to produce the final endpoint/response variable for modelling within macro Part 3.

Note the weight is, total expected ELLIPTA duration within the period of interest. The proportion of weight to apply per monthly Analysis value is m1+m2+m3/ Total expected ELLIPTA duration within the period of interest.

### Percentage of ELLIPTA doses taken (daily adherence) - Sensitivity Analysis

Sensitivity analyses will be performed estimating the treatment effect by utilizing a generalized linear model (GLM) and not running the multiple imputation process. The model will follow a binomial distribution with the logit link function.

The sensitivity analyses will be performed for the following primary and secondary endpoints relating to the percentage of ELLIPTA doses taken between

- the beginning of Month 4 and the end of Month 6
- the beginning of Month 1 and the end of Month 6
- o the beginning of Month 1 and the end of Month 3

Model assumptions will be checked by using standardised residual plots. Missing data will be assumed to be MAR.

The weighting strategy is to be applied as detailed above.

#### Percentage of ELLIPTA doses taken (daily adherence) Endpoint

#### **Seeds for Multiple Imputations Macros**

Seeds for all planned MI analyses were determined in advance using the following SAS code and documented within this RAP prior to unblinding:

```
data temp;
```

```
do i = 1 to 6;
    number=round(10000*ranuni(0),1);
    output;
    end;
run;
proc print;
run;
```

#### Part 1B Macro Seed for Parameter Estimation Using Bayesian MCMC Procedure

| Endpoint | Input Dataset | Macro Seed |
|-------------------------------|--------------------|------------|
| Percentage of Daily Adherence | Observed Dataset A | 2124 |
| | Observed Dataset B | 5071 |

| Endpoint | Multiple Imputation Method | Macro Seed | Output Dataset |
|---|---|---|---|
| Percentage of Daily Adherence | MAR | 8517 | MAR Dataset A |
| | J2R | 6888 | J2R Dataset A |
| | MAR | 6388 | MAR Dataset B |
| | J2R | 8674 | J2R Dataset B |

#### 10.5.3.2. MDI Device Sensor Assessments

#### Percentage of Rescue Free Days Endpoint

#### Overview of Calculation

- 1. Create a dataset (Observed Data A) to calculate the monthly <u>observed</u> percentage of MDI rescue free days values (from month 1 to month 6) accounting for the following,
  - a. number of days MDI rescue medication was used (at least once per day)
  - b. number of days post MDI rescue use sensor permanent discontinuation
  - c. the intermittent missing daily MDI rescue use data due to device incident
  - d. MDI Rescue free days (i.e. none of the above).
- 2. Duplicate the observed monthly MDI rescue free values dataset (Observed Dataset A). Using the values in the duplicate dataset (Dataset B), impute the month where the sensor was permanently discontinued before the end of that month (and therefore presents a monthly adherence rate based on partly observed sensor data for that month) as missing unless the participant is a study completer.
- 3. Using each of the two observed datasets (Observed Dataset A and Observed Dataset B), create four separate imputed datasets (J2R-Dataset A, J2R-Dataset B, MAR-Dataset A, MAR-Dataset B) that account for the two imputation methods (J2R or MAR) that may be applied to participants data after discontinuation of the MDI rescue sensor or withdrawal from study. Imputation will be carried out using observed monthly MDI rescue free rates for months 1 to 6. 1000 draws will be used. Completely missing intermediate monthly values will be assumed MAR. The multiple imputation will be implemented using the methods described in Carpenter, 2013, using the macros (Part1A, Part1B, Part2A and Part2B) available from <a href="https://missingdata.lshtm.ac.uk/2017/04/06/gsk-five-macros/">https://missingdata.lshtm.ac.uk/2017/04/06/gsk-five-macros/</a> using seeds documented in the RAP for the respective endpoint.
- 4. The Observed Datasets (A and B), imputed datasets (J2R-Dataset A, J2R-Dataset B, MAR-Dataset A, MAR-Dataset B) and the timing of the intercurrent events; permanent discontinuation of the MDI rescue sensor and withdrawal from study; will be used to create an analysis dataset (Dataset C) that identifies the proportion of each month to be assigned as observed data, J2R imputed data or MAR imputed data. The strategy for handling intercurrent events is described in Section 7.2.2.3 Strategy for Intercurrent (Post-Randomisation) Events.

Within each imputation draw, for each missing month, the observed and any imputed data will be combined to provide a percentage of rescue free days value. The values for months 4 to 6 will be combined to create the value for the respective secondary endpoint analysis and the weight to be assigned to each participant.

5. Analyse using Multiple Imputation macro Part3

- Perform ANCOVA on the endpoint for each imputed dataset to obtain treatment effect estimate and standard error
- b. Combine estimates across imputations using Rubin's rules

The intercurrent events identified as part of this secondary endpoint estimand and derivation are detailed in full in Section 7.2.2.3 Strategy for Intercurrent (Post-Randomisation) Events. Below are two schematics of the intercurrent event patterns and their estimation rules.

#### **Intercurrent Event Patterns**



e Discontinuation of MDI rescue sensor S Withdrawal from study

#### Intercurrent Event 'Estimation Rules' 1-4



#### Intercurrent Events related to CIS

In order to implement the intercurrent event strategy detailed in Section 7.2.2.3 Strategy for Intercurrent (Post-Randomisation) Events, it is necessary to determine if and when the reasons for permanent discontinuations related to CIS occur.

The date and reason for withdrawing from the study will be determined from the study conclusion page of the eCRF.

Study discontinuation reasons classified as related to CIS are as follows:

• Withdrew consent – dissatisfaction with the connected inhaler system (CIS)

#### Percentage of Rescue Free Days Endpoint

#### Monthly Percentage of Rescue Free Days - Calculation

STEP 1: Creating the observed adherence dataset (Observed Dataset A)

To determine the monthly <u>observed</u> percentage of rescue free days values (Observed Dataset A) the following should be applied for each month:

For Baseline Analysis Month, for each participant create a count of each of the following types of Days

- D1 = Rescue use recorded
- D2 = Device incident
- D3 = Post discontinuation of MDI rescue sensor
- D4 = MDI rescue free

D5=D1 + D2 + D3 + D4, i.e. The total number of days within the Baseline Analysis Month; the total number of days between Beginning Timepoint and Ending Timepoint as defined in Table 5 in Section 10.2 Appendix 2: Assessment Windows.

For Analysis Month 1, 2, 3, 4 and 5, for each participant create a count of each of the following types of days:

- D1 = Rescue use recorded
- D2 = Device incident
- D3 = Post discontinuation of MDI rescue sensor
- D4 = MDI rescue free
- D5 = D1 + D2 + D3 + D4, i.e. The total number of days within the Analysis Month; the total number of days between Beginning Timepoint and Ending Timepoint as defined in Table 5 in Section 10.2 Appendix 2: Assessment Windows.

For Analysis Month 6, for each participant create a count of each of the following types of days:

- D1 = Rescue use recorded
- D2 = Device incident
- D3 = Post discontinuation of MDI rescue sensor
- D4 = MDI rescue free
- D5 = D1 + D2 + D3 + D4, i.e. the total number of days within Analysis Month 6; the total number of days between Beginning Timepoint and Ending Timepoint as defined in Table 5 in Section 10.2 Appendix 2: Assessment Windows.

The following observations from the sensor and eCRF will be required to determine the above Days and the differences between missing at random due to device/sensor incident and non-adherent days.

- Device malfunction date
- Sensor malfunction date
- Permanent discontinuation of MDI rescue sensor
- First and last individual sensor synchronisation dates

The first and last individual sensor synchronisation dates will be provided in the sensor dataset. These dates will be used to assess whether missing observations are due to rescue free days or data being missing at random due to device/sensor malfunction.

For each Analysis Month, the Observed MDI rescue free days (%) for that month will be calculated as follows:

Monthly observed MDI rescue free days (%) = 
$$\left(\frac{D4}{D5 - D2 - D3}\right) \times 100$$

#### STEP 2: Creating the modified observed MDI rescue free dataset (Observed Dataset B)

The Observed Dataset A will be duplicated. Using the values in the duplicate dataset (Observed Dataset B) the Analysis Month where the MDI rescue sensor was permanently discontinued before the end of that month (and therefore presents a monthly rescue free rate based on partly observed sensor data for that month) will be imputed as missing; i.e.in Dataset B, if within an Analysis Month (D3>0 and D3<D5) then set monthly value for that Analysis Month to missing. (Note: unless the participant is a completer in which case do not set the value to missing for that Analysis Month).

#### STEP 3: Creating the reference imputed datasets under MAR and J2R method

Using each of the two observed datasets (Observed Dataset A and Observed Dataset B) monthly values, create four separate reference imputed datasets (J2R-Dataset A, J2R-Dataset B, MAR-Dataset A, MAR-Dataset B) that account for the two imputation methods (J2R or MAR). Completely missing intermediate monthly values will be assumed MAR.

The multiple imputation will be implemented using the methods described in Carpenter, 2013 using macros, Part1A, Part1B, Part2A and Part2B (available from <a href="https://missingdata.lshtm.ac.uk/2017/04/06/gsk-five-macros/">https://missingdata.lshtm.ac.uk/2017/04/06/gsk-five-macros/</a>). The seeds are documented at the end of Section 10.5.3.2 and 1000 draws will be used in the relevant macros parameters.

Due to the range of the rescue free days percentages being limited between 0 and 100, the multiple imputation process can generate percentages outside the possible range of values (< 0% or > 100%). A cap will be put in place where values imputed < 0 will be set as 0 and values imputed as > 100 set as 100.

#### STEP 4: Creating the Monthly Analysis values dataset

For each month within each participant create a count of each of the following durations based on intercurrent events: Let,

r1 = MDI rescue sensor still in use

r2 = MDI rescue sensor discontinued but MDI rescue use ongoing until study withdrawal

r3 = MDI rescue discontinued at study withdrawal (includes days post withdrawal from the study). Note, if participant is a completer then for Analysis Month 6, r3=0.

r4 = r1 + r2 + r3

Note: it is assumed that MDI rescue use is not discontinued until permanent discontinuation of the study. Therefore, discontinuation date of MDI rescue use is the same date as permanent discontinuation of study

Set participants monthly values to observed, MARA, MARB, J2RA, J2RB imputation, no data each with a r1, r2, r3 duration.

Examples include to following:

 A participant who prematurely discontinues sensor after 20 days of Analysis Month 5 and withdraws from study after 5 days of Analysis Month 6

| Subject<br>Id | Draw | Month | A | В | J2RA | J2RB | MARA | MARB | r1 | r2 | r3 | r4 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Х | 1 | 1 | 77 | 77 | 77 | 77 | 77 | 77 | 28 | 0 | 0 | 28 |
| X | 1 | 2 | 82 | 82 | 82 | 82 | 82 | 82 | 28 | 0 | 0 | 28 |
| Х | 1 | 3 | 87 | 87 | 87 | 87 | 87 | 87 | 28 | 0 | 0 | 28 |
| Х | 1 | 4 | 77 | 77 | 77 | 77 | 77 | 77 | 28 | 0 | 0 | 28 |
| X | 1 | 5 | 71 | | 71 | 77 | 71 | 78 | 20 | 8 | 0 | 28 |
| X | 1 | 6 | | | 80 | 79 | 77 | 76 | 0 | 5 | 23 | 28 |

 A participant who concurrently prematurely discontinues sensor and withdraws from study after 20 days of Analysis Month 5

| Subject<br>Id | Draw | Month | Α | В | J2RA | J2RB | MARA | MARB | r1 | r2 | r3 | r4 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| X | 1 | 1 | 77 | 77 | 77 | 77 | 77 | 77 | 28 | 0 | 0 | 28 |
| X | 1 | 2 | 80 | 80 | 80 | 80 | 80 | 80 | 28 | 0 | 0 | 28 |
| X | 1 | 3 | 79 | 79 | 79 | 79 | 79 | 79 | 28 | 0 | 0 | 28 |
| X | 1 | 4 | 75 | 75 | 75 | 75 | 75 | 75 | 28 | 0 | 0 | 28 |
| Х | 1 | 5 | 83 | | 83 | 77 | 83 | 79 | 20 | 0 | 8 | 28 |
| Х | 1 | 6 | | | 77 | 77 | 75 | 80 | 0 | 0 | 28 | 28 |

A participant who completes the study after 27 days in Analysis Month 6

| Subject<br>Id | Draw | Month | Α | В | J2RA | J2RB | MARA | MARB | r1 | r2 | r3 | r4 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Х | 1 | 1 | 77 | 77 | 77 | 77 | 77 | 77 | 28 | 0 | 0 | 28 |
| Х | 1 | 2 | 82 | 82 | 82 | 82 | 82 | 82 | 28 | 0 | 0 | 28 |
| Х | 1 | 3 | 87 | 87 | 87 | 87 | 87 | 87 | 28 | 0 | 0 | 28 |
| Х | 1 | 4 | 77 | 77 | 77 | 77 | 77 | 77 | 28 | 0 | 0 | 28 |
| Х | 1 | 5 | 80 | 80 | 80 | 80 | 80 | 80 | 28 | 0 | 0 | 28 |
| Х | 1 | 6 | 82 | 82 | 82 | 82 | 82 | 82 | 15 | 12 | 0 | 27 |

For Arms 1 and 2,

• If the sensor is in use for at least a day within a month, r1>0 then let the analysis value be a combined value (weighted average) of the J2RA observed and MARB imputed values, by taking a proportion of each value based on the proportion of days the sensor is in use and not in use in that month

Analysis value =  $r1/r4 \times (value from J2RA) + (r2+r3)/r4 \times (value from MARB)$ Note the weight is, r4

• Else if the sensor was not used in the month, r1=0 then let the analysis value be the imputed value, Analysis value = value from J2RA dataset (which is the imputed value)

Implement special case of MAR post-early discontinuation of study by identifying participants where the MDI rescue sensor is prematurely discontinued and the participant concurrently withdraws from the study. Where study withdrawal has not been discontinued after the sensor but on the same day, r2=0.

• If the sensor is in use for at least a day within a month, r1>0 then let the analysis value be a combined value (weighted average) of the J2RA observed and MARB imputed values, by taking a proportion of each value based on the proportion of days the MDI rescue was in use and not in use in that month

Analysis Value =  $r1/r4 \times (value from J2RA) + r3/r4 \times (value from MARB)$ Note the weights are r4

Else if the sensor was not used in the month, r1=0 then let the analysis value be the imputed value,
 Analysis value = value from MARA dataset (which is the imputed value)

For Arm 3 and 4.

• If the sensor is in use for at least a day within a month, r1>0 then let the analysis value be a combined value (weighted average) of the J2RA observed and J2RB imputed values, by taking a proportion of each value based on the proportion of days the MDI sensor is in use and not in use in that month

Analysis value =  $r1/r4 \times (value from J2RA) + (r2+r3)/r4 \times (value from J2RB)$ Note the weight is, r4

• Else if the sensor was not used in the month, r1=0 then let the analysis value be the imputed value, Analysis value = value from J2RA dataset (which is the imputed value)

Implement special case of MAR post-early discontinuation of study by identifying participants where the MDI rescue sensor is prematurely discontinued and the participant concurrently withdraws from the study and study withdrawal reason is <u>not</u> related to CIS. Where study withdrawal has not been discontinued after the sensor but on the same day, r2=0.

• If the sensor is in use for at least a day within a month, r1>0 then let the analysis value be a combined value (weighted average) of the J2RA observed and MARB imputed values, by taking a proportion of each value based on the proportion of days the MDI rescue was in use and not in use in that month

Analysis Value =  $r1/r4 \times (value from J2RA) + r3/r4 \times (value from MARB)$ Note the weights are r4

• Else if the sensor was not used in the month, r1=0 then let the analysis value be the imputed value, Analysis value = value from MARA dataset (which is the imputed value)

Implement special case of J2R post-early discontinuation of study by identifying participants where the MDI rescue sensor is prematurely discontinued and the participant concurrently withdraws from the study and study withdrawal reason <u>is</u> related to CIS. Where study withdrawal has not been discontinued after the sensor but on the same day, r2=0.

• If the sensor is in use for at least a day within a month, r1>0 then let the analysis value be a combined value (weighted average) of the J2RA observed and J2RB imputed values, by taking a proportion of each value based on the proportion of days the MDI rescue was in use and not in use in that month

Analysis Value = r1/r4 x (value from J2RA) + r3/r4 x (value from J2RB) Note the weights are r4

Else if the sensor was not used in the month, r1=0 then let the analysis value be the imputed value,
 Analysis value = value from J2RA dataset (which is the imputed value)

STEP 5: Secondary Endpoint Percentage of Rescue Free Days Endpoint calculation

The calculations presented in the previous steps support the final derivation of the following secondary endpoint, the percentage of rescue free days between

o the beginning of Month 4 and the end of Month 6

For participants who complete the study during the endpoint period of interest:

Analysis Endpoint is the average of monthly Analysis Values over the number of months in the endpoint period of interest, i.e.

Month 4 to Month 6

For participants who prematurely discontinue the study during the endpoint period of interest for reasons related or not related to CIS, the MAR or J2R imputation assumes participants would have continued in the study until the end of the period of interest. The weight is the total duration within the endpoint period of interest. This weight will be applied to each month within the period of interest and results summed together to produce the final endpoint/response variable for modelling within macro Part 3.

Note the weight is, total expected study duration within the period of interest. The proportion of weight to apply per monthly Analysis value is r1+r2+r3/ Total expected study duration within the period of interest.

#### **Seeds for Multiple Imputations Macros**

Seeds for all planned MI analyses were determined in advance using the following SAS code and documented within this RAP prior to unblinding:

```
data temp;
do i = 1 to 6;
number=round(10000*ranuni(0),1);
output;
end;
run;
proc print;
```

run;

### Part 1B Macro Seed for Parameter Estimation Using Bayesian MCMC Procedure

| Endpoint | Input Dataset | Macro Seed |
|--------------------------------|--------------------|------------|
| Percentage of Rescue Free Days | Observed Dataset A | 9170 |
| | Observed Dataset B | 5337 |

# Part 2B Macro Seeds for Multiple Imputation of Datasets

| Endpoint | Multiple Imputation Method | Macro Seed | Output Dataset |
|---|---|---|---|
| Percentage of Rescue Free Days | MAR | 2553 | MAR Dataset A |
| | J2R | 8350 | J2R Dataset A |
| | MAR | 4380 | MAR Dataset B |
| | J2R | 2045 | J2R Dataset B |

#### 10.5.3.3. Patient Reported Outcomes

#### Asthma Control Test (ACT)

The ACT is a validated self-administered questionnaire utilising 5 questions to assess asthma control during the past 4 weeks on a 5-point categorical scale (1 to 5).

By answering all 5 questions, a participant with asthma can obtain a score that may range between 5 and 25, with higher scores indicating better control. An ACT total score of 5 to 19 suggests that the participant's asthma is unlikely to be well controlled. A score of 20 to 25 suggests that the participant's asthma is likely to be well controlled. The minimally important difference (MID) for ACT is 3 [Schatz, 2009].

The total score is calculated as the sum of the scores from all 5 questions [Nathan,2004], provided all scores are non-missing; if any individual scores are missing then the overall score will be set to missing. The ACT total scores calculated using the electronic version on the ePRO device will be used; i.e. total scores will not be rederived from the individual question responses.

ACT will be completed on an ePRO device at the clinical study site and at the times detailed in Appendix 1: Schedule of Activities.

#### Asthma Symptom Utility Index (ASUI)

The ASUI is a 10-item self-administered questionnaire with 4 questions on asthma symptoms (Cough, wheeze, shortness of breath, awakening at night) and 1 question about the side effects of asthma medications [Revicki, 1998].

For each symptom, there are 2 dimensions; frequency and severity. The questionnaire is based on a 2-week patient recall of symptoms with response options of 0 to 4 for frequency (not at all, 1 to 3 days, 4 to 7 days, and 8 to 14 days) and severity (not applicable, mild, moderate and severe).

ASUI score ranges from 0 (worst possible symptoms) to 1 (no symptoms) and the MID of the ASUI is considered to be 0.09 [Bime, 2012]. If the response to any question is missing then the ASUI is also set to missing.

A multi-attributable utility theory was used to construct a model for calculating ASUI utilities from individual patient responses [Revicki, 1998]. The multi-attributable utility function is:

$$ASUI = 1.200 \times (s_1 \times s_2 \times s_3 \times s_4 \times s_5) - 0.200$$

where ASUI is the utility of the symptom state on a scale where the best state (no symptoms) has a score of 1 and worst possible symptoms (severe symptoms for 8 to 14 days) has a score of 0; and  $i_s$  is the score for the level on symptom i. The table below shows the coefficients for calculating the ASUI scores:

| | Symptom (Attribute) | | | | |
|---|---|---|---|---|---|
| Level, d | Cough, S <sub>1</sub> | Wheeze, S <sub>2</sub> | Dyspnoea, | Awaken at | Medication Side |
| | | | S <sub>3</sub> | Night, S₄ | Effects, S <sub>5</sub> |
| 1 None | 1.0 | 1.0 | 1.0 | 1.0 | 1.0 |
| 2 Mild, 1-3 | 0.985 | 0.962 | 0.946 | 0.955 | 0.970 |
| 3 Mild, 4-7 | 0.963 | 0.940 | 0.920 | 0.931 | 0.954 |
| 4 Mild, 8-14 | 0.935 | 0.913 | 0.885 | 0.899 | 0.930 |
| 5 Moderate, 1-3 | 0.955 | 0.913 | 0.892 | 0.909 | 0.924 |
| 6 Moderate, 4-7 | 0.920 | 0.886 | 0.860 | 0.880 | 0.900 |
| 7 Moderate, 8- | 0.875 | 0.851 | 0.818 | 0.845 | 0.862 |
| 14 | | | | | |
| 8 Severe, 1-3 | 0.863 | 0.810 | 0.771 | 0.821 | 0.824 |
| 9 Severe, 4-7 | 0.813 | 0.772 | 0.729 | 0.781 | 0.789 |
| 10 Severe, 8-14 | 0.751 | 0.729 | 0.681 | 0.734 | 0.730 |

ASUI will be completed on an ePRO device at the clinical study site and at the times detailed in Appendix 1: Schedule of Activities.

#### St. George's Respiratory Questionnaire (SGRQ)

The St. George's Respiratory Questionnaire is a well-established instrument, comprising a 50-item questionnaire designed to measure Quality of Life in patients with diseases of airway obstruction, measuring symptoms, impact, and activity.

The questions are designed to be self-completed by the participant with a recall over the past 4 weeks [Jones, 1992].

Scores are expressed as the percentage of overall impairment with 100 equalling to the worst possible health status and 0 indicating the best possible health status.

Scoring in each domain of the SGRQ (Symptoms, Activity, Impacts) and the Total score are described in the St George's Respiratory Questionnaire Manuel (Version 2.3, 2009).

SGRQ will be completed on an ePRO device at the clinical study site and at the times detailed in Appendix 1: Schedule of Activities.

#### **Patient Activation Measure (PAM-13)**

Patient Activation Measure will be used to assess the knowledge, skills and confidence a person has in managing their own health and health care.

The PAM contains a series of 13 statements designed to assess the extent of a patient's activation. These statements are about beliefs, confidence in the management of health-related tasks and self-assessed knowledge. Patients are asked to rate the degree to which they agree or disagree with each statement. These answers are combined to provide a single score of between 0 and 100, which represents the patients' concept of themselves as an active manager of their health and health care. There is no specified timeframe on which responses should be based, the questionnaire is suitable to be used to measure changes in activation over time and can be performed before and after an intervention [Hibbard, 2004].

The 13 items have four possible response options: (1) disagree strongly, (2) disagree, (3) agree and (4) agree strongly, and an additional "Not applicable" option. The total PAM score is then calculated by dividing the raw score over the number of items answered (not including the non-applicable items) and multiplied by 13. This score is then transformed to a scale with a range of 0-100 based on calibration tables and proprietary PAM algorithm (<a href="http://www.insigniahealth.com/">http://www.insigniahealth.com/</a>). The score will be provided for analysis.

#### Medication Adherence Report Scale for Asthma (MARS-A)

The MARS-A is a 10-item questionnaire where medication use is rated on a 5-point Likert scale (1 indicating 'always' to 5 indicating 'never'). It has been validated as a self-reported measure of adherence with ICS for patients with asthma, and includes generic ("I use it regularly every day") and lung condition-specific questions about medication use ("I only use it when I feel breathless") [Cohen, 2009].

The MARS-A 10-Score will be calculated for each participant as the sum of scores for each of the ten questions divided by the number of non-missing responses to the ten questions.

If some responses are missing the MARS-A 10-score is calculated as follows for each participant:

• If eight or more of the questions have been answered, the missing responses for that participant will be imputed to the average score

 If less than eight of the questions have been answered, the overall MARS-A 10-score for that participant will be set to missing

MARS-A will be completed on an ePRO device at the clinical study site and at the times detailed in Appendix 1: Schedule of Activities.

#### **Beliefs in Medicine Questionnaire (BMQ)**

The BMQ questionnaire consists of the BMQ Specific, which measures perceptions of specific medicines, and the BMQ General, which measures more general beliefs about medicines. All items are scored on a 5-point Likert scale ranging from Strongly Disagree (1) to Strongly Agree (5).

The BMQ Specific questionnaire is formed of the 6 item Necessity and 12 item Concern scales, and the General questionnaire is formed of the 4 item Benefit, 5 item Harm and 3 item Overuse scales.



Scores obtained for individual items within scales are summed together to provide a total score. The BMQ Specific and General will be completed on an ePRO device at the clinical study site and at the times detailed in Appendix 1: Schedule of Activities.

#### **Biomarkers**

#### **PEF and FeNO**

- Participants should not use their rescue medication for at least 6 hours before each FeNO and PEF assessment, unless essential for clinical need. Participants should also withhold ICS/LABA for (1 dosing interval) approximately 12-24 hours prior to FeNO and PEF assessment.
- PEF and FeNO will be taken in triplicate at the times detailed in Appendix 1: Schedule of Activities. All 3
  measures will be recorded in the eCRF.
- The maximum value from the 3 measures taken at each visit will be used in the calculation of the FeNO and PEF endpoints.

#### **Severe Asthma Exacerbations**

#### General

Missing onset or resolution dates will be handled as follows:

- Single event with missing onset and/or resolution dates:
  - (a) Missing onset date: set onset date = study treatment start date
  - (b) Missing resolution date: set resolution date = study treatment stop date
  - (c) Both missing: imputed per both (a) and (b)
- Multiple events, one event with some missing onset/resolution dates; on the assumption any partial date information does not occur during the other events:
  - (a) Missing onset date: set onset date = max[(resolution date of the nearest previous event) + 1 day, study treatment start date]
  - (b) Missing resolution date: set resolution date = min[(onset date of the nearest subsequent event)- 1 day, study treatment stop date]
  - (c) Both missing: determine the largest gap between study treatment start date and first event onset date, between first event resolution date and next event(s) onset dates (if any), between last event resolution date and study treatment stop date. If there is more than one gap which is the largest, then take the first occurrence. Then impute as follows:

onset date = (onset date of largest gap) + 1 day

resolution date = (resolution date of largest gap) + 1 day

### 10.5.4. Safety

#### **Adverse Events**

 Adverse events will be coded using the current MedDRA coding dictionary at the time of reporting providing a Preferred Term (PT) and a System Organ Class (SOC) for analysis and reporting.

#### **ADRs and SAEs of Special Interest**

ADR and SAE groups of special interest have been defined as SAEs which are included in specified areas of interest for Relvar/Breo. They are identified by groupings of preferred terms based on the Medical Dictionary for Regulatory Activities (MedDRA) dictionary version used in each reporting effort. Groupings or subgroups may be defined, based on relevant combination of preferred terms, or on Standardised MedDRA queries (SMQs).

SAEs of special interest will be confirmed prior to final data, based on the MedDRA version in use at the time

# 10.6. Appendix 6: Reporting Standards for Missing Data

# 10.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Participant study completion (as specified in the protocol) is defined as completing all visits of the study including the follow-up phone contact.</li> <li>Withdrawn participants will not be replaced in the study.</li> <li>All available data from participants who are withdrawn from the study will be included in listings and where possible any available data from withdrawn participants will be included in summaries or analyses, unless otherwise specified.</li> </ul> |

# 10.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in participant listing displays. If all data for a specific visit are missing, the visit will be excluded from the display.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and will be displayed as such.</li> </ul> |
| MMRM<br>Analysis | All the available assessments taken at scheduled visits will be included in the repeated measures models in which missing data are not explicitly imputed but the correlation between visits for all participants is used to adjust the estimate of treatment effect considering any missing data. |
| Rescue Free<br>Days<br>Endpoint | Handling of missing sensor data is detailed in Section 7.2.2.3 Strategy for Intercurrent (Post-Randomisation) Events, as well Section 10.5.3.2 MDI Device Sensor Assessments. |
| ACT | Handling of missing ACT data is detailed in Section 7.2.3.3 Strategy for Intercurrent (Post-Randomisation) Events. |
| Other PROs | Handling of missing PRO data is detailed in Section 7.3.3.4 Strategy for Intercurrent (Post-Randomisation) Events, as well in Section 10.5.3.3 Patient Reported Outcomes. |

# 10.6.3. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in participant listing displays. |
| Adverse<br>Events | The eCRF does not allow partial dates to be captured for AEs. All dates will either be complete or missing. |
| | Completely missing start or end dates will remain missing, with no imputation applied. |
| | Where AE onset dates are missing then the AE will be considered on-treatment. |
| Concomitant<br>Medications | <ul> <li>The eCRF allows partial dates to be captured for concomitant medications.</li> <li>Partial dates for any concomitant medications recorded in the eCRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be</li> </ul> </li> </ul> |
| | used for the month If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month. |

| Element | Reporting Detail |
|---|---|
| | The answers to the questions "Taken Prior to Study?" and "Ongoing?" which are recorded in the eCRF will also be taken into consideration to determine if the medication was started pre-treatment or continued post-treatment. In each case, should the answers suggest a different classification than the dates, the medication will be summarized in all possible classifications (pre-/during/post-treatment) in which it could conceivably have been taken. |
| Exacerbations | Exacerbations are treated in the same way as AEs. |

# 10.7. Appendix 7: Abbreviations & Trade Marks

# 10.7.1. Abbreviations

| Abbreviation | Description |
|--------------|-----------------------------------------------------|
| ACT | Asthma Control Test |
| ADaM | Analysis Data Model |
| ADR | Adverse Drug Reaction |
| AE | Adverse Event |
| ANCOVA | Analysis of Covariance |
| A&R | |
| ASUI | Analysis and Reporting Asthma Symptom Utility Index |
| ATC | Anatomical Therapoutical Chamical |
| | Anatomical Therapeutical Chemical |
| BMQ | Beliefs in Medicine Questionnaire |
| CDISC | Clinical Data Interchange Standards Consortium |
| Cl | Confidence Interval |
| CIS | Connected Inhaler System |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| DM | Data Management |
| DPI | Dry powder inhaler |
| eCRF | Electronic Case Record Form |
| ER | Emergency Room |
| EW | Early Withdrawal |
| FeNO | Fractional exhaled Nitric Oxide |
| GLM | Generalized Linear Model |
| GSK | GlaxoSmithKline |
| HCP | Healthcare Professional |
| HCRU | Health Care Resource Utilization |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| ICF | Informed Consent Form |
| ICS | Inhaled Corticosteroid |
| IDSL | Integrated Data Standards Library |
| ITT | Intent-To-Treat |
| J2R | Jump to reference |
| LABA | Long-Acting Beta2-Agonist |
| MAR | Missing At Random |
| MARS-A | Medication Adherence Report Scale for Asthma |
| MDI | Metered dose inhaler |
| MMRM | Mixed Model Repeated Measures |
| PAM | Patient Activation Measure |
| PDMP | Protocol Deviation Management Plan |
| PEF | Peak Expiratory Flow |
| PRO | Patient Reported Outcomes |
| PT | Preferred Term |
| L * * | |

| Abbreviation | Description |
|--------------|--------------------------------------------|
| QC | Quality Control |
| RAP | Reporting & Analysis Plan |
| RFD | Rescue Free Day |
| RAMOS | Randomisation & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| S&P | Statistics and Programming |
| SD | Standard Deviation |
| SDL | Source Data Lock |
| SDTM | Study Data Tabulation Model |
| SGRQ | St. Georges Respiratory Questionnaire |
| SI | System Independent |
| SMQ | Standardised MedDRA Queries |
| SOC | System Organ Class |
| TRU | Total Rescue Use |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |

# 10.7.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| BREO |
| ELLIPTA |
| RELVAR |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| ACT |
| ASUI |
| BMQ |
| MARS-A |
| MedDRA |
| PAM-13 |
| RAMOS NG |
| SAS |
| SGRQ |

## 10.8. Appendix 8: List of Data Displays

# 10.8.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------------|--------------|
| Study Population | 1.01 to 1.44 | 1.01 to 1.02 |
| Efficacy | 2.01 to 2.41 | 2.01 to 2.22 |
| Safety | 3.01 to 3.29 None | |
| Section | List | ings |
| ICH Listings | 1 to 19 | |
| Other Listings | 20 to 44 | |

# 10.8.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 9: Example Mock Shells for Data Displays: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|----------------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | Not applicable | SAFE_Tn | SAFE_Ln |

#### NOTES:

• Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 10.8.3. Deliverables

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| SAC [2] | Final Statistical Analysis Complete |
| DRY RUN [1] | Dry Run |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# 10.8.4. Study Population Tables

| Study I | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | Screened | IDSL_SP1 | Summary of Subject Populations | See Section 4 for population details | SAC [2]<br>DRY RUN [1] |
| 1.2. | Enrolled | IDSL_ES6 | Summary of Screening Status and Reasons for Screen Failure | | SAC [2]<br>DRY RUN [1] |
| 1.3. | Enrolled | IDSL_ES6 | Summary of Run-in Status and Reasons for Run-In Failure | | SAC [2]<br>DRY RUN [1] |
| 1.4. | ITT | POP_T1 | Summary of Attendance at Each Visit | Note: Visit 2/3/4 subjects may be randomised or re-entered into run-in up 3 times if ACT ≥ 20. Note: Visits 6/7/8/9 are Healthcare Professional Dashboard reviews for Arm 1 and Arm 3. | SAC [2]<br>DRY RUN [1] |
| 1.5. | ITT | IDSL_ES1 | Summary of Subject Disposition for the Subject Conclusion Record | | SAC [2]<br>DRY RUN [1] |
| 1.6. | ITT | IDSL_ES4 | Summary of Subject Disposition at Each Study Epoch | | SAC [2]<br>DRY RUN [1] |
| 1.7. | ITT | IDSL_SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | | SAC [2]<br>DRY RUN [1] |
| 1.8. | ITT | POP_T2 | Summary of Relvar/Breo ELLIPTA Sensor Status | | SAC [2]<br>DRY RUN [1] |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.9. | ITT | POP_T2 | Summary of Salbutamol MDI Sensor Status | | SAC [2]<br>DRY RUN [1] |
| 1.10. | ITT | POP_T3 | Summary of App Status | | SAC [2]<br>DRY RUN [1] |
| 1.11. | Enrolled | IDSL_NS1 | Summary of Number of Subjects Enrolled by Country and Site ID | Disclosure display Add "No Treatment" column Do by page by country to help fit all columns in one width. | SAC [2]<br>DRY RUN [1] |
| 1.12. | ITT | IDSL_NS1 | Summary of Number of Subjects Enrolled by Country and Site ID | Do by page by country for consistency with above display | SAC [2]<br>DRY RUN [1] |
| 1.13. | ITT | IDSL_IE1 | Summary of Inclusion/Exclusion Criteria Deviations | | SAC [2]<br>DRY RUN [1] |
| 1.14. | ITT | IDSL_DV1 | Summary of Important Protocol Deviations | | SAC [2]<br>DRY RUN [1] |
| Demog | raphic and Basel | ine Characteris | tics | | |
| 1.15. | ITT | IDSL_DM1 | Summary of Demographic Characteristics | Include, Gender, Age (years), Age group categories: 18-64, 65-84 and >=85, Ethnicity, Height, Weight, BMI | SAC [2]<br>DRY RUN [1] |
| 1.16. | ITT | IDSL_DM1 | Summary of Demographic Characteristics by Country | | SAC [2]<br>DRY RUN [1] |
| 1.17. | Enrolled | IDSL_DM11 | Summary of Age ranges | Disclosure displays / Categories: 18-64, 65-84 and >=85. Include "No Treatment" column | SAC [2]<br>DRY RUN [1] |

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.18. | ITT | IDSL_DM5 | Summary of Race and Racial Combinations | | SAC [2]<br>DRY RUN [1] |
| 1.19. | ITT | IDSL_DM6 | Summary of Race and Racial Combination Details | | SAC [2]<br>DRY RUN [1] |
| Medica | l Conditions | | | | |
| 1.20. | ITT | IDSL_MH4 | Summary of Current Medical Conditions | | SAC [2]<br>DRY RUN [1] |
| 1.21. | ITT | IDSL_MH4 | Summary of Past Medical Conditions | | SAC [2]<br>DRY RUN [1] |
| 1.22. | ITT | IDSL_FH1 | Summary of Family History of Cardiovascular Risk Factors | | SAC [2]<br>DRY RUN [1] |
| 1.23. | ITT | IDSL_SU1 | Summary of Substance Use at Screening | Include Smoking History, for the<br>Current and Former Smokers<br>include Years smoked,<br>Cigarettes/Day, Smoking Pack<br>Years | SAC [2]<br>DRY RUN [1] |
| Disease | e Characteristics | | | | • |
| 1.24. | ITT | POP_T4 | Summary of Asthma Duration at Screening | | SAC [2]<br>DRY RUN [1] |
| 1.25. | ITT | POP_T5 | Summary of Exacerbation History at Screening | | SAC [2]<br>DRY RUN [1] |
| 1.26. | ITT | POP_T6 | Summary of Screening and Randomisation Peak Expiratory Flow (PEF) | Summarize using the maximum value at visit | SAC [2]<br>DRY RUN [1] |
| Study F | Study Population Tables | | | | | | | |
|---|---|---|---|---|---|--|--|--|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] | | | |
| 1.27. | ITT | POP_T6 | Summary of Screening and Randomisation Peak Expiratory Flow (PEF) by Country | Summarize using the maximum value at visit | SAC [2]<br>DRY RUN [1] | | | |
| 1.28. | ITT | POP_T6 | Summary of Screening and Randomisation Fractional Exhaled Nitric Oxide (FeNO) | Summarize using the maximum value at visit | SAC [2]<br>DRY RUN [1] | | | |
| Concor | nitant Medicatior | ıs | | | | | | |
| 1.29. | ITT | IDSL_CM1 | Summary of Concomitant Medications Taken in the Run-in, Medications Given for Severe Exacerbation | | SAC [2]<br>DRY RUN [1] | | | |
| 1.30. | ITT | IDSL_CM1 | Summary of On-Treatment Asthma Concomitant Medications, Medications Given for Severe Exacerbation | | SAC [2]<br>DRY RUN [1] | | | |
| 1.31. | ITT | IDSL_CM1 | Summary of On-Treatment Asthma Concomitant Medications | | SAC [2]<br>DRY RUN [1] | | | |
| 1.32. | ITT | IDSL_CM1 | Summary of Post-Treatment Asthma Concomitant Medications | | SAC [2]<br>DRY RUN [1] | | | |
| 1.33. | ITT | IDSL_CM1 | Summary of Run-in Treatment Asthma Concomitant Medications | | SAC [2]<br>DRY RUN [1] | | | |
| 1.34. | ITT | IDSL_CM1 | Summary of On-Treatment Non-Asthma Concomitant Medications | | SAC [2]<br>DRY RUN [1] | | | |
| 1.35. | ITT | IDSL_CM1 | Summary of Post-Treatment Non-Asthma Concomitant Medications | | SAC [2]<br>DRY RUN [1] | | | |
| 1.36. | ITT | IDSL_CM1 | Summary of Run-in Treatment Non-Asthma Concomitant Medications | | SAC [2]<br>DRY RUN [1] | | | |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.37. | ITT | IDSL_CM1 | Summary of Asthma Concomitant Medications Taken Prior to Screening | Ensure the observations dates are pre-screening visit 1 (there is a specific prior conmeds page in eCRF | SAC [2]<br>DRY RUN [1] |
| Exposu | re and Treatmer | nt Compliance | | | |
| 1.38. | ITT | POP_T7 | Summary of Exposure to Study Medication | Post-randomisation treatment exposure | SAC [2]<br>DRY RUN [1] |
| 1.39. | ITT | POP_T8 | Summary of the Frequency of Puffs Per Day – ELLIPTA Sensor | Programming Note: Repeat for Months 2, 3, 4, 5, 6, Months 4-6, Months 1-6 and Months 1-3. Frequency of puffs per day over the baseline and on-treatment period as defined in the Assessment Windows of RAP | SAC [2]<br>DRY RUN [1] |
| 1.40. | ITT | POP_T8 | Summary of the Frequency of Puffs Per Day – MDI Sensor | Programming Note: Repeat for Months 2, 3, 4, 5, 6, Months 4-6, Months 1-6 and Months 1-3. Frequency of puffs per day over the baseline and on-treatment period as defined in the Assessment Windows of RAP | SAC [2]<br>DRY RUN [1] |

| Study F | Population Tables | S | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.41. | ITT | POP_T9 | Summary of Treatment Compliance | Post-randomisation compliance Note: Treatment compliance = (Total number of inhalation taken / Expected Inhalation x (Stop date - Start date + 1)) x 100 where Total Number of Inhalations Taken is the total number of doses taken from all inhalers, Expected Inhalations is equal to 1 and Start Date and Stop Date are the earliest treatment start date on or post randomisation and the latest treatment stop date recorded for all the inhalers. | SAC [2]<br>DRY RUN [1] |
| Others | L | | 1 | 1 | |
| 1.42. | ITT | POP_T10 | Summary of Incidence of Preferred Time of Dosing over the<br>Treatment Period | | SAC [2]<br>DRY RUN [1] |
| 1.43. | ITT | POP_T11 | Summary of HCP Dashboard Review by Visit | Note: Visits 6/7/8/9 are Healthcare<br>Professional Dashboard reviews for<br>Arm 1 and Arm 3<br>[1] Action taken – Email/Text/Phone<br>Contact | SAC [2]<br>DRY RUN [1] |
| 1.44. | ITT | POP_T12 | Summary of Prior Prescription Details | | SAC [2]<br>DRY RUN [1] |

# 10.8.5. Study Population Figures

| Study F | Study Population Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Relvar/l | Breo ELLIPTA A | dherence | | | |
| 1.1. | ITT | POP_F1 | Frequency of ELLIPTA Puffs Per Day– ELLIPTA Sensor | Programming Note: Repeat for<br>Period: Month 1, 2, 3, 4, 5, 6, Month<br>4-6, Month 1-3, Month 1-6. | SAC [2]<br>DRY RUN [1] |
| 1.2. | ITT | POP_F1 | Frequency of MDI Puffs Per Day – MDI Sensor | Programming Note: Repeat for<br>Period: Month 1, 2, 3, 4, 5, 6, Month<br>4-6, Month 1-3, Month 1-6. | SAC [2]<br>DRY RUN [1] |

# 10.8.6. Efficacy Tables

| Efficacy | Efficacy Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Relvar/l | Breo ELLIPTA A | dherence | | | |
| 2.1. | ITT | EFF_T1 | Summary of Monthly Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 1 and the end of month 6 as determined by the maintenance sensor – Observed Data | Use the observed monthly values (month 1, 2, 3, 4, 5, 6) [1] Baseline adherence is calculated using up to the last 28 days of daily adherence data during the run-in period. | SAC [2]<br>DRY RUN [1] |

| Efficacy | Efficacy Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.2. | ITT | EFF_T2 | Summary of Statistical Analysis of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor | Present comparisons Arm 1,2,3,4 v<br>Arm 5 | SAC [2]<br>DRY RUN [1] |
| 2.3. | ITT | EFF_T2 | Summary of Statistical Analysis of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor – Generalised Linear Model (Sensitivity Analysis) | Present comparisons Arm 1,2,3,4 v<br>Arm 5 | SAC [2] |
| 2.4. | ITT | EFF_T3 | Summary of Statistical Analysis of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor by Baseline ACT Total Score Group | Subgroup analysis output Update footer with interaction between treatment group arm and baseline ACT Total Score Group | SAC [2]<br>DRY RUN [1] |
| 2.5. | ITT | EFF_T3 | Summary of Statistical Analysis of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor by Age Group | Subgroup analysis output Update footer with interaction between treatment group arm and baseline ACT Total Score Group | SAC [2]<br>DRY RUN [1] |
| 2.6. | ITT | EFF_T4 | Summary of Statistical Analysis of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 1 and the end of month 3 as determined by the maintenance sensor | Present comparisons Arms 1,2,3,4 v Arm 5 | SAC [2]<br>DRY RUN [1] |
| 2.7. | ITT | EFF_T4 | Summary of Statistical Analysis of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 1 and the end of month 3 as determined by the maintenance sensor – Generalised Linear Model (Sensitivity Analysis) | Present comparisons Arm 1,2,3,4 v<br>Arm 5 | SAC [2] |

| Efficacy | / Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.8. | ITT | EFF_T4 | Summary of Statistical Analysis of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 1 and the end of month 6 as determined by the maintenance sensor | Present comparisons Arms 1,2,3,4 v Arm 5 | SAC [2]<br>DRY RUN [1] |
| 2.9. | ITT | EFF_T4 | Summary of Statistical Analysis of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 1 and the end of month 6 as determined by the maintenance sensor – Generalised Linear Model (Sensitivity Analysis) | Present comparisons Arm 1,2,3,4 v<br>Arm 5 | SAC [2] |
| 2.10. | ITT | EFF_T5 | Summary of Statistical Analysis of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor – Impact of Feedback of Sensor Data to HCP | Present comparisons Arm 1 v 2,<br>Arm 3 v 4 | SAC [2]<br>DRY RUN [1] |
| 2.11. | ITT | EFF_T6 | Summary of Statistical Analysis of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor – Impact of Feedback on Rescue Medication Use | Present comparisons Arm 1 v 3,<br>Arm 2 v 4 | SAC [2]<br>DRY RUN [1] |
| Salbuta | mol MDI Rescue | Medication Use | | | l |
| 2.12. | ITT | EFF_T1 | Summary of Monthly Percentage of Rescue Free Days between the beginning of month 1 and then end of month 6 as determined by the rescue medication sensor – Observed Data | Use the observed monthly values (month 1, 2, 3, 4, 5, 6) [1] Baseline rescue free use is calculated using up to the last 28 days of daily rescue use data during the run-in period. | SAC [2]<br>DRY RUN [1] |
| 2.13. | ITT | EFF_T4 | Summary of Statistical Analysis of Percentage of Rescue Free Days between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor | Present comparisons Arms 1,2,3,4 v Arm 5 | SAC [2]<br>DRY RUN [1] |

| Efficacy | y Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.14. | ITT | EFF_T1 | Summary of Total Rescue Medication Use as determined by the maintenance sensor | | SAC [2]<br>DRY RUN [1] |
| Asthma | Control Test (A | CT) | | | |
| 2.15. | ITT | EFF_T1 | Summary of Asthma Control Test (ACT) Total Score | Programming Note: Add screening visit score. [1] Baseline ACT total score is taken at Randomisation visit. | SAC [2]<br>DRY RUN [1] |
| 2.16. | ITT | EFF_T4 | Summary of the Statistical Analysis of Change from Baseline (Randomisation) in ACT Total Score at Month 6 | | SAC [2]<br>DRY RUN [1] |
| 2.17. | ITT | EFF_T12 | Summary of Percentage of Subjects Who Have Either an ACT Total Score >= 20 and/ or >= 3 Point Increase from Baseline in ACT Total Score | See SLS T2.1 | SAC [2]<br>DRY RUN [1] |
| 2.18. | ITT | EFF_T13 | Summary of the Statistical Analysis of Percentage of Patients Who Have an ACT Total Score of >=20 at Month 6 | | SAC [2]<br>DRY RUN [1] |
| 2.19. | ITT | EFF_T13 | Summary of the Statistical Analysis of Percentage of Patients with an Increase from Baseline ≥3 in ACT Total Score at Month 6 | | SAC [2]<br>DRY RUN [1] |
| 2.20. | ITT | EFF_T13 | Summary of the Statistical Analysis of Percentage of Patients Who Have Either an ACT Total Score of ≥ 20 and/or an Increase from Baseline of ≥ 3 in ACT Total Score at Month 6 | | SAC [2]<br>DRY RUN [1] |
| Unsche | duled Health Ca | re Utilisation | | | |
| 2.21. | ITT | EFF_T14 | Summary of Unscheduled Asthma Related Healthcare Utilisation During the Study | | SAC [2]<br>DRY RUN [1] |
| 2.22. | ITT | EFF_T22 | Summary of Primary Care Visits relating to HCP Dashboard Review | | SAC [2]<br>DRY RUN [1] |

| Efficacy | / Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Severe | On-treatment Ex | acerbations | | | |
| 2.23. | ITT | EFF_T15 | Summary of Severe On-Treatment and Post-Treatment Asthma Exacerbations | Exacerbation duration and rates will only be determined from those events that have dates of onset and resolution | SAC [2]<br>DRY RUN [1] |
| | | | | Include a total column | |
| Asthma | Symptom Utility | / Index (ASUI) | | | |
| 2.24. | ITT | EFF_T1 | Summary of Asthma Symptom Utility Index (ASUI) Score | Programming Note: Add screening visit score. Decimal places need to be increased by 2 dp for all values. [1] Baseline ASUI total score is taken at Randomisation visit.Note: | SAC [2]<br>DRY RUN [1] |
| 2.25. | ITT | EFF_T16 | Summary of Statistical Analysis of Percentage of Patients Meeting a Responder Threshold of ≥ 0.09 Points Improvement (Increase) from Baseline (Randomisation) for the ASUI Total Score at Visit 10 (Month 6) | | SAC [2]<br>DRY RUN [1] |
| 2.26. | ITT | EFF_T4 | Summary of Statistical Analysis of Change from Baseline (Randomisation) in Asthma Symptom Utility Index (ASUI) Score at Visit 10 (Month 6) | | SAC [2]<br>DRY RUN [1] |
| St. Geo | rge's Respirator | y Questionnaire | (SGRQ) | | |
| 2.27. | ITT | EFF_T1 | Summary of St. George's Respiratory Questionnaire (SGRQ) Total Score | Programming Note: Add screening visit score. [1] Baseline SGRQ total score is taken at Randomisation visit. | SAC [2]<br>DRY RUN [1] |

| Efficacy | / Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.28. | ITT | EFF_T13 | Statistical Analysis of Percentage of Patients Meeting a Responder Threshold of ≥ 4 Points Improvement (Decrease) from Baseline (Randomisation) for the SGRQ Total Score at Visit 10 (Month 6) | | SAC [2]<br>DRY RUN [1] |
| 2.29. | ITT | EFF_T4 | Summary of Statistical Analysis of Change from Baseline (Randomisation) in St. George's Respiratory Questionnaire (SGRQ) at Visit 10 (Month 6) | | SAC [2]<br>DRY RUN [1] |
| Patient | <b>Activation Meas</b> | ure (PAM-13) | | | |
| 2.30. | ITT | EFF_T1 | Summary of Patient Activation Measure (PAM) 13 Total Score | Programming Note: Add randomisation visit score. [1] Baseline PAM-13 total score is taken at Screening visit. | SAC [2]<br>DRY RUN [1] |
| Medicat | tion Adherence F | Rating Scale As | thma (MARS-A) | | |
| 2.31. | ITT | EFF_T1 | Summary of Medication Adherence Report Scale-Asthma (MARS-A) Total Score | Programming Note: Add randomisation visit score. [1] Baseline MARS-A total score is taken at Screening visit. | SAC [2]<br>DRY RUN [1] |
| Beliefs | about Medicines | (BMQ) | | | |
| 2.32. | ITT | EFF_T1 | Summary of BMQ General Benefit Total Score | Programming Note: Add randomisation visit score. [1] Baseline BMQ total score is taken at Screening visit. | SAC [2]<br>DRY RUN [1] |
| 2.33. | ITT | EFF_T1 | Summary of BMQ General Harm Total Score | Programming Note: Add randomisation visit score. [1] Baseline BMQ total score is taken at Screening visit. | SAC [2]<br>DRY RUN [1] |

| Efficacy | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.34. | ITT | EFF_T1 | Summary of BMQ General Overuse Total Score | Programming Note: Add randomisation visit score. [1] Baseline BMQ total score is taken at Screening visit. | SAC [2]<br>DRY RUN [1] |
| 2.35. | ΙΤΤ | EFF_T1 | Summary of BMQ Specific Necessity Total Score | Programming Note: Add randomisation visit score. [1] Baseline BMQ total score is taken at Screening visit. | SAC [2]<br>DRY RUN [1] |
| 2.36. | ITT | EFF_T1 | Summary of BMQ Specific Concern Total Score | Programming Note: Add randomisation visit score. [1] Baseline BMQ total score is taken at Screening visit. | SAC [2]<br>DRY RUN [1] |
| Medical | Device Incident | S | | | |
| 2.37. | ITT | EFF_T21 | Summary of Medical Device Incidents (Sensors) | | SAC [2]<br>DRY RUN [1] |
| Fraction | nal Exhaled Nitri | Oxide (FeNO) | and Peak Expiratory Flow (PEF) | | |
| 2.38. | ITT | EFF_T1 | Summary of Fractional Exhaled Nitric Oxide (FeNO) | Programming Note: Add screening visit reading. [1] Baseline FeNO readings are taken at Randomisation visit. | SAC [2]<br>DRY RUN [1] |
| 2.39. | ITT | EFF_T23 | Summary of Change from Baseline (Randomisation) in Fractional Exhaled Nitric Oxide (FeNO) at Month 6 (Visit 10) by Percentage of ELLIPTA doses taken (daily adherence) between the beginning of Month 4 and the end of Month 6 Group | The adherence observations should be those taken from the analysis dataset holding the observed % values. These should be grouped in quantiles using the 25th, 50th and 75th percentiles as the data group boundaries. | SAC [2]<br>DRY RUN [1] |

| Efficacy | Efficacy Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.40. | ITT | EFF_T1 | Summary of Peak Expiratory Flow (PEF) | Programming Note: Add screening visit reading. [1] Baseline FeNO readings are taken at Randomisation visit. | SAC [2]<br>DRY RUN [1] |
| 2.41. | ITT | EFF_T23 | Summary of Change from Baseline (Randomisation) in Peak Expiratory Flow (PEF) at Month 6 (Visit 10) by Percentage of ELLIPTA doses taken (daily adherence) between the beginning of Month 4 and the end of Month 6 Group | The adherence observations should be those taken from the analysis dataset holding the observed % values. These should be grouped in quantiles using the 25th, 50th and 75th percentiles as the data group boundaries | SAC [2]<br>DRY RUN [1] |

# 10.8.7. Efficacy Figures

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Relvar/I | Breo ELLIPTA A | dherence | | | |
| 2.1. | ITT | EFF_F5 | Box plot of Monthly Percentage of ELLIPTA doses taken (daily adherence) as determined by the maintenance sensor – Observed Data | Month 1, 2, 3, 4, 5, and 6, ave month 1-3, ave month 4-6, ave month 1-6 across the x-axis. Monthly observed % value on the y-axis. Present each treatment over each month, off-set from one another | SAC [2]<br>DRY RUN [1] |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.2. | ITT | EFF_F3 | Adjusted Treatment Differences for Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor – Comparisons Arm 1,2,3,4 v Arm 5 | ANCOVA Primary endpoint analysis Present "Treatment Arm Difference (95% CI) versus Arm 5" on y-axis and "Treatment Arms" Arm 1, Arm 2, Arm 3 and Arm 4 on the x-axis. | SAC [2]<br>DRY RUN [1] |
| 2.3. | ITT | EFF_F4 | Summary of Interaction Tests for Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor - Comparisons Arm 1,2,3,4 v Arm 5 | Footer: the results displays are from an ANCOVA adjusted for randomised treatment arm, baseline adherence, duration of run-in (visits), country, gender [1] age (years), covariate, and two-way interaction between randomised treatment arm and covariate [2] covariate, two-way interaction between randomised treatment group and covariate. | SAC [2]<br>DRY RUN [1] |
| 2.4. | ITT | EFF_F2 | Scatter Plot of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor (Observed values) by Age | Requires the primary endpoint observed value, each treatment arm presented with a unique symbol/pattern | SAC [2]<br>DRY RUN [1] |
| 2.5. | ITT | EFF_F2 | Scatter Plot of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor (Observed values) by Baseline ACT Total Score | Requires the primary endpoint observed value, each treatment arm presented with a unique symbol/pattern | SAC [2]<br>DRY RUN [1] |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.6. | ITT | EFF_F3 | Adjusted Treatment Differences for Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor – Impact of Feedback of Sensor Data to HCP | ANCOVA Present comparisons Arm 1 v 2, Arm 3 v 4 Present "Treatment Arm Difference (95% CI)" on y-axis and "Treatment Arms" "Arm 1 vs Arm 2" and "Arm 3 vs Arm 4" on the x-axis | SAC [2]<br>DRY RUN [1] |
| 2.7. | ITT | EFF_F3 | Adjusted Treatment Differences for Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor – Impact of Feedback on Rescue Medication Use | ANCOVA Present comparisons Arm 1 v 3, Arm 2 v 4 Present "Treatment Arm Difference (95% CI)" on y-axis and "Treatment Arms" "Arm 1 vs Arm 3" and "Arm 2 vs Arm 4" on the x-axis | SAC [2]<br>DRY RUN [1] |
| 2.8. | ITT | EFF_F3 | Adjusted Treatment Differences for Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 1 and the end of month 3 as determined by the maintenance sensor – Comparisons Arm 1,2,3,4 v Arm 5 | ANCOVA Present comparisons<br>Arms 1,2,3,4 v Arm 5<br>Present "Treatment Arm Difference<br>(95% CI) versus Arm 5" on y-axis<br>and "Treatment Arms" Arm 1, Arm<br>2, Arm 3 and Arm 4 on the x-axis. | SAC [2]<br>DRY RUN [1] |
| 2.9. | ITT | EFF_F3 | Adjusted Treatment Differences for Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 1 and the end of month 6 as determined by the maintenance sensor – Comparisons Arm 1,2,3,4 v Arm 5 | ANCOVA Present comparisons Arms 1,2,3,4 v Arm 5 Present "Treatment Arm Difference (95% CI) versus Arm 5" on y-axis and "Treatment Arms" Arm 1, Arm 2, Arm 3 and Arm 4 on the x-axis. | SAC [2]<br>DRY RUN [1] |

| Efficacy | r: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Salbuta | mol MDI Rescue | Medication Use | | | |
| 2.10. | ITT | EFF_F5 | Box plot of Monthly Percentage of Rescue Free Days as determined by the rescue medication MDI sensor | Month 1, 2, 3, 4, 5, and 6, ave month 4-6 across the x-axis. Monthly observed % value on the y-axis. Present each treatment over each month, off-set from one another | SAC [2]<br>DRY RUN [1] |
| 2.11. | ITT | EFF_F3 | Adjusted Treatment Differences for Percentage of Rescue Free Days between the beginning of month 4 and the end of month 6 as determined by the rescue medication MDI sensor – Comparisons Arm 1,2,3,4 v Arm 5 | ANCOVA Present "Treatment Arm Difference (95% CI) versus Arm 5" on y-axis and "Treatment Arms" Arm 1, Arm 2, Arm 3 and Arm 4 on the x-axis. | SAC [2]<br>DRY RUN [1] |
| Asthma | Control Test (A | CT) | | | |
| 2.12. | ITT | EFF_F3 | Summary of ACT Total Score | Present "ACT Total Score (Mean± SD)" on y-axis and "Visit" on x-axis Baseline, Visit 5 (Month 1), Visit 10 (Month 6). Present mean ACT Total Score ± SD separately for treatment group at each visit, connecting the means with a solid line. Distinguish the treatment groups by different line types. [1] Baseline FeNO readings are taken at Randomisation visit. | SAC [2]<br>DRY RUN [1] |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.13. | ITT | EFF_F3 | Summary of Statistical Analysis for Change from Baseline (Randomisation) in ACT Total Score at Month 6 | (MMRM) Present "Treatment Arm Difference (95% CI) versus Arm 5" on y-axis and "Visit" on x-axis Visit 5 (Month 1), Visit 10 (Month 6). Present Difference and 95% CI change from baseline in treatment arm difference and CI separately for treatment group at each visit. Distinguish the treatment groups by different line types. | SAC [2]<br>DRY RUN [1] |
| 2.14. | ITT | EFF_F1 | Forest Plot for Odds Ratio of Percentage of Subjects Who Have Either an ACT Total Score >= 20 and/or Increase from Baseline of >= 3 in ACT Total Score at Visit 10 (Month 6) | See example display for full visual. Present each treatment comparison per page. Within the plot Favours Arm 5 should on the left and Favour Arm x on the right per page. Three odds ratios should be presented, one for each of the ACT responder models – • ACT Total Score of >=20 • ACT Total Score Increase from Baseline ≥3 • ACT Total Score of ≥ 20 and/or an Increase from Baseline of ≥ 3 | SAC [2]<br>DRY RUN [1] |

| Efficacy | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Asthma | Symptom Utility | / Index (ASUI) | | | |
| 2.15. | ITT | EFF_F3 | Summary of ASUI Total Score | Present "ASUI Total Score (Mean ± SD)" on y-axis and "Visit" on x-axis Baseline, Visit 5 (Month 1), Visit 10 (Month 6). Present mean ASUI Total Score ± SD separately for treatment group at each visit, connecting the means with a solid line. Distinguish the treatment groups by different line types. Note: Baseline ASUI total score is taken at Randomisation visit. | SAC [2]<br>DRY RUN [1] |
| 2.16. | ITT | EFF_F3 | Summary of Statistical Analysis for Change from Baseline (Randomisation) in ASUI Total Score at Visit 10 (Month 6) | (MMRM) Present "Treatment Arm Difference (95% CI) versus Arm 5" on y-axis and "Visit" on x-axis Visit 5 (Month 1), Visit 10 (Month 6). Present Difference and 95% CI change from baseline in treatment arm difference and CI separately for treatment group at each visit. Distinguish the treatment groups by different line types. | SAC [2]<br>DRY RUN [1] |
| 2.17. | ITT | EFF_F1 | Forest Plot for Odds Ratio of Percentage of Patients Meeting a Responder Threshold of ≥ 0.09 Points Improvement from Baseline (Randomisation) for the ASUI Total Score at Visit 10 (Month 6) | See example display for full visual. Present each treatment comparison per page. Within the plot Favours Arm 5 should on the left and Favour Arm x on the right per page. Odds ratio should be presented for logistic reg. analysis • ASUI | SAC [2]<br>DRY RUN [1] |

| Efficacy | /: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| St. Geo | rge's Respirator | y Questionnaire | (SGRQ) | | |
| 2.18. | ITT | EFF_F3 | Summary of SGRQ Total Score | Present "SGRQ Total Score (Mean ± SD)" on y-axis and "Visit" on x-axis Baseline, Visit 5 (Month 1), Visit 10 (Month 6). Present mean SGRQ Total Score ± SD separately for treatment group at each visit, connecting the means with a solid line. Distinguish the treatment groups by different line types. Note: Baseline SGRQ total score is taken at Randomisation visit. | SAC [2]<br>DRY RUN [1] |
| 2.19. | ΤΤ | EFF_F3 | Summary of Statistical Analysis for Change from Baseline (Randomisation) in SGRQ Total Score at Visit 10 (Month 6) | (MMRM) Present "Treatment Arm Difference (95% CI) versus Arm 5" on y-axis and "Visit" on x-axis Visit 5 (Month 1), Visit 10 (Month 6). Present Difference and 95% CI change from baseline in treatment arm difference and CI separately for treatment group at each visit. Distinguish the treatment groups by different line types. | SAC [2]<br>DRY RUN [1] |
| 2.20. | ITT | EFF_F1 | Forest Plot for Odds Ratio of Percentage of Patients Meeting a Responder Threshold of ≥ 4 Points Improvement from Baseline (Randomisation) for the SGRQ Total Score at Visit 10 (Month 6) | See example display for full visual. Present each treatment comparison per page. Within the plot Favours Arm 5 should on the left and Favour Arm x on the right per page. Odds ratio should be presented, for logistic reg. analysis • SGRQ | SAC [2]<br>DRY RUN [1] |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Fraction | nal Exhaled Nitri | c Oxide (FeNO) | and Peak Expiratory Flow (PEF) | | |
| 2.21. | ITT | EFF_F2 | Scatter Plot of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor (observed values) by Change from Baseline (Randomisation) in FeNO at Month 6 (Visit 10) | Requires the primary endpoint observed value, each treatment arm presented with a unique symbol/pattern | SAC [2]<br>DRY RUN [1] |
| 2.22. | ITT | EFF_F2 | Scatter Plot of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor (observed values) by Change from Baseline (Randomisation) in PEF at Month 6 (Visit 10) | Requires the primary endpoint observed value, each treatment arm presented with a unique symbol/pattern | SAC [2]<br>DRY RUN [1] |

# 10.8.8. Safety Tables

| Safety: Table | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse Eve | ents (AEs) | | | | |
| 3.1. | ITT | SAFE_T1 | Overview of On-Treatment and Post-Treatment Non-<br>Serious AEs leading to Withdrawal, Non-Serious ADRs and<br>SAEs | Include total column | SAC [2]<br>DRY RUN [1] |
| 3.2. | ITT | SAFE_T1 | Overview of Run-In Treatment Non-Serious AEs leading to Withdrawal, Non-Serious ADRs and SAEs | Include total column | SAC [2]<br>DRY RUN [1] |

| afety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.3. | Not in ITT | SAFE_T1 | Overview of Run-In Treatment Non-Serious AEs leading to Withdrawal, Non-Serious ADRs and SAEs for Subjects not in ITT | Total column only | SAC [2]<br>DRY RUN [1] |
| 3.4. | ITT | IDSL_AE15 | Summary of Common (>=1%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | Include total column. Do not apply rounding. Footnote: Non-serious Adverse Events includes non-serious ADRs and non-serious AEs leading to withdrawal Disclosure table. | SAC [2]<br>DRY RUN [1] |
| 3.5. | ITT | IDSL_AE15 | Summary of Common (>=1%) Run-In Treatment Non-<br>Serious Adverse Events by System Organ Class and<br>Preferred Term (Number of Subjects and Occurrences) | Include total column only. Do not apply rounding. Footnote: Non-serious Adverse Events includes nonserious ADRs and non-serious AEs leading to withdrawal Disclosure table. | SAC [2]<br>DRY RUN [1] |
| 3.6. | Not in ITT | IDSL_AE15 | Summary of Common (>=1%) Run-In Treatment Non-<br>Serious Adverse Events by System Organ Class and<br>Preferred Term (Number of Subjects and Occurrences) for<br>Subjects not in ITT | Include total column only. Do not apply rounding. Footnote: Non-serious Adverse Events includes non-serious ADRs and non-serious | SAC [2]<br>DRY RUN [1 |

| Safety: Tabl | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| | | | | AEs leading to withdrawal | |
| | | | | Disclosure table. | |
| Adverse Dru | g Reactions (AD | DRs) | | | |
| 3.7. | ITT | IDSL_AE1 | Summary of On-Treatment Adverse Drug Reactions | Include total column. All ADRs (Non-serious and Serious) | SAC [2]<br>DRY RUN [1] |
| 3.8. | ITT | IDSL_AE1 | Summary of Post-Treatment Adverse Drug Reactions | Include total column. All ADRs (Non-serious and Serious) | SAC [2]<br>DRY RUN [1] |
| 3.9. | ITT | IDSL_AE1 | Summary of On-Treatment Serious Adverse Drug Reactions | Include total column | SAC [2]<br>DRY RUN [1] |
| 3.10. | ITT | IDSL_AE1 | Summary of Post-Treatment Serious Adverse Drug<br>Reactions | Include total column | SAC [2]<br>DRY RUN [1] |
| 3.11. | ITT | IDSL_AE1 | Summary of On-Treatment Non-Serious Adverse Drug Reactions | Include total column | SAC [2]<br>DRY RUN [1] |
| 3.12. | ITT | IDSL_AE1 | Summary of Post-Treatment Non-Serious Adverse Drug Reactions | Include total column | SAC [2]<br>DRY RUN [1] |

| Safety: Table | es | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Serious Adv | erse Events (SA | Es) | | | |
| 3.13. | ITT | IDSL_AE16 | Summary of Serious Adverse Events by System Organ<br>Class and Preferred Term (Number of Subjects and<br>Occurrences) | Include total column | SAC [2]<br>DRY RUN [1] |
| 3.14. | ITT | IDSL_AE16 | Summary of Run-In Treatment Serious Adverse Events by<br>System Organ Class and Preferred Term (Number of<br>Subjects and Occurrences) | Include total column | SAC [2]<br>DRY RUN [1] |
| 3.15. | Not in ITT | IDSL_AE16 | Summary of Run-In Treatment Serious Adverse Events by<br>System Organ Class and Preferred Term (Number of<br>Subjects and Occurrences) for Subjects not in ITT | Include total column | SAC [2]<br>DRY RUN [1] |
| 3.16. | ITT | IDSL_AE1 | Summary of On-Treatment Serious Adverse Events | Include total column | SAC [2]<br>DRY RUN [1] |
| 3.17. | ITT | IDSL_AE1 | Summary of Post-Treatment Serious Adverse Events | Include total column | SAC [2]<br>DRY RUN [1] |
| Adverse Eve | ents leading to V | Vithdrawal | | 1 | |
| 3.18. | ITT | IDSL_AE1 | Summary of All On-treatment or Post-Treatment Adverse<br>Events Leading to Permanent Discontinuation of Study Drug<br>or Withdrawal from Study | Footnote: All Adverse Events includes ADRs, SAEs and Non-serious AEs leading to withdrawal Include total column | SAC [2]<br>DRY RUN [1] |

| Safety: Table | es | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.19. | ITT | IDSL_AE1 | Summary of All On-treatment or Post-Treatment Serious<br>Adverse Events Leading to Permanent Discontinuation of<br>Study Drug or Withdrawal from Study | Include total column | SAC [2]<br>DRY RUN [1] |
| 3.20. | ITT | IDSL_AE1 | Summary of On-treatment or Post-Treatment Non-Serious<br>Adverse Events Leading to Permanent Discontinuation of<br>Study Drug or Withdrawal from Study | Include total column | SAC [2]<br>DRY RUN [1] |
| 3.21. | ITT | IDSL_AE1 | Summary of On-treatment or Post-Treatment Adverse Drug<br>Reactions Leading to Permanent Discontinuation of Study<br>Drug or Withdrawal from Study | Include total column | SAC [2]<br>DRY RUN [1] |
| Adverse Eve | ents of Special Ir | nterest | | | 1 |
| 3.22. | ITT | IDSL_AE1 | Summary of On-Treatment Non-Serious Adverse Drug<br>Reactions of Special Interest | Footnote: [1] This special interest group/subgroup was defined using Special MedDRA Queries Include total column | SAC [2]<br>DRY RUN [1] |
| 3.23. | ITT | IDSL_AE1 | Summary of On-Treatment Serious Adverse Drug Reactions of Special Interest | Footnote: [1] This special interest group/subgroup was defined using Special MedDRA Queries Include total column | SAC [2]<br>DRY RUN [1] |

| Safety: Table | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.24. | ITT | IDSL_AE1 | Summary of On-Treatment Adverse Drug Reactions of Special Interest | Footnote: [1] This special interest group/subgroup was defined using Special MedDRA Queries | SAC [2]<br>DRY RUN [1] |
| | | | | Include total column | |
| 3.25. | ITT | IDSL_AE1 | Summary of On-Treatment Serious Adverse Events of Special Interest | Footnote: [1] This special interest group/subgroup was defined using Special MedDRA Queries | SAC [2]<br>DRY RUN [1] |
| | | | | Include total column | |
| Most Comm | only Reported E | vents/Reactions | | | |
| 3.26. | ITT | SAFE_T2 | Top Ten Most Commonly Reported On-Treatment Adverse Events Per Treatment Group | Footnote: All Adverse Events includes ADRs, SAEs and Non-serious AEs leading to withdrawal | SAC [2]<br>DRY RUN [1] |
| | | | | Include total column | |
| 3.27. | | ITT SAFE_T2 | Top Ten Most Commonly Reported On-Treatment Adverse | ADRs only | SAC [2]<br>DRY RUN [1] |
| J.Z1 . | ITT | | Drug Reactions Per Treatment Group | Include total column | 2777 17077[1] |

| Safety: Table | es | | | | |
|---|---|---|---|---|---|
| No. | No. Population IDSL / Example Shell | | Title | Programming Notes | Deliverable<br>[Priority] |
| Plain Langua | age Summary D | isplays | | | |
| 3.28. | ITT | IDSL_AE15 | Summary of Common (>=1%) Serious Drug-Related<br>Adverse Events by System Organ Class and Preferred<br>Term (Number of Subjects and Occurrences) | Include total column | SAC [2]<br>DRY RUN [1] |
| 3.29. | ITT | IDSL_AE15 | Summary of Common (>=1%) Non-Serious Drug-Related Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | Footnote: Non-serious Adverse Events includes non- serious ADRs and non-serious AEs leading to withdrawal Include total column | SAC [2]<br>DRY RUN [1] |

# 10.8.9. ICH Listings

| ICH: Li | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1. | Screened | IDSL_ES7 | Listing of Reasons for Screen Failure | | SAC [2] |
| 2. | Enrolled | IDSL_ES7 | Listing of Reasons for Run-in Failure | | SAC [2] |
| 3. | Screened | IDSL_ES9 | Listing of Subjects Who Were Rescreened | | SAC [2] |
| 4. | ITT | IDSL_ES2 | Listing of Reasons for Study Withdrawal | | SAC [2] |
| 5. | ITT | IDSL_SD2 | Listing of Reasons for Study Treatment Discontinuation | | SAC [2] |
| 6. | ITT | IDSL_TA1 | Listing of Planned and Actual Treatments | Planned arm is determine from the RANDALL dataset and Actual treatment arm received determine from the eCRF data | SAC [2] |
| Expos | ure | | | | |
| 7. | ITT | IDSL_EX3 | Listing of Exposure | | SAC [2] |
| Protoc | ol Deviations | | | | |
| 8. | ITT | IDSL_DV2 | Listing of Important Protocol Deviations | | SAC [2] |
| 9. | ITT | IDSL_IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC [2] |
| Demog | graphic and Bas | eline Characteris | tics | | |
| 10. | ITT | IDSL_DM2 | Listing of Demographic Characteristics | Include Height, Weight, BMI in the listing | SAC [2] |
| 11. | ITT | IDSL_DM9 | Listing of Race | | SAC [2] |

| ICH: L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | se Events | | | | |
| 12. | ITT | IDSL_AE8 | Listing of All Adverse Events | Footnote: All Adverse Events includes ADRs, SAEs and Nonserious AEs leading to withdrawal | SAC [2] |
| 13. | ITT | IDSL_AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC [2] |
| 14. | ITT | IDSL_AE2 | Listing of Relationship Between Adverse Event System Organ Class, Preferred Term and Verbatim Text | | SAC [2] |
| 15. | Not in ITT | IDSL_AE8 | Listing of All Adverse Events for Subjects not in Intent-to-Treat Population | Footnote: All Adverse Events includes ADRs, SAEs and Nonserious AEs leading to withdrawal | SAC [2] |
| Seriou | s and Other Sig | nificant Adverse | Events | | |
| 16. | ITT | IDSL_AE8 | Listing of Fatal Serious Adverse Events | Fatal and Non-Fatal SAEs are combined into a single listing for ClinPharm studies (i.e., "Listing of Serious Adverse Events"). | SAC [2] |
| 17. | ITT | IDSL_AE8 | Listing of Non-Fatal Serious Adverse Events | Fatal and Non-Fatal SAEs are combined into a single listing for ClinPharm studies (i.e., "Listing of Serious Adverse Events"). | SAC [2] |
| 18. | ITT | IDSL_AE14 | Listing of Reasons for Considering as a Serious Adverse Event | | SAC [2] |
| 19. | ITT | IDSL_AE8 | Listing of All Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | Footnote: All Adverse Events includes ADRs, SAEs and Nonserious AEs leading to withdrawal | SAC [] |

### 10.8.10. Non-ICH Listings

| Non-IC | CH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | |
| Study | Population | | | | <u> </u> |
| 20. | Enrolled | POP_L1 | Listing of Subjects Screened but Not in the Intent-to-Treat Population | | SAC [2] |
| 21. | ITT | POP_L2 | Listing of Subjects by Country | | SAC [2] |
| 22. | ITT | POP_L3 | Listing of Family History of Cardiovascular Risk Factors | | SAC [2] |
| 23. | ITT | IDSL_SU2 | Listing of Substance Use | | SAC [2] |
| 24. | ITT | POP_L4 | Listing of Asthma History | | SAC [2] |
| 25. | ITT | POP_L5 | Listing of Prescription Details | | SAC [2] |
| 26. | ITT | POP_L6 | Listing of Preferred time of dosing | | SAC [2] |
| 27. | ITT | POP_L7 | Listing of HCP Dashboard Review | | SAC [2] |
| 28. | ITT | POP_L8 | Listing of Treatment Compliance | | SAC [2] |
| Medica | al Conditions | | | | |
| 29. | ITT | IDSL_MH2 | Listing of Medical Conditions | | SAC [2] |

| Non-IC | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Conco | mitant Medicatio | ons | | | |
| 30. | ITT | IDSL_CM3 | Listing of Concomitant Medications | Note: IDSL shell in development. Required for ClinPharm studies instead of a corresponding table. Not required for studies where a table is produced. | SAC [2] |
| 31. | ITT | IDSL_CM6 | Relationship between ATC Level 1, Ingredient and Verbatim Text | | SAC [2] |
| Advers | se Events of Spe | cial Interest | | | |
| 32. | ITT | SAFE_L1 | Listing of Adverse Event of Special Interest Group,<br>Subgroup, Sub-SMQ and Preferred Term | | SAC [2] |
| Device | Malfunction | | | | |
| 33. | Enrolled | SAFE_L2 | Listing of Relvar/Breo Ellipta Sensor Status | | SAC [2] |
| 34. | Enrolled | SAFE_L3 | Listing of Salbutamol MDI Sensor Status | | SAC [2] |
| 35. | ITT | SAFE_L4 | Listing of Sensor App Status | | SAC [2] |
| 36. | ITT | SAFE_L5 | Listing of Device Malfunction | | SAC [2] |

| Non-IC | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | tle Programming Notes | |
| Efficac | ; <b>у</b> | | | | |
| 37. | ITT | EFF_L1 | Listing of Relvar/Breo ELLIPTA Adherence | | SAC [2] |
| 38. | ITT | EFF_L2 | Listing of Salbutamol MDI Rescue Free Days and Total Rescue Use | | SAC [2] |
| 39. | ITT | EFF_L3 | Listing of Patient Reported Outcome Questionnaire Total Scores – ACT, ASUI, MARS-A, PAM-13 and SGRQ | | SAC [2] |
| 40. | ITT | EFF_L3 | Listing of Patient Reported Outcome Questionnaire Total<br>Scores – BMQ | Replace the different questionnaire headings with the separate scales of the BMQ general and specific | SAC [2] |
| 41. | ITT | EFF_L4 | Listing of Severe Asthma Exacerbations | | SAC [2] |
| 42. | ITT | EFF_L5 | Listing of Unscheduled Asthma Related Healthcare Utilisation | | SAC [2] |
| 43. | ITT | EFF_L11 | Listing of Peak Expiratory Flow (PEF) and Fractional Exhaled Nitric Oxide (FeNO) Results | | SAC [2] |
| Cardio | vascular Events | (Patient profiles) | | | |
| 44. | Enrolled | IDSL_DEATH | Listing of All Cause Deaths | | SAC [2] |

#### 10.9. Appendix 9: Example Mock Shells for Data Displays

#### **STUDY POPULATION TABLES**

POP\_T1


Population: Intent-to-Treat

Table 1.4 Summary of Attendance at Each Visit

| Visit | Arm 1<br>(N=XXX) | Arm 2<br>(N=XXX) | Arm 3<br>(N=XXX) | Arm 4<br>(N=XXX) | Arm 5<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Visit 1 (Screening) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Visit 2 (Run-In) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Visit 3 (Run-In) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Visit 4 (Run-In) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Visit 5 (Month 1) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Visit 6 (Month 2) | xxx (xxx%) | N/A | xxx (xxx%) | N/A | N/A | xxx (xxx%) |
| Visit 7 (Month 3) | xxx (xxx%) | N/A | xxx (xxx%) | N/A | N/A | xxx (xxx%) |
| Visit 8 (Month 4) | xxx (xxx%) | N/A | xxx (xxx%) | N/A | N/A | xxx (xxx%) |
| Visit 9 (Month 5) | xxx (xxx%) | N/A | xxx (xxx%) | N/A | N/A | xxx (xxx%) |
| Visit 10 (Month 6) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Visit 11 (Follow-Up) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Early Withdrawal | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

Note: Visit 2/3/4 subjects may be randomised or re-entered into run-in up 3 times if ACT  $\geq$  20. Note: Visits 6/7/8/9 are Healthcare Professional Dashboard reviews for Arm 1 and Arm 3.

Protocol: 207040

Population: Intent-to-Treat


Table 1.8 Summary of Relvar/Breo ELLIPTA Sensor Status

| | Arm 1<br>(N=XXX) | Arm 2<br>(N=XXX) | Arm 3<br>(N=XXX) | Arm 4<br>(N=XXX) | Arm 5<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Number of Subjects who Activated a Sensor | xxx | XXX | xxx | xxx | xxx | XXX |
| Number of Sensors Activated | XXX | XXX | XXX | XXX | XXX | XXX |
| Was the Sensor Returned? | | | | | | |
| Yes | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| No | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Reason sensor was not returned | | | | | | |
| Lost | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Subject Lost to Follow-up | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Other | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Did the sensor malfunction? | | | | | | |
| Yes | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| No | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Did the subject permanently stop using their activated sensor during the Study | | | | | | |
| Yes | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| No | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |


Population: Intent-to-Treat

# Table 1.8 Summary of Relvar/Breo ELLIPTA Sensor Status

| | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Total |
|---|---|---|---|---|---|---|
| | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Did the subject permanently stop using sensors from the study Yes No | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

Note: Did the subject permanently stop using their activated sensor during the Study – How many activated sensors the subject permanently stopped using during the study.

Note: Did the subject permanently stop using sensors from the study - These the number of subjects who did not activate a new sensor after permanently stopping their previous sensor while still on the study.


207040


POP\_T2

Protocol: 207040

Population: Intent-to-Treat

Table 1.9 Summary of Salbutamol MDI Sensor Status

Programming note: Repeat as per Table 1.xxx


Population: Intent-to-Treat

Table 1.10 Summary of App Status

| | Arm 1<br>(N=XXX) | Arm 2<br>(N=XXX) | Arm 3<br>(N=XXX) | Arm 4<br>(N=XXX) | Arm 5<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Did subject permanently discontinue form the Sensor App during the study? | | | | | | |
| n | XXX | XXX | xxx | XXX | XXX | xxx |
| No | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Yes | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

Note: As reported by data collected in the eCRF.


Population: Intent-to-Treat

Table 1.24 Summary of Asthma Duration at Screening

| | Arm 1<br>(N=XXX) | Arm 2<br>(N=XXX) | Arm 3<br>(N=XXX) | Arm 4<br>(N=XXX) | Arm 5<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| | | | ( | | ( | |
| Duration of Asthma | | | | | | |
| n | XXX | XXX | XXX | XXX | XXX | XXX |
| < 6 months | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| >= 6 month to < 1 year | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| >= 1 year to < 5 years | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| >= 5 years to < 10 years | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| >= 10 years | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |


Example : POP\_T5 Protocol : 207040

Population : Intent-to-Treat

Table 1.25
Summary of Asthma Exacerbation History at Screening

| | Arm 1<br>(N=xxx) | Arm 2<br>(N=xxx) | Arm 3<br>(N=xxx) | Arm 4<br>(N=xxx) | Arm 5<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|---|---|
| Total number of exacerbations during the | 12 months prior to screening | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| 0 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| 1 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >1 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Number of exacerbations during the 12 m | onths prior to screening | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX | XX |

Note: Number of severe asthma exacerbations reported in the 12 months prior to Screening (Visit 1)
POP\_T5

Protocol: 207040

Population: Intent-to-Treat 

Table 1.25
Summary of Asthma Exacerbation History at Screening

| | Arm 1<br>(N=xxx) | Arm 2<br>(N=xxx) | Arm 3<br>(N=xxx) | Arm 4<br>(N=xxx) | Arm 5<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|---|---|
| Did not require oral/systemic corticosteroids (not involving hospitalisation) | | | | | | |
| . , | VV | VV | VV | VV | VV | VV |
| n<br>o | XX | XX | XX | XX | XX | XX |
| 0 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| 1 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >1 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Required oral/systemic corticosteroids (not involving hospitalisation) | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| 0 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| 1 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| ·<br>>1 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Required hospitalisation | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| <br>N | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| 1 | | | | xx (xx%) | xx (xx%) | ` , |
| 1 | xx (xx%) | xx (xx%) | xx (xx%) | , , | , , | xx (xx%) |
| >1 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

Note: Number of severe asthma exacerbations reported in the 12 months prior to Screening (Visit 1).

Example: POP\_T6 Protocol: 207040

Population: Intent-to-Treat


Table 1.26
Summary of Screening and Baseline (Randomisation) Peak Expiratory Flow (PEF)

| | | Arm 1<br>(N=XXX) | Arm 2<br>(N=XXX) | Arm 3<br>(N=XXX) | Arm 4<br>(N=XXX) | Arm 5<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|---|
| Screening Pre-<br>bronchodilator PEF<br>(L/min) | n | ххх | xxx | <br>xxx | XXX | XXX | XXX |
| | Mean | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | Min. | XX | XX | XX | XX | XX | XX |
| | Max. | XXX | XXX | XXX | XXX | XXX | XXX |
| Baseline Pre-<br>bronchodilator PEF<br>(L/min) | n | xxx | xxx | xxx | XXX | XXX | XXX |
| , | Mean | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | Min. | XX | XX | XX | XX | XX | XX |
| | Max. | XXX | XXX | XXX | XXX | XXX | XXX |


207040

Example: POP\_T6 Protocol: 207040

Population: Intent-to-Treat


Table 1.27

Summary of Screening and Baseline (Randomisation) Peak Expiratory Flow (PEF) by Country

Country: xxxxxx

Programming note: Repeat on subsequent pages by Country in alphabetical order.

Example: POP\_T6
Protocol:207040

Population: Intent-to-Treat


Table 1.28
Summary of Screening and Baseline (Randomisation) Exhaled Nitric Oxide (FeNO)

| | | Arm 1<br>(N=xx) | Arm 2<br>(N=xx) | Arm 3<br>(N=xx) | Arm 4<br>(N=xx) | Arm 5<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| Screening FeNO (ppb) | n | XXX | XXX | XXX | XXX | XXX | XXX |
| Me<br>SI<br>Me | Mean | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | Min. | XX | XX | XX | XX | XX | XX |
| | Max. | XXX | XXX | XXX | XXX | XXX | XXX |
| Baseline FeNO (ppb) | n | XXX | XXX | XXX | xxx | xxx | XXX |
| (1.7) | Mean | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | Min. | XX | XX | XX | XX | XX | XX |
| | Max. | XXX | XXX | XXX | XXX | XXX | XXX |

Example: POP\_T7: Protocol: 207040

Population: Intent-to-Treat


Table 1.38 Summary of Exposure to Study Medication

| Overall | | Arm 1<br>(N=xx) | Arm 2<br>(N=xx) | Arm 3<br>(N=xx) | Arm 4<br>(N=xx) | Arm 5<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| Exposure (days) [1] | N | XXX | XXX | XXX | XXX | XXX | xxx |
| | Mean | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | Min.<br>Max. | XX<br>XXX | XX<br>XXX | XX<br>XXX | xx | XX | XX |
| Total Subject Years (years) | | xxx | XXX | XXX | XXX | XXX | XXX |
| Range of Exposure | <= 6 weeks | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| | <= 12 weeks | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| | <= 18 weeks | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| | <= 24 weeks | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| | > 24 weeks | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |

<sup>[1]</sup> Exposure to study medication = treatment stop date – randomisation date + 1, regardless of dosage modification.

Example POP\_T8 Protocol: 207040

Population: Intent-to-Treat

Table 1.39 Summary of the Frequency of Puffs Per Day – ELLIPTA Relvar/Breo Sensor

| Period | | Arm 1<br>(N=xx) | Arm 2<br>(N=xx) | Arm 3<br>(N=xx) | Arm 4<br>(N=xx) | Arm 5<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| Baseline | Number of subjects | XX | XX | XX | XX | XX | XX |
| | Number of subject days | XX | XX | XX | XX | XX | XX |
| | 0 per day [1] | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| | 1 per day | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| | 2 per day | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| | 3 per day | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| | 4 per day | xx (%) | xx (%) | xx (%) | xx (̂%) | xx (̂%) | xx (%) |
| | >=5 per day | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| Month 1 | Number of subjects | XX | XX | XX | XX | XX | xx |
| | Number of subject days | XX | XX | XX | XX | XX | XX |
| | 0 per day [1] | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| | 1 per day | xx (%) | xx (%) | xx (%) | xx (̂%) | xx (̂%) | xx (%) |
| | 2 per day | xx (̈%) | xx (̂%) | xx (`%) | xx (̂%) | xx (̂%) | xx (̂%) |
| | 3 per day | xx (%) | xx (%) | xx (%) | xx (̂%) | xx (̂%) | xx (%) |
| | 4 per day | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| | >=5 per day | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |

Note: Number of subject days are number of days a subject has contributed to in that time period [1]: 0 per day can constitute of: No puffs recorded, Device Incidents, or Post discontinuation of ELLIPTA maintenance sensor

Programming Note: Repeat for Months 2, 3, 4, 5, 6, Months 4-6, Months 1-6 and Months 1-3.

Example POP\_T8 Protocol: 207040

Population: Intent-to-Treat


Table 1.40 Summary of the Frequency of Puffs Per Day – MDI Sensor

| Period | | Arm 1<br>(N=xx) | Arm 2<br>(N=xx) | Arm 3<br>(N=xx) | Arm 4<br>(N=xx) | Arm 5<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| Baseline | Number of subjects | XX | XX | XX | XX | XX | XX |
| | Number of subject days | XX | XX | XX | XX | XX | XX |
| | 0 per day [1] | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| | 1 per day | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| | 2 per day | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| | 3 per day | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| | 4 per day | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| | 5 per day | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| | 6 per day | xx (%) | xx (̂%) | xx (%) | xx (̂%) | xx (`%) | xx (%) |
| | 7 per day | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| | 8 per day | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| | >=9 per day | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| Month 1 | Number of subjects | XX | XX | XX | XX | XX | XX |
| | Number of subject days | XX | XX | XX | XX | XX | XX |
| | 0 per day [1] | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| | 1 per day | xx (%) | xx (̂%) | xx (`%) | xx (`%) | xx (`%) | xx (̂%) |
| | 2 per day | xx (̈%) | xx (̂%) | xx (`%) | xx (`%) | xx (`%) | xx (̂%) |
| | 3 per day | xx (%) | xx (̂%) | xx (`%) | xx (`%) | xx (`%) | xx (̂%) |
| | 4 per day | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| | 5 per day | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| | • | | • • | | | • • | • • |

Note: Number of subject days are number of days a subject has contributed to in that time period

<sup>[1]: 0</sup> per day can constitute of: No puffs recorded, Device Incidents, or Post discontinuation of MDI maintenance sensor Programming Note: Repeat for Months 2, 3, 4, 5, 6 and Months 4-6.

Example POP\_T9 Protocol:207040

Population: Intent-to-Treat


Table 1.41 Summary of Treatment Compliance

| Overall Compliance (%) | Arm 1<br>(N=xx) | Arm 2<br>(N=xx) | Arm 3<br>(N=xx) | Arm 4<br>(N=xx) | Arm 5<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|---|---|
| n | XXX | XXX | XXX | XXX | XXX | XXX |
| Mean | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| Min. | XX | XX | XX | XX | XX | XX |
| Max. | XXX | XXX | XXX | XXX | XXX | XXX |
| < 80% | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| 80% - < 100% | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| 100% - < 120% | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >=120% | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |

Example POP\_T10
Protocol:207040

Population: Intent-to-Treat


Table 1.42 Summary of Incidence of Preferred Time of Dosing Over the Treatment Period

| % | Arm 1<br>(N=xxx) | Arm 2<br>(N=xxx) | Arm 3<br>(N=xxx) | Arm 4<br>(N=xxx) | Arm 5<br>(N=xxx) |
|---|---|---|---|---|---|
| | \ / | , , | , , | , , | \ / |
| n | xxx | XXX | XXX | XXX | XXX |
| Mean | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| Min. | XX | XX | XX | XX | XX |
| Max. | XXX | XXX | XXX | XXX | XXX |

Note: A subject is considered as having taken their dose at their preferred time if the actuation time from the Relvar/Breo ELLIPTA sensor is recorded  $\pm 1$  hour of their preferred time as captured on the eCRF at screening

Example POP\_T11 Protocol:207040

Population: Intent-to-Treat


Table 1.43 Summary of HCP Dashboard Review by Visit

### Visit: Visit 5

| Actions taken post review | Arm 1<br>(N=xxx) | Arm 3<br>(N=xxx) |
|---|---|---|
| n | XXX | XXX |
| No action taken | xxx (xx%) | xxx (xx%) |
| Action Taken | xxx (xx%) | xxx (xx%) |
| Discuss adherence | xxx (xx%) | xxx (xx%) |
| Discuss rescue medication | xxx (xx%) | xxx (xx%) |
| Subject was called in for an unscheduled clinic visit | xxx (xx%) | xxx (xx%) |
| Other | xxx (xx%) | xxx (xx%) |

Programming note: Repeat subsequent pages by visits 6,7,8, 9 and 10 and Unscheduled

Example: POP\_T12 Protocol: 207040

Population: Intent-to-Treat

Table 1.44

| Summary of Asthma Maintenance Therapy | Prescription Details in the Pr | revious 12 M | onths | | |
|---|---|---|---|---|---|
| | Arm 1 | Arm 3 | Arm 4 | Arm 5 | |
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx |
| Actual number of prescriptions requested in previous 12 months | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX |
| Number of prescriptions requested/prescribed to be 100% compliant in previo | ous 12 months | | | | |
| n | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX |
| Prescription Compliance in previous 12 months (%) | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX |

Note: Prescription compliance is calculated as 100\*(Actual number of prescriptions)/(Number of prescriptions requested/prescribed to be 100% compliant)

# **STUDY POPULATION FIGURES**

Example : POP\_F1 Protocol : 207040

Population : Intent-to-Treat


Figure 1.02
Frequency of ELLIPTA Puffs Per Day

Period: Baseline



Note: 0 Puffs per day can constitute of: No puffs recorded, Device Incidents, or Post discontinuation of ELLIPTA maintenance sensor Programming Note: Repeat for Period: Month 1, 2, 3, 4, 5, 6, Month 4-6, Month 1-3, Month 1-6.

# **EFFICACY TABLES**

Example: EFF\_T1 Protocol: 207040


Population : Intent-to-Treat

Table 2.01

Summary of Monthly Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 1 and end of month 6 as determined by the maintenance sensor – Observed Monthly Data

| Month | | Arm 1<br>(N=xxx) | Arm 2<br>(N=xxx) | Arm 3<br>(N=xxx) | Arm 4<br>(N=xxx) | Arm 5<br>(N=xxx) |
|---|---|---|---|---|---|---|
| | | | • | | · | <u> </u> |
| Baseline (%) | n | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Month 1 (%) | n | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Average Month 1 to 6 (%) | n | VV | vv | VV | vv | VV |
| Average Month 1 to 0 (76) | Mean | XX | XX | XX | XX | XX |
| | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD<br>Madian | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |

Programming note: Continue table to include all monthly timelines (month 3, month 4, month 5, month 6, average month 4-6, average month 1-3, average month 1-6)

Example: EFF\_T2
Protocol: 207040

Population : Intent-to-Treat


Table 2.02

Summary of Statistical Analysis of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor

| Month 4 to 6 (%) | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 |
|---|---|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| n | XX | XX | XX | XX | XX |
| LS Mean (Std Error) | XX.X | XX.X | XX.X | XX.X | XX.X |
| CIS Arm vs Arm 5<br>Difference<br>95% C.I.<br>p-value | xx.x<br>(x.xx, x.xx)<br>xx.xxx | xx.x<br>(x.xx, x.xx)<br>xx.xxx | xx.x<br>(x.xx, x.xx)<br>xx.xxx | xx.x<br>(x.xx, x.xx)<br>xx.xxx | |

<sup>[1]</sup> Monthly adherence values were weighted by amount of observed data available and time on ELLIPTA between month 4 and 6


207040

Example : EFF\_T3

Protocol : 207040 

Population: Intent-to-Treat

Table 2.xx

Summary of Statistical Analysis of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor by Baseline ACT Total Score Group

Table 2.xx

Summary of Statistical Analysis of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor by Age Group

Example : EFF\_T4
Protocol : 207040

Population : Intent-to-Treat

Table 2.xx

Summary of Statistical Analysis of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 1 and the end of month 3 as determined by the maintenance sensor

| Month 1 to 3 (%) | Arm 1<br>(N=xxx) | Arm 2<br>(N=xxx) | Arm 3<br>(N=xxx) | Arm 4<br>(N=xxx) | Arm 5<br>(N=xxx) |
|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX |
| LS Mean (Std Error) | XX.X | XX.X | XX.X | XX.X | XX.X |
| CIS Arm vs Arm 5 | | | | | |
| Difference | XX.X | XX.X | XX.X | XX.X | |
| 95% C.I. | (x.xx, x.xx) | (x.xx, x.xx) | (x.xx, x.xx) | (x.xx, x.xx) | |
| p-value | XX.XXX | XX.XXX | XX.XXX | XX.XXX | |

Example: EFF\_T4
Protocol: 207040

Population : Intent-to-Treat

Table 2.xx

Summary of Statistical Analysis of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 1 and the end of month 6 as determined by the maintenance sensor

| Month 1 to 6 (%) | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 |
|---|---|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| n | xx | XX | XX | XX | XX |
| LS Mean (Std Error) | xx.x | XX.X | XX.X | XX.X | XX.X |
| CIS Arm vs Arm 5<br>Difference<br>95% C.I.<br>p-value | xx.x<br>(x.xx, x.xx)<br>xx.xxx | XX.X<br>(X.XX, X.XX)<br>XX.XXX | XX.X<br>(x.xx, x.xx)<br>XX.xxx | xx.x<br>(x.xx, x.xx)<br>xx.xxx | |

Example: EFF\_T5
Protocol: 207040

Population : Intent-to-Treat

Table 2.xx

Summary of Statistical Analysis of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor – Impact of Feedback of Sensor Data to HCP

| Month 4 to 6 (%) | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 |
|---|---|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| n | XX | xx | XX | XX | XX |
| LS Mean (Std Error) | XX.X | xx.x | XX.X | XX.X | XX.X |
| CIS Arm 1 vs Arm 2<br>Difference<br>95% C.I.<br>p-value | xx.x<br>(x.xx, x.xx)<br>xx.xxx | | | | |
| CIS Arm 3 vs Arm 4<br>Difference<br>95% C.I.<br>p-value | | | xx.x<br>(x.xx, x.xx)<br>xx.xxx | | |

Example: EFF\_T6
Protocol: 207040

Population : Intent-to-Treat


Table 2.xx

Summary of Statistical Analysis of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor – Impact of Feedback on Rescue Medication Use

| Month 4 to 6 (%) | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 |
|---|---|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| n | XX | XX | xx | xx | XX |
| LS Mean (Std Error) | XX.X | XX.X | xx.x | xx.x | XX.X |
| CIS Arm 1 vs Arm 3<br>Difference<br>95% C.I.<br>p-value | xx.x<br>(x.xx, x.xx)<br>xx.xxx | | | | |
| CIS Arm 2 vs Arm 4<br>Difference<br>95% C.I.<br>p-value | | xx.x<br>(x.xx, x.xx)<br>xx.xxx | | | |

Example: EFF\_T1 Protocol: 207040

Population : Intent-to-Treat

Table 2.xx

Summary of Monthly Percentage of Rescue Free Days between the beginning of month 1 and then end of month 6 as determine by the MDI rescue medication sensor

– Observed Data

| Month | | Arm 1<br>(N=xxx) | Arm 2<br>(N=xxx) | Arm 3<br>(N=xxx) | Arm 4<br>(N=xxx) | Arm 5<br>(N=xxx) |
|---|---|---|---|---|---|---|
| Deceline (0/) | | Vo. | V0/ | VV | <b>VO</b> / | VV |
| Baseline (%) | n<br>Maara | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Manda 4 (0) | _ | | | | | |
| Month 1 (%) | n | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Average Month 1 to 6 (%) | n | xx | XX | XX | XX | XX |
| Avoidge Month 1 to 6 (70) | Mean | XX.X | | | | |
| | | | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |

Programming note: Continue table to include all monthly timelines (month 2, month 3, month 4, month 5, month 6, average month 4-6)

Example: EFF\_T4
Protocol: 207040

Population : Intent-to-Treat


Table 2.xx

Summary of Statistical Analysis of Percentage of Rescue Free Days between the beginning of month 4 and then end of month 6 as determine by the MDI rescue

| Month 4 to 6 (%) | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 |
|---|---|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| n | XX | XX | XX | XX | XX |
| LS Mean (Std Error) | XX.X | XX.X | XX.X | XX.X | XX.X |
| CIS Arm vs Arm 5 | | | | | |
| Difference | xx.x | XX.X | XX.X | xx.x | |
| 95% C.I. | (x.xx, x.xx) | (X.XX, X.XX) | (X.XX, X.XX) | (x.xx, x.xx) | |
| p-value | xx.xxx | XX.XXX | XX.XXX | xx.xxx | |

medication sensor

<sup>[1]</sup> Monthly adherence values were weighted by amount of observed data available and time on ELLIPTA between month 4 and 6

Example : EFF\_T1 Protocol : 207040

 Population : Intent-to-Treat

Table 2.xx Summary of Total Rescue Use as Determined by the Maintenance Sensor

| Month | | Arm 1<br>(N=xxx) | Arm 2<br>(N=xxx) | Arm 3<br>(N=xxx) | Arm 4<br>(N=xxx) | Arm 5<br>(N=xxx) |
|---|---|---|---|---|---|---|
| Baseline | n | VV | VV | VV | VV | VV |
| Daseille | n<br>Mean | XX | XX | XX | XX | XX |
| | SD | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Month 1 | n | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Average Month 1 to 6 | n | XX | XX | XX | XX | XX |
| · | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| | IVIAA. | ** | ^^ | ^^ | ^^ | ^^ |

Programming note: Continue table to include all monthly timelines (month 2, month 3, month 4, month 5, month 6, average month 4-6)

Example: EFF\_T1
Protocol: 207040

Population : Intent-to-Treat


## Table 2.xx Summary of Asthma Control Test (ACT) Total Score

| Visit | | Arm 1<br>(N=xxx) | Arm 2<br>(N=xxx) | Arm 3<br>(N=xxx) | Arm 4<br>(N=xxx) | Arm 5<br>(N=xxx) |
|---|---|---|---|---|---|---|
| Baseline [1] | n | XX | XX | XX | XX | XX |
| Dascinic [1] | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | | | | | |
| | | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Visit 5 (Month 1) | n | xx | xx | XX | XX | XX |
| , , | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | x.xx | x.xx | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Change from Baseline at Visit 5 | n | XX | XX | XX | XX | XX |
| (Month 1) | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| , | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |

<sup>[1]</sup> Baseline ACT total score is taken at randomisation visit.

Programming note: repeat for Visit 10 (Month 6), Change from Baseline at Visit 10 (Month 6), Early Withdrawal, Change from Baseline at Early withdrawal

Example: EFF\_T4
Protocol: 207040

Population: Intent-to-Treat

Table 2.xx
Summary of the Statistical Analysis of Change from Baseline (Randomisation) in ACT Total Score at Visit 10 (Month 6)

| | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 |
|---|---|---|---|---|---|
| | (N=xxx) | (N=xxx) | N=xxx) | (N=xxx) | (N=xxx) |
| n | xx | xx | xx | xx | xx |
| LS Mean Change (SE) | xx.xx (x.xxx) | xx.xx (x.xxx) | xx.xx (x.xxx) | xx.xx (x.xxx) | xx.xx (x.xxx) |
| CIS Arm vs. Arm 5<br>Difference<br>95% CI<br>p-value | xx.x<br>(xx.x, xx.x)<br>x.xxx | xx.x<br>(xx.x, xx.x)<br>x.xxx | xx.x<br>(xx.x, xx.x)<br>x.xxx | xx.x<br>(xx.x, xx.x)<br>x.xxx | |

Note: The analysis method was an MMRM adjusted for randomised treatment arm, (visit), baseline ACT total score, randomised treatment arm-by-visit interaction, baseline ACT total score-by-visit interaction, gender, age, country and subject fitted as a random factor.

Note: The Restricted Maximum Likelihood (REML) estimation approach was used with a default covariance structure of unstructured.

Programming note: Should computational issues be encountered when using an unstructured covariance structure, other structures including AR1 and CS should be considered and the second footnote updated as appropriate.

Example : EFF\_T12
Protocol : 207040
Population : Intent-to-Treat


Table 2.xx

Summary of Percentage of Subjects Who Have Either an ACT Total Score of >= 20 and/or >= 3 Point Increase from Baseline (Randomisation) in ACT Total Score

| Visit | | Arm 1<br>(N=xxx) | Arm 2<br>(N=xxx) | Arm 3<br>(N=xxx) | Arm 4<br>(N=xxx) | Arm 5<br>(N=xxx) |
|---|---|---|---|---|---|---|
| Visit 5 (Month<br>1) | n | XXX | XXX | XXX | xxx | XXX |
| , | ACT Total Score >= 20 and/or >= 3 Point Increase from Baseline | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx<br>(xx%) | xxx (xx%) |
| | ACT Total Score >= 20 | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx<br>(xx%) | xxx (xx%) |
| | >= 3 Point Increase from Baseline | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx<br>(xx%) | xxx (xx%) |
| Visit 10 (Month 6) | n | XXX | XXX | XXX | XXX | xxx |
| 0) | ACT Total Score >= 20 and/or >= 3 Point Increase from Baseline | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx<br>(xx%) | xxx (xx%) |
| | ACT Total Score >= 20 | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx<br>(xx%) | xxx (xx%) |
| | >= 3 Point Increase from Baseline | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx<br>(xx%) | xxx (xx%) |

Example : EFF\_T13 Protocol : 207040

Population : Intent-to-Treat

Table 2.xx
Summary of the Statistical Analysis of Percentage of Subjects Who Have an ACT Total Score of ≥ 20 at Visit 10 (Month 6)

| | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 |
|---|---|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| n | xxx | xxx | xxx | xxx | xxx |
| Responder [1] | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Non-Responder | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| CIS Arm v Arm 5<br>Adjusted Odds Ratio<br>95% C.I.<br>p-value | X.XX<br>(X.XX, X.XX)<br>X.XX | x.xx<br>(x.xx, x.xx)<br>x.xx | x.xx<br>(x.xx, x.xx)<br>x.xx | x.xx<br>(x.xx, x.xx)<br>x.xx | |

Note: The analysis method was logistic regression adjusted for randomised treatment arm, baseline ACT total score, country, gender and age

<sup>[1]</sup> Responder is defined as an ACT total score >= 20.

Example : EFF\_T13 Protocol : 207040

Population : Intent-to-Treat

Table 2.xx

Summary of the Statistical Analysis of Percentage of Subjects with an Increase from Baseline (Randomisation) ≥3 in ACT Total Score at Visit 10 (Month 6)

| | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 |
|---|---|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| n | xxx | xxx | xxx | xxx | xxx |
| Responder [1] | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Non-Responder | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| CIS Arm v Arm 5<br>Adjusted Odds Ratio<br>95% C.I.<br>p-value | x.xx<br>(x.xx, x.xx)<br>x.xx | x.xx<br>(x.xx, x.xx)<br>x.xx | x.xx<br>(x.xx, x.xx)<br>x.xx | x.xx<br>(x.xx, x.xx)<br>x.xx | |

Note: The analysis method was logistic regression adjusted for randomised treatment arm, baseline ACT total score, country, gender and age

<sup>[1]</sup> Responder is defined as an increase from baseline of >= 3 in ACT total score.

Example : EFF\_T13 Protocol : 207040

Population : Intent-to-Treat

Table 2.xx

Summary of the Statistical Analysis of Percentage of Subjects Who Have Either an ACT Total Score of >=20 and/or an Increase from Baseline (Randomisation) of >=3 in ACT Total Score at Visit 10 (Month 6)

| | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 |
|---|---|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| n | xxx | xxx | xxx | xxx | xxx |
| Responder [1] | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Non-Responder | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| CIS Arm v Arm 5<br>Adjusted Odds Ratio<br>95% C.I.<br>p-value | X.XX<br>(X.XX, X.XX)<br>X.XX | x.xx<br>(x.xx, x.xx)<br>x.xx | x.xx<br>(x.xx, x.xx)<br>x.xx | x.xx<br>(x.xx, x.xx)<br>x.xx | |

Note: The analysis method was logistic regression adjusted for randomised treatment arm, baseline ACT total score, country, gender and age

<sup>[1]</sup> Responder is defined as an ACT total score >= 20 and/or an increase from baseline of >= 3.

Example : EFF\_T14
Protocol : 207040
Population : Intent-to-Treat


Table 2.xx Summary of Unscheduled Asthma Related Healthcare Resource Utilisation During the Study

| | | Arm 1<br>(N=XXX) | Arm 2<br>(N=XXX) | Arm 3<br>(N=XXX) | Arm 4<br>(N=XXX) | Arm 5<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Had unscheduled healthcare utilisation | n (%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Number of telephone calls | n<br>0<br>1<br>2<br>3<br>>3<br>Total [1] | xxx<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx | xxx<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx | xxx<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx | xxx<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx | xxx<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx |
| Number of home visits (Day) | n<br>0<br>1<br>2<br>3<br>>3<br>Total [1] | xxx<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx (%) | xxx<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx (%) | xxx<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx | xxx<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx | xxx<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx (%)<br>xxx |

<sup>[1]</sup> Total number of days/contacts across all subjects.

Example : EFF\_T14
Protocol : 207040
Population : Intent-to-Treat


Table 2.xx Summary of Unscheduled Asthma Related Healthcare Resource Utilisation During the Study

| | | Arm 1<br>(N=XXX) | Arm 2<br>(N=XXX) | Arm 3<br>(N=XXX) | Arm 4<br>(N=XXX) | Arm 5<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Number of home visits (Night) | n | XXX | XXX | XXX | XXX | XXX |
| Training of the tree (Trigging | 0 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | 1 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | 2 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | 2<br>3 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | >3 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | Total [1] | XXX | XXX | XXX | XXX | XXX |
| Number of office/practice visits | n | XXX | XXX | xxx | XXX | XXX |
| riames of ones, present visits | 0 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | 1 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | 2 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | 2<br>3 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | >3 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | Total [1] | XXX | xxx | XXX | XXX | XXX |
| Number of urgent care/outpatient visits | n | Xxx | xxx | XXX | XXX | XXX |
| <b>9</b> | 0 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | 1 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | 2 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | 3 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | >3 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | Total [1] | XXX | XXX | XXX | XXX | XXX |
| | | ,,,,, | ,,,,, | | ,,,,, | , |

<sup>[1]</sup> Total number of days/ contacts across all subjects.

Example : EFF\_T14
Protocol : 207040
Population : Intent-to-Treat


Table 2.xx Summary of Unscheduled Asthma Related Healthcare Resource Utilisation During the Study

| | | Arm 1<br>(N=XXX) | Arm 2<br>(N=XXX) | Arm 3<br>(N=XXX) | Arm 4<br>(N=XXX) | Arm 5<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Number of emergency room visits | n | XXX | XXX | XXX | XXX | XXX |
| | 0 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | 1 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | 2 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | 3 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | >3 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | Total [1] | xxx | XXX | XXX | XXX | XXX |
| Number of days inpatient hospitalisation days | n | XXX | XXX | XXX | XXX | XXX |
| , , | 0 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | 1 | xxx (̂%) | xxx (%) | xxx (̂%) | xxx (`%) | xxx (̈%) |
| | 2 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (%) |
| | 3 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (`%) |
| | >3 | xxx (%) | xxx (%) | xxx (%) | xxx (%) | xxx (`%) |
| | Total [1] | xxx ` ´ | xxx ` ´ | xxx ` ´ | xxx | xxx `´ |

<sup>[1]</sup> Total number of days/ contacts across all subjects.

Example : EFF\_T22 Protocol : 207040

Population : Intent-to-Treat


Table 2.xx Summary of Primary Care Visits relating to HCP Dashboard Review

| | Arm 1<br>(N=XXX) | Arm 2<br>(N=XXX) | Arm 3<br>(N=XXX) | Arm 4<br>(N=XXX) | Arm 5<br>(N=XXX) |
|---|---|---|---|---|---|
| Number of Subjects called in for an unscheduled clinic visit | XX | XX | XX | xx | XX |
| Number of unscheduled clinic visits | XX | XX | XX | XX | XX |

Example: EFF\_T15
Protocol: 207040


Population: Intent-to-Treat

Table 2.xx Summary of Severe On-Treatment and Post-Treatment Asthma Exacerbations

Time: On-Treatment

| | Arm 1<br>(N=xxx) | Arm 2<br>(N=xxx) | Arm 3<br>(N=xxx) | Arm 4<br>(N=xxx) | Arm 5<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|---|---|
| No. of subjects with one or more severe asthma exacerbation | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Total no. of severe asthma exacerbations | XX | XX | XX | XX | XX | XX |
| Number of severe asthma exacerbations per subject 0 1 > 1 | xx (xx%)<br>xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%)<br>xx (xx%) |
| Duration of severe asthma exacerbation (days) [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX | XX |

<sup>[1]</sup> Summary only includes exacerbations for which a date of onset and resolution were provided in the eCRF. Programming Note: Repeat for Post-Treatment


Example : EFF\_T15 Protocol : 207040

Population : Intent-to-Treat

Table 2.xx

Summary of Severe On-Treatment and Post-Treatment Asthma Exacerbations

Time: On-Treatment

| | Arm 1<br>(N=xxx) | Arm 2<br>(N=xxx) | Arm 3<br>(N=xxx) | Arm 4<br>(N=xxx) | Arm 5<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|---|---|
| No. of subjects with an expecthation outcome | | | | | | |
| No. of subjects with an exacerbation outcome Resolved | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Fatal | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Not resolved | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| No. of subjects with exacerbations: | | | | | | |
| Requiring use of systemic/oral corticosteroids | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Leading to hospitalisation | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Requiring emergency room visit | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| No. of subjects with exacerbations requiring intubation | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| No. of subjects with exacerbations leading to withdrawal from study | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Annual severe asthma exacerbation rate [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX | XX |

<sup>[1]</sup> Summary only includes exacerbations for which a date of onset and resolution were provided in the eCRF..

Example EFF\_T1 Protocol : 207040

Population : Intent-to-Treat


Table 2.xx Summary of Asthma Symptom Utility Index (ASUI) Score

| Visit | | Arm 1<br>(N=xxx) | Arm 2<br>(N=xxx) | Arm 3<br>(N=xxx) | Arm 4<br>(N=xxx) | Arm 5<br>(N=xxx) |
|---|---|---|---|---|---|---|
| Baseline [1] | n | XX | XX | XX | XX | XX |
| [] | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | xx | XX | XX | XX | XX |
| Visit 5 (Month 1) | n | XX | XX | XX | XX | XX |
| , | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | x.xx | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | xx | XX | XX | XX | XX |
| Change from Baseline at Visit 5 | n | XX | XX | XX | XX | XX |
| (Month 1) | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| , | SD | X.XX | x.xx | X.XX | x.xx | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |

<sup>[1]</sup> Baseline ASUI total score is taken at randomisation visit.

Programming note: repeat, Visit 10 (Month 6), Change from Baseline at Visit 10 (Month 6), Early Withdrawal

Example EFF\_T16

Protocol : 207040 

Population : Intent-to-Treat

Table 2.xx

Summary of Statistical Analysis of Percentage of Subjects Meeting a Responder Threshold of 0.09 Points Improvement (Increase) from Baseline (Randomisation) for the ASUI Total Score at Visit 10 (Month 6)

| | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 |
|---|---|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| n | xxx | xxx | xxx | xxx | xxx |
| Responder [1] | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Non-Responder | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| CIS Arm v Arm 5<br>Adjusted Odds Ratio<br>95% C.I.<br>p-value | X.XX<br>(X.XX, X.XX)<br>X.XX | x.xx<br>(x.xx, x.xx)<br>x.xx | x.xx<br>(x.xx, x.xx)<br>x.xx | x.xx<br>(x.xx, x.xx)<br>x.xx | |

Note: The analysis method was logistic regression adjusted for randomised treatment arm, baseline ASUI total score, country, gender and age

<sup>[1]</sup> Responder is defined as an ASUI total score >= 0.09 points increase from baseline.


Example: EFF\_T4
Protocol: 207040

Population: Intent-to-Treat

Table 2.xx

Summary of the Statistical Analysis of Change from Baseline (Randomisation) in Asthma Symptom Utility Index (ASUI) Total Score at Visit 10 (Month 6)

| | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 |
|---|---|---|---|---|---|
| | (N=xxx) | (N=xxx) | N=xxx) | (N=xxx) | (N=xxx) |
| n | xx | xx | xx | xx | xx |
| LS Mean Change (SE) | xx.xx (x.xxx) | xx.xx (x.xxx) | xx.xx (x.xxx) | xx.xx (x.xxx) | xx.xx (x.xxx) |
| CIS Arm vs. Arm 5<br>Difference<br>95% CI<br>p-value | xx.x<br>(xx.x, xx.x)<br>x.xxx | xx.x<br>(xx.x, xx.x)<br>x.xxx | xx.x<br>(xx.x, xx.x)<br>x.xxx | xx.x<br>(xx.x, xx.x)<br>x.xxx | |

Note: The analysis method was an MMRM adjusted for randomised treatment arm, visit, baseline ASUI total score, randomised treatment arm-by-visit interaction, baseline ASUI total score-by-visit interaction, gender, age, country and subject fitted as a random factor.

Note: The Restricted Maximum Likelihood (REML) estimation approach was used with a default covariance structure of unstructured.

Programming note: Should computational issues be encountered when using an unstructured covariance structure, other structures including AR1 and CS should be considered and the second footnote updated as appropriate.

Example : EFF\_T1
Protocol : 207040
Population : Intent-to-Treat


Table 2.xx Summary of St. George's Respiratory Questionnaire (SGRQ) Total Score

| Visit | | Arm 1<br>(N=xxx) | Arm 2<br>(N=xxx) | Arm 3<br>(N=xxx) | Arm 4<br>(N=xxx) | Arm 5<br>(N=xxx) |
|---|---|---|---|---|---|---|
| Baseline [1] | n | xx | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | x.xx | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Visit 5 (Month 1) | n | XX | XX | XX | XX | XX |
| , | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | x.xx | X.XX | x.xx | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Change from Baseline at Visit 5 | n | XX | XX | XX | XX | XX |
| (Month 1) | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| , | SD | X.XX | x.xx | X.XX | x.xx | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |

<sup>[1]</sup> Baseline SGRQ total score is taken at randomisation visit

Programming note: repeat for Visit 10 (Month 6), Change from Baseline at Visit 10 (Month 6), Early Withdrawal


Example : EFF\_T13 Protocol : 207040

Population : Intent-to-Treat

Table 2.xx

Summary of the Statistical Analysis of Percentage of Subjects Meeting a Responder Threshold of ≥4 Points Improvement (Decrease) from Baseline (Randomisation) for the SGRQ Total Score at Visit 10 (Month 6)

| | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 |
|---|---|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| n | xxx | xxx | xxx | xxx | xxx |
| Responder [1] | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Non-Responder | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| CIS Arm v Arm 5<br>Adjusted Odds Ratio<br>95% C.I.<br>p-value | X.XX<br>(X.XX, X.XX)<br>X.XX | x.xx<br>(x.xx, x.xx)<br>x.xx | x.xx<br>(x.xx, x.xx)<br>x.xx | x.xx<br>(x.xx, x.xx)<br>x.xx | |

Note: The analysis method was logistic regression adjusted for randomised treatment arm, baseline SGRQ total score, country, gender and age

<sup>[1]</sup> Responder is defined as SGRQ total score >= 4 points decrease from baseline.

Example : EFF\_T Protocol : 207040


Population : Intent-to-Treat

Table 2.xx
Summary of the Statistical Analysis of Change from Baseline (Randomisation) in SGRQ at Visit 10 (Month 6)

| | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 |
|---|---|---|---|---|---|
| | (N=xxx) | (N=xxx) | N=xxx) | (N=xxx) | (N=xxx) |
| n | xx | xx | xx | xx | xx |
| LS Mean Change (SE) | xx.xx (x.xxx) | xx.xx (x.xxx) | xx.xx (x.xxx) | xx.xx (x.xxx) | xx.xx (x.xxx) |
| CIS Arm vs. Arm 5<br>Difference<br>95% CI<br>p-value | xx.x<br>(xx.x, xx.x)<br>x.xxx | xx.x<br>(xx.x, xx.x)<br>x.xxx | xx.x<br>(xx.x, xx.x)<br>x.xxx | xx.x<br>(xx.x, xx.x)<br>x.xxx | |

Note: The analysis method was an MMRM adjusted for randomised treatment arm, visit, baseline SGRQ total score, randomised treatment arm-by-visit interaction, baseline SGRQ total score-by-visit interaction, gender, age, country and subject fitted as a random factor.

Note: The Restricted Maximum Likelihood (REML) estimation approach was used with a default covariance structure of unstructured.

Programming note: Should computational issues be encountered when using an unstructured covariance structure, other structures including AR1 and CS should be considered and the second footnote updated as appropriate.

Example : EFF\_T1
Protocol : 207040
Population : Intent-to-Treat


Table 2.xx Summary of Patient Activation Measure (PAM) 13 Total Score

| Visit | | Arm 1<br>(N=xxx) | Arm 2<br>(N=xxx) | Arm 3<br>(N=xxx) | Arm 4<br>(N=xxx) | Arm 5 (N=xxx) |
|---|---|---|---|---|---|---|
| Baseline [1] | n | xx | XX | XX | XX | XX |
| Dascinic [1] | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Visit 5 (month 1) | n | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |

<sup>[1]</sup> Baseline PAM-13 total score is taken from Screening Visit

Programming note: repeat for Randomisation Visit, Change from Baseline at Visit 5 (Month 1), Visit 10 (Month 6), Change from Baseline at Visit 10 (Month 6), Early Withdrawal

Note: The total PAM score is calculated by dividing the raw score over the number of items answered and multiplied by 13. This score is then transformed to a scale within a range of 0-100 based on calibration tables and proprietary PAM algorithm.

Example : EFF\_T28
Protocol : 207040
Population : Intent-to-Treat


Table 2.xx Summary of Medication Adherence Report Scale - Asthma (MARS-A) Total Score

| Visit | | Arm 1<br>(N=xxx) | Arm 2<br>(N=xxx) | Arm 3<br>(N=xxx) | Arm 4<br>(N=xxx) | Arm 5<br>(N=xxx) |
|---|---|---|---|---|---|---|
| Baseline [1] | n | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | x.xx | X.XX | x.xx | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Visit 5 (Month 1) | n | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |

<sup>[1]</sup> Baseline MARS-A 10 total score is taken from screening visit.

Note: MARS-A 10 Total Score is based on the mean score across all ten questions per visit.

Programming note: repeat for Randomisation visit, Change from Baseline at Visit 5 (Month 1), Visit 10 (Month 6), Change from Baseline at Visit 10 (Month 6), Early Withdrawal

EFF\_T19 Protocol:207040 Population: Intent-to-Treat


Table 2.xx Summary of Beliefs in Medicine Questionnaire (BMQ) General Benefit Total Score

| Visit | | Arm 1<br>(N=xxx) | Arm 2<br>(N=xxx) | Arm 3<br>(N=xxx) | Arm 4<br>(N=xxx) | Arm 5<br>(N=xxx) |
|---|---|---|---|---|---|---|
| D 1: 141 | | | | | | |
| Baseline [1] | n | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Visit 5 (Month 1) | n | xx | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |

[1] Baseline BMQ total score is taken from screening visit.

Note: BMQ Score is based on the total score across all items within the BMQ measure

Programming note: repeat for Randomisation visit, Change from Baseline at Visit 5 (Month 1), Visit 10 (Month 6), Change from Baseline at Visit 10 (Month 6), Early Withdrawal

#### Repeat for:

Table 2.28 Summary of Beliefs in Medicine Questionnaire (BMQ) General Harm Total Score Programming note: Use the items as presented in RAP

Table:2.29 Summary of Beliefs in Medicine Questionnaire (BMQ) General Overuse Total Score

Programming note: Use the items as presented in RAP

Table: 2.30 Summary of Beliefs in Medicine Questionnaire (BMQ) Specific Necessity Total Score

Programming note: Use the items as presented in RAP

Table:2.31 Summary of Beliefs in Medicine Questionnaire (BMQ) Specific Concern Total Score

Programming note: Use the items as presented in RAP

EFF\_T21 Protocol:207040

Population: Intent-to-Treat


Table 2.xx Summary of Medical Device Incidents (Sensors)

| | | Arm 1<br>(N=xxx) | Arm 2<br>(N=xxx) | Arm 3<br>(N=xxx) | Arm 4<br>(N=xxx) | Arm 5<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|---|---|---|
| Relvar/Breo ELLIPTA Sensor | Number of incidents<br>Subjects with at least one<br>incident | xxx<br>xxx (xx%) | xxx<br>xxx (xx%) | xxx<br>xxx (xx%) | xxx<br>xxx (xx%) | xxx<br>xxx (xx%) | xxx<br>xxx (xx%) |
| SABA MDI Sensor | Number of incidents<br>Subjects with at least one<br>incident | xxx<br>xxx (xx%) | xxx<br>xxx (xx%) | xxx<br>xxx (xx%) | xxx<br>xxx (xx%) | xxx<br>xxx (xx%) | xxx<br>xxx (xx%) |

Note: Devices incidents are classed as sensor malfunctions as noted in the eCRF.

EFF\_T1
Protocol:207040
Population: Intent-to-Treat


Table 2.xx Summary of Fractional Exhaled Nitric Oxide (FeNO)

| Visit | | Arm 1<br>(N=xxx) | Arm 2<br>(N=xxx) | Arm 3<br>(N=xxx) | Arm 4<br>(N=xxx) | Arm 5<br>(N=xxx) |
|---|---|---|---|---|---|---|
| Baseline [1] | n | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | xx | XX | XX | XX | XX |
| Visit 5 (Month 1) | n | XX | XX | XX | XX | XX |
| , | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Change from Baseline at Visit 5 | n | XX | XX | XX | XX | XX |
| ŭ | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |

<sup>[1]</sup> Baseline FeNO reading is taken from the Randomisation visit.

Programming note: repeat for Screening visit, Visit 10 (Month 6), Change from Baseline at Visit 10 (Month 6), 4, Early Withdrawal,


EFF\_T23 Protocol:207040

Population: Intent-to-Treat

Table 2.xx

Summary of Change from Baseline (Randomisation) in Fractional Exhaled Nitric Oxide (FeNO) at Month 6 (Visit 10) by Percentage of ELLIPTA doses taken (daily adherence) between the beginning of Month 4 and the end of Month 6 Group

Adherence: <range of quartile %>

| Visit | | Arm 1<br>(N=xxx) | Arm 2<br>(N=xxx) | Arm 3<br>(N=xxx) | Arm 4<br>(N=xxx) | Arm 5<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|---|---|---|
| Baseline | n | XX | XX | XX | XX | XX | XX |
| Buschile | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | | | | | | |
| | | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX | XX |
| Visit 10 (Month 6) | n | XX | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX | XX |
| Change from Baseline at Visit 10 | n | XX | XX | XX | XX | XX | XX |
| 3 | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | x.xx | X.XX | x.xx |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX | XX |
| | Max. | /// | /// | <b>XX</b> | <b>A</b> A | <b>7</b> /1 | <b>AA</b> |

EFF\_T23

Protocol:207040

Population: Intent-to-Treat


Table 2.xx

Summary of Change from Baseline (Randomisation) in Peak Expiratory Flow (PEF) at Month 6 (Visit 10) by Percentage of ELLIPTA doses taken (daily adherence) between the beginning of Month 4 and the end of Month 6 Group

Adherence: <range of quartile %>

| Visit | | Arm 1<br>(N=xxx) | Arm 2<br>(N=xxx) | Arm 3<br>(N=xxx) | Arm 4<br>(N=xxx) | Arm 5<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|---|---|---|
| Baseline | n | XX | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | x.xx | x.xx | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX | XX |
| | Max. | XX | XX | xx | XX | XX | XX |
| Visit 10 (Month 6) | n | XX | XX | XX | XX | XX | XX |
| visit to (Month o) | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | | | | | | |
| | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX | XX |
| Change from Baseline at Visit 10 | n | XX | XX | xx | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX | XX |
| FFF T1 | | 701 | 701 | 701 | 701 | 701 | 701 |

EFF\_T1

Protocol:207040


Population: Intent-to-Treat

Table 2.xx Summary of Peak Expiratory Flow (PEF) (Litres/min)

| Visit | | Arm 1<br>(N=xxx) | Arm 2<br>(N=xxx) | Arm 3<br>(N=xxx) | Arm 4<br>(N=xxx) | Arm 5<br>(N=xxx) |
|---|---|---|---|---|---|---|
| Baseline [1] | n | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | xx | XX | XX | XX | XX |
| Visit 5 (Month 1) | n | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | xx | xx | XX | XX | XX |
| Change from Baseline at Visit 5 | n | XX | XX | XX | XX | XX |
| 3 | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |

[1] Baseline PEF reading is taken from the randomisation visit.

Programming note: repeat for Visit 10 (Month 6), Change from Baseline at Visit 10 (Month 6), 4, Early Withdrawal

#### **EFFICACY FIGURES**

Example: EFF\_F1 Protocol: 207040

Protocol: 207040 
Population: Intent-to-Treat

Figure 2.xx

Forest Plot for Odds Ratio of Either an ACT Total Score >= 20 and/or Increase from Baseline of >= 3 in ACT Total Score at Visit 10 (Month 6)

Treatment Group: Arm 1



\*=Proportion of responders, defined as ACT Total Score >= 20 and/ or Increase from Baseline of >= 3 in ACT Total Score at Visit 10 (Month 6)

Note: The analysis method was logistic regression adjusted for randomised treatment arm, baseline ACT total score, country, gender and age

Programming note: page 1 comparison between Arm 5 and Arm 1, following pages present the remaining Arm 5 v 2,3,4 treatment arm comparison

Example: EFF\_F2 Protocol: 207040

Population: Intent-to-Treat


Figure 2.xx

Scatter Plot of Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor (Observed values) by Age



Programming Note: Requires the primary endpoint observed value, each treatment arm presented with a unique symbol/pattern. Be consistent with symbols/colours across all figures.


Example: EFF\_F3 Protocol: 207040

Population: Intent-to-Treat

Figure 2.xx
Summary of Statistical Analysis for Change from Baseline (Randomisation) in ACT Total Score at Month 6



Programming Note: Present "Change from Baseline ACT Total Score" on y-axis and "Visit" on x-axis Baseline, Visit 5 (Month 1), Visit 10 (Month 6). Present mean ACT Total Score +- SD separately for treatment group at each visit, connecting the means with a solid line. Distinguish the treatment groups by different line types.


Example: EFF\_F4
Protocol: 207040

Population: Intent-to-Treat

Figure 2.xx
Summary of Interaction Tests for Percentage of ELLIPTA doses taken (daily adherence) between the beginning of month 4 and the end of month 6 as determined by the maintenance sensor - - Comparisons Arm 1,2,3,4 v Arm 5



Note: The results displays are from an ANCOVA adjusted for randomised treatment arm, baseline adherence, duration of run-in (visits), country, gender

[1] age (years), covariate, and two-way interaction between randomised treatment arm and covariate

[2] covariate, two-way interaction between randomised treatment group and covariate.

Example: EFF\_F5

Protocol: 207040 

Population: Intent-to-Treat

Figure 2.xx
Box plot of Monthly Percentage of ELLIPTA doses taken (daily adherence) as determined by the maintenance sensor



Analysis Month

Note: Baseline adherence is calculated using up to the last 28 days of daily adherence data during the run-in period.

#### **SAFETY TABLES**

Example: SAFE\_T1 Page 1 of X Protocol: 207040

Population: Intent-to-Treat

Table 3.1 Overview of On-Treatment and Post-Treatment Non-Serious AEs leading to Withdrawal, Non-Serious ADRs and SAEs

| | Arm 1<br>(N=XXX) | Arm 2<br>(N=XXX) | Arm 3<br>(N=XXX) | Arm 4<br>(N=XXX)) | Arm 5<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Any Non-Serious AE | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Any Non-Serious ADR's | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Any On-Treatment Non-Serious ADRs | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Any Post-Treatment Non-Serious ADRs | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Any AEs leading to permanent discontinuation of study drug or withdrawal from study [1] | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Any SAE | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Any On-Treatment SAEs | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Any Post-Treatment SAEs | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Any On-Treatment Serious ADRs | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Any Post-Treatment Serious ADRs | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Any On-Treatment Fatal SAEs | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Any Post-Treatment Fatal SAEs | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |

Footnote: [1] Includes both on-treatment and post-treatment Non-Serious Adverse events leading to withdrawal, Non-serious ADRs and SAEs


SAFE\_T2: Protocol: 207040

Population: Intent-to-Treat

Table 3.xx
Top Ten Most Commonly Reported On-Treatment Adverse Events Per Treatment Group

| Dictionary-Derived Term | Arm 1<br>(N=XXX) | Arm 2<br>(N=XXX) | Arm 3<br>(N=XXX) | Arm 4<br>(N=XXX) | Arm 5<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Viral upper respiratory tract infection | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Headache | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Chronic obstructive pulmonary disease | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Upper respiratory tract infection | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Influenza | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Pneumonia | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Pharyngitis | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Back pain | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Hypertension | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Bronchitis | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Cough | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

Note: The 10 most frequent preferred terms in Arm 1, Arm 2, Arm 3, Arm 4 and Arm 5.


SAFE\_T2:
Protocol: 207040

Population: Intent-to-Treat

Table 3.xx
Top Ten Most Commonly Reported On-Treatment Adverse Drug Reactions Per Treatment Group

| Dictionary-Derived Term | Arm 1<br>(N=XXX) | Arm 2<br>(N=XXX) | Arm 3<br>(N=XXX) | Arm 4<br>(N=XXX) | Arm 5<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Viral company and instance tracet infection | , (, o, 0/ ) | var (var0/ ) | var (var0/ ) | \\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\ | \\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\ | vo. (vo.0/ ) |
| Viral upper respiratory tract infection<br>Headache | xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%) |
| Chronic obstructive pulmonary disease | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Upper respiratory tract infection | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Influenza | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Pneumonia | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Pharyngitis | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Back pain | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Hypertension | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Bronchitis | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

Note: The 10 most frequent preferred terms in Arm 1, Arm 2, Arm 3, Arm 4 and Arm 4, and the 10 most frequent in Arm 5 are presented.

#### **LISTINGS**

POP\_L1

Protocol: 207040
Population: Enrolled

## Listing xx Listing of Subjects Screened but Not in the Intent-to-Treat Population

| Treatment | Site Id./<br>Unique Subject Id. | Disposition Status | Reason for Screen Failure/Run-in/Withdrawal |
|---|---|---|---|
| Arm 1 | xxxxxx/<br>xxxxxx.xxxxxxxxxxxxxxxxxxxxxxxx | Early Withdrawal | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | xxxxxx/<br>xxxxxx.xxxxxxxxxxxxxxxxxxxxxxxx | Early Withdraw | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| Arm 3 | xxxxxx/<br>xxxxxx.xxxxxx | Early Withdrawal | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | xxxxxx/<br>xxxxxx.xxxxxxxxxxxx | Early Withdraw | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| Non Treatment | xxxxxx/<br>xxxxxx.xxxxxxx | Screen Failure | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | xxxxxx/<br>xxxxxx.xxxxxxxxxxxxxxxxxxxxxxxx | Rin-in Failure | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

POP\_L2


Population: Intent-to-Treat

#### Listing xx Listing of Subjects by Country

| Country | Investigator<br>Name | Subject | Treatment Arm |
|----------------|----------------------|---------|---------------|
| Netherlands | PPD | | ARM1 |
| | | | ARM3 |
| | | | ARM4 |
| United Kingdom | | | ARM2 |

POP\_L3


Population: Intent-to-Treat

Listing xx
Listing of Family History of Cardiovascular Risk Factors

| Site Id. | J | |
|----------|-----------------|--------------------|
| Unique | Subject Id. ARM | Family History [1] |
| PPD | | |
| | ARM1 | Yes |
| | | Unknown |
| | ARM3 | Unknown |
| | | Yes |
| | ARM4 | Unknown |

Footnote: [1] Family history of premature coronary artery disease in women < 65 years or men < 55 years in first degree relatives only (e.g., biological mother or father, biological brother or sister, biological son or daughter).

POP\_L4

Protocol: 207040

Population: Intent-to-Treat


### Listing xx Listing of Asthma History

| | | | | Number of Asthma | | |
|---|---|---|---|---|---|---|
| | | | Dura | tion of Asthma | | ons in Last 12 Months_ |
| Treatment | Inv. | Subj. | Years | Months | Type 1^ | Type 2# |
| Arm 1 | xxxxx | XXXX | XX | XX | XX | xx |
| | | XXXX | XX | XX | XX | XX |
| | | XXXX | XX | XX | XX | XX |
| | | XXXX | XX | XX | XX | XX |
| | XXXXX | XXXX | XX | XX | XX | XX |
| | | XXXX | XX | XX | XX | XX |
| | | XXXX | XX | XX | XX | XX |
| | | XXXX | XX | XX | XX | xx |
| Arm 2 | XXXXX | XXXX | XX | XX | XX | XX |
| | | XXXX | XX | XX | XX | XX |
| | | XXXX | XX | XX | XX | XX |
| | | XXXX | XX | XX | XX | XX |
| | XXXXX | XXXX | XX | XX | XX | XX |
| | | XXXX | XX | XX | XX | XX |
| | | XXXX | XX | XX | XX | XX |
| | | XXXX | XX | XX | XX | XX |

<sup>^</sup>Type 1: Required oral/systemic corticosteroids (not involving hospitalization) #Type 2: Required hospitalization

POP\_L5 Protocol:207040 Population: All Subjects Enrolled


Listing xx Listing of Prescription Details

| Site Id./<br>Unique Subject Id. | Actual number of prescriptions [1] | Number of prescriptions needing 100% compliance [2] |
|---|---|---|
| PPD | 4 | 11 |
| | 8 | 5 |

<sup>[1]</sup> Actual number of asthma maintenance therapy prescriptions requested by subject or prescribed for subject.

<sup>[2]</sup> Number of asthma maintenance therapy prescriptions requested or prescribed that would be needed to be 100% compliant.

POP\_L6


Population: Intent-to-Treat

Listing xx
Listing of Preferred time of dosing

| Site Id<br>Unique | l./ Treatment Arm<br>e Subject Id. | Preferred time | Incidence of Preferred time (%) |
|---|---|---|---|
| PPD | 1 | 15:30 | 57.34% |
| | 2 | 9:00 | 89.23% |

Note: A subject is considered as having taken their dose at their preferred time if the actuation time from the Relvar/Breo ELLIPTA sensor is recorded  $\pm 1$  hour of their preferred time as captured on the eCRF at screening

POP\_L7 Protocol:207040 Population: Intent-to-Treat


Listing xx
Listing of HCP Dashboard Review

| | ite Id./<br>nique Subject Id. | Treatment | Visit | Date of Dashboard data review | Was action taken | Action(s) Taken |
|---|---|---|---|---|---|---|
| PP | D | Arm 4 | Xxxxxxx | 12DEC2008 | N | Discuss adherence |
| | | Arm 2 | xxxxxx | 03FEB2009 | Υ | Discuss rescue medication |


Population: Intent-to-Treat

Listing xx Listing of Treatment Compliance

| Site Id. | / Protocol Subject Id. prescribed dose | Start Date/<br>Study Day | Stop Date/<br>Study Day | Overall Compliance |
|---|---|---|---|---|
| Onique | | | Study Day | |
| PPD | 200/25 mcg QD | PPD | PPD | 71 |
| | ŭ | 1 | 1 | |
| | 200/25 mcg QD | PPD | PPD | 107 |
| | | 1 | 1 | |

Protocol: 207040

Population: Intent-to-Treat


## Listing xx Listing of Adverse Event of Special Interest Group, Subgroup, Sub-SMQ and Preferred Term

| AESI Group | AESI Subgroup | Sub-SMQ | Preferred Term |
|---|---|---|---|
| Adrenal suppression | | | ACTH stimulation test abnormal<br>Addison's disease<br>Adrenal androgen deficiency<br>Adrenal atrophy<br>Adrenal insufficiency |


Population: ITT

Listing xx Listing of Relvar/Breo ELLIPTA Sensor Status

| Site id/<br>Subj. | atment | Date of Sensor activation | Serial<br>Number | Sensor<br>return<br>status | Sensor return date | Reasons for not returning the Sensor | Date of Sensor malfunction | permanently stopping the use of Sensor |
|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|

PPD

Population: Enrolled

Listing xx Listing of Salbutamol MDI Sensor Status

| Site id/<br>Subj. | Treatment | Date of Sensor activation | Serial<br>Number | Sensor<br>return<br>status | Sensor<br>return date | Reasons for not returning the Sensor | Date of Sensor malfunction | Date of permanently stopping the use of Sensor |
|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|

PPD

SAFE\_L4


Population: Intent-to-Treat

Listing xx Listing of Sensor App Status

| Site id./<br>Subj. | Arm | Date of permanent discontinuation/study day |
|--------------------|-------|---------------------------------------------|
| PPD | Arm 1 | PPD 23 |
| | Arm 5 | PPD 43 |

SAFE\_L5 Protocol: 207040

Page 1 of x Population: ITT

# Listing xx Listing of Device Malfunction

| Site id.<br>Subj. | / Arm | Date of malfunction | Malfunctioning device type | Reasons for device malfunction |
|---|---|---|---|---|
| PPD | Arm 2 | 07FEB2008 | ELLIPTA | Dose counter is ambiguous |
| | Arm 4 | 12FEB2008 | Rescue Medication | Inhaler is cracked or broken apart |

EFF\_L1 Protocol: 207040

Protocol: 207040
Population: Intent-to-Treat

Listing xx
Listing of Relvar/Breo ELLIPTA Adherence – Observed Data

| | Site id./<br>Subj. | Arm | Month | Day | | Number of Days | Adherence (%) |
|---|---|---|---|---|---|---|---|
| PPD | Arm 2 | Baseline | Adherence | recorded | 28 | 100% | |
| | | | Device inc | ident | 0 | | |
| | | | Post disco | ntinuation of maintenance Sensor | 0 | | |
| | | | Non-adher | ent | 0 | | |
| | | Month 1 | Adherence | recorded | 20 | 71.42% | |
| | | | Device inc | ident | 0 | | |
| | | | Post disco | ntinuation of maintenance Sensor | 0 | | |
| | | | Non-adher | ent | 8 | | |
| | Arm 4 | Baseline | Adherence | recorded | 28 | 100% | |
| | | | Device inc | ident | 0 | | |
| | | | Post disco | ntinuation of maintenance Sensor | 0 | | |
| | | | Non-adher | ent | 0 | | |
| | | Month 1 | Adherence | recorded | 18 | | |
| | | | Device inc | ident | 1 | | |
| | | | Post disco | ntinuation of maintenance Sensor | 0 | | |
| | | | Non-adher | ent | 9 | | |

Programming Note: Repeat for Month 2, 3, 4, 5 and 6


EFF\_L2 Protocol: 207040

Population: Intent-to-Treat

Listing xx
Listing of Salbutamol MDI Rescue Free Days and Total Rescue Use – Observed Data

| Site id./<br>Subj. | Arm | Month | Day | Number of Days | Rescue Free (%) | Total Rescue Use (Puffs) |
|---|---|---|---|---|---|---|
| PPD | Arm 1 | Baseline | Rescue use recorded | 9 | 67.86% | 15 |
| | | | Device incident | 0 | | |
| | | | Post discontinuation of MDI rescue sensor | 0 | | |
| | | | MDI rescue free | 19 | | |
| | | Month 1 | Rescue use recorded | 20 | 28.58% | 42 |
| | | | Device incident | 0 | | |
| | | | Post discontinuation of MDI rescue sensor | 0 | | |
| | | | MDI rescue free | 8 | | |
| | Arm 3 | Baseline | Rescue use recorded | 0 | 100% | 0 |
| | | | Device incident | 0 | | |
| | | | Post discontinuation of MDI rescue sensor | 0 | | |
| | | | MDI rescue free | 28 | | |
| | | Month 1 | Rescue use recorded | 18 | | 29 |
| | | | Device incident | 1 | | |
| | | | Post discontinuation of MDI rescue sensor | 0 | | |
| | | | MDI rescue free | 9 | | |

Programming Note: Repeat for Month 2, 3, 4, 5 and 6

EFF\_L3


Population: ITT

Listing xx
Listing of Patient Reported Outcome Questionnaire Total Scores

Treatment: Arm 1

| | Visit/ | | | Total Score | | | |
|---------|-------------|-----|------|-------------|--------|------|-----|
| Inv./ | Study Date/ | | | | | | |
| Subj. | Study Day | ACT | ASUI | MARS-A | PAM-13 | SGRQ | BMQ |
| xxxxxx/ | XXXXX | | | | | | |
| XXXXX | DDMMMYYYY/ | | | | | | |
| | XX | | | | | | |

EFF\_L4


Population: Intent-to-Treat

# Listing xx Listing of Severe Asthma Exacerbations

| Treatment/ Inv./<br>Subj. | Days Since<br>1st Dose of<br>Onset | Date of<br>Onset/<br>Resolution | Outcome | Withdrawn<br>from<br>Study<br>Treatment? | Systemic/<br>Oral Corti-<br>costeroids<br>Taken? | Antibiotics<br>Taken? | A medication<br>Taken? | Hospitalized/<br>ER Visit/<br>Intubated? |
|---|---|---|---|---|---|---|---|---|
| xxxxxxx/<br>xxx/<br>xxxxx | XX | DDMMMYYYY/<br>DDMMMYYYY | XXXXXX | XXX | XXX | XXX | xxx | xxx/xxx/xxx |
| xxxxxxx/<br>xxx/<br>xxxxx | xx | DDMMMYYYY/<br>DDMMMYYYY | xxxxxx | XXX | XXX | XXX | XXX | xxx/xxx/xxx |
| xxxxxxx/<br>xxx/<br>xxxxx | XX | DDMMMYYYY/<br>DDMMMYYYY | xxxxxx | XXX | XXX | XXX | XXX | xxx/xxx/xxx |
| xxxxxxx/<br>xxx/<br>xxxxx | XX | DDMMMYYYY/<br>DDMMMYYYY | xxxxxx | XXX | XXX | XXX | XXX | xxx/xxx/xxx |
| ^^^^ | XX | DDMMMYYYY/<br>DDMMMYYYY | xxxxxx | XXX | xxx | XXX | XXX | xxx/xxx/xxx |

EFF\_L5


Population: Intent-to-Treat

## Listing xx Listing of Unscheduled Asthma Related Healthcare Utilisation

Treatment: Placebo

| , | Number of<br>Number of Home Visits | | physician urgent office/ care/ | Number of urgent care/ | Number of _ | Number of Inpatient Hospitalisation Days | | |
|---|---|---|---|---|---|---|---|---|
| Inv./ | Telephone | | | practice | outpatient | emergency | T 011 | General |
| Subj. | Calls | Day<br> | Night<br> | visits | visits<br> | room visits | ICU | Ward<br> |
| xxxxxx/ | X | X | X | Х | Х | x | X | X |
| xxxxxx. | | | | | | | | |
| XXXXXX | | | | | | | | |

EFF\_L11


Population: Intent-to-Treat

### Listing xx Listing of Peak Expiratory Flow (PEF) and Fractional Exhaled Nitric Oxide (FeNO) Results

| Site<br>I.D/<br>Subj. | Treatment<br>Arm | Visit | Date | PEF (unit) | FeNO (ppb) | FeNO Flow rate (mL/sec) |
|---|---|---|---|---|---|---|
| XXXX | xxxx | xxxxxxxx<br>xxxxxxxx | DDMMMYYYY<br>DDMMMYYYY | xxxxxxxx<br>xxxxxxxx | xxxxxxxx<br>xxxxxxxx | |

...

. . . .

Programming Note: Include the FeNO flow rate (mL/sec)